E-mail: lyudmill@niaid.nih.gov

## INNER-CITY ASTHMA CONSORTIUM

## **PROTOCOL ICAC-30**

# Mechanisms Underlying Asthma Exacerbations Prevented and Persistent with Immune-Based Therapy: A Systems Approach Phase 2

## **MUPPITS-2**

## Version 9.0 / 11Jan2021

Study Sponsor(s) The Division of Allergy, Immunology, and Transplantation

(DAIT), The National Institute of Allergy and Infectious

Diseases (NIAID)

NIAID Funding Mechanism Grants 1 UM1 Al114271-01 and UM2Al117870

IND Sponsor/Number IND sponsor: DAIT NIAID, IND# 136355

Study Drug Manufacturer/Provider GlaxoSmithKline

| - | | |
|---|---|---|
| PROTOCOL CO-CHAIR — | MEDICAL MONITOR – | BIOSTATISTICIAN — |
| DANIEL J. JACKSON, MD | PETER J. GERGEN, MD, MPH | CYNTHIA VISNESS, PHD |
| Associate Professor of Pediatrics | Division of Allergy, Immunology, | Senior Research Scientist |
| University of Wisconsin School of | and Transplantation – NIAID/NIH | Rho, Inc. |
| Medicine and Public Health | 5601 Fishers Lane, Room 6B58 | 2635 E NC Hwy 54 |
| 600 Highland Avenue | Rockville, MD 20892 MSC 9827 | Durham, NC 27713 |
| CSC K4/936 | Phone: (240) 627-3545 | Phone: (919) 408-8000 |
| Madison, WI 53792 | Fax: (301) 480-4258 | Fax: (919) 408-0999 |
| Phone: (608) 263-7686 | E-mail: pgergen@niaid.nih.gov | E-mail: |
| Fax: (608) 265-2207 | | cindy_visness@rhoworld.com |
| E-mail: djj@medicine.wisc.edu | | |
| PROTOCOL CO-CHAIR — | Project Manager – | REGULATORY OFFICER - |
| WILLIAM W. BUSSE, MD | LISA GAGALIS, RN, BSN | LYUDMILA LYAKH, MD, PHD |
| Professor of Medicine | Division of Allergy, Immunology, | Office of Regulatory Affairs |
| University of Wisconsin School of | and Transplantation | Division of Allergy, Immunology, |
| Medicine and Public Health | National Institute of Allergy and | and Transplantation |
| Ultratec Building, Rm. 129 | Infectious Diseases | National Institute of Allergy and |
| 5901 Research Park Blvd | 5601 Fishers Lane, Room 6B53 | Infectious Diseases |
| Madison, WI 53719 | Rockville, MD 20852-9828, USA | 5601 Fishers Lane, Room 7B39 |
| Phone: (608) 263-6183 | Phone: (240) 472-1823 | Rockville, MD 20892-9828, USA |
| Fax: (608) 261-1191 | Fax: (301) 480-4258 | Phone: (240) 627-3530 |
| Email: wwb@medicine.wisc.edu | E-mail: <u>lisa.gagalis@nih.gov</u> | Fax: (301) 480-1537 |

## **Confidentiality Statement**

The information contained within this document is not to be disclosed in any way without the prior permission of the Protocol Chair,

or the Division of Allergy, Immunology, and Transplantation, National Institute of Allergy and Infectious Diseases of the National Institutes of Health.



| INVESTIGATOR SIGNATURE PAGE | |
|---|---|
| Protocol: ICAC-30 | Version/Date: 9.0 / 11Jan2021 |
| Title: Mechanisms Underlying Asthma Exacerbations | Prevented and Persistent with Immune-Based |
| Therapy: A Systems Approach Phase 2 | |
| Study Sponsor: The Division of Allergy, Immunology, a | and Transplantation (DAIT), The National |
| Institute of Allergy and Infectious Diseases (NIAID) | |
| INSTRUCTIONS: | |
| The original signature page must be kept for your records signature page (*as described below) to the DAIT Regulat | , , , |
| RMC email address for the protocol/network: | |
| DAITRegulatory_ICAC (SM) < DAITRegulatory_ICAC@p | opdi.com> |
| I confirm that I have read the above protocol in the lat according to the principles of Good Clinical Practice (Grederal Regulations (CFR) – 45 CFR part 46 and 21 CFR Conference on Harmonisation (ICH) document Integrate E6(R1): Guideline for Good Clinical Practice E6(R2). Furth legal and regulatory requirements. | CP) as described in the United States Code of parts 50, 56, and 312, and in the International ted Addendum to ICH |
| As the site Principal Investigator, I agree to carry out th | |
| and understand that no changes can be made to this p | • |
| IRB and NIAID. All personnel involved in the conduct of Protection Training. | f this study have completed Human Subjects |
| I agree to ensure that all staff members involved in the obligations in meeting the above commitments. | e conduct of this study are informed about their |
| [*The site Principal Investigator should sign and date at ti | he indicated location below. A written |
| signature/date is acceptable (e.g., scanned and sent via e | email as a PDF version). An electronic signature is |
| also acceptable (e.g., sent via email as a PDF version).] | |
| Site Principal Investigator (Print) | |
| Site Principal Investigator (Signature) | <br>Date |

## **Protocol Synopsis**

| Title | Mechanisms Underlying Asthma Exacerbations Prevented and<br>Persistent with Immune-Based Therapy: A Systems Approach Phase 2 |
|---|---|
| Short Title | Protocol ICAC-30 MUPPITS-2 |
| Clinical Phase | II |
| Number of Sites | Multiple |
| IND Sponsor/Number | IND sponsor: DAIT NIAD IND#: 136355 |
| Study Objectives | The primary objective of the study is to determine if phenotype-directed use of mepolizumab reduces the rate of asthma exacerbations as defined by the need for systemic corticosteroid treatment in urban children and adolescents (ages 6-17) with difficult-to-control exacerbation-prone asthma and peripheral blood eosinophils ≥150 cells/μl. Secondary objectives are: 1. To determine whether mepolizumab will lead to an improved Composite Asthma Severity Index (CASI)¹ 2. To determine whether mepolizumab will improve quality of life as assessed by the physician-patient global assessment² 3. To determine whether mepolizumab improves lung function as assessed by spirometry and impulse oscillometry 4. To determine whether mepolizumab increases the time to first asthma exacerbation 5. To separately determine whether mepolizumab reduces the rate of asthma exacerbations in study participants who do not fit the FDA-approved dosing table for omalizumab therapy and in study participants who fit the FDA-approved dosing table for omalizumab therapy 6. To assess the safety of mepolizumab treatment |
| Study Design | Protocol ICAC-30 MUPPITS-2 is a multicenter, double-blind, placebo-<br>controlled, randomized trial of mepolizumab adjunctive therapy for the<br>prevention of asthma exacerbations in urban children and adolescents |

| | with difficult-to-control exacerbation-prone asthma and peripheral blood eosinophils ≥150 cells/μl. |
|---|---|
| Primary Endpoint(s) | The primary endpoint is the number of asthma exacerbations during the 12-month treatment period. |
| Secondary Endpoint(s) | <ol> <li>CASI during the treatment period</li> <li>Quality of life as measured by the physician-patient global assessment</li> <li>Lung function as assessed by spirometry and IOS during the treatment period</li> <li>Time to first asthma exacerbation during the treatment period</li> <li>Number of reported adverse events and serious adverse events, including their severity and treatment relatedness</li> </ol> |
| Accrual Objective | 290 |
| Study Duration | 15 months recruitment + 12 months treatment |
| Agent/Treatment Description | <ul> <li>Mepolizumab (anti-IL-5 antagonist monoclonal antibody) by subcutaneous injection every 4 weeks at the following doses: <ul> <li>Age 12 years and above: 100 mg</li> <li>Age 6-11 years: 40mg</li></ul></li></ul> |
| Inclusion Criteria | <ol> <li>Participant and/or parent guardian must be able to understand and provide informed consent and age-appropriate assent</li> <li>Are male and female aged 6-17 years, inclusive at randomization</li> <li>Have a primary place of residence in one of the pre-selected recruitment census tracts as outlined in the Protocol ICAC-30 Recruitment Manual of Operations</li> <li>Participants who do not live in the pre-selected census tracts but live within the Office of Management and Budget (OMB) defined Metropolitan Statistical Area and have publicly-funded health insurance will qualify for inclusion.</li> </ol> |

- 4. Have had a diagnosis of asthma made > 1 year prior to recruitment; participants who received an asthma diagnosis by a clinician ≤ 1 year prior to recruitment must report that their respiratory symptoms were present for more than 1 year prior to recruitment
- Have had at least two asthma exacerbations in the prior year (defined as a requirement for systemic corticosteroids and/or hospitalization)
- 6. At Visit 0 (Screening), have the following requirement for asthma controller medication: for participants aged 6 to 11 years, treatments with at least fluticasone 250 mcg dry powder inhaler (DPI) one puff twice daily or its equivalent and for participants aged 12 years and older, treatment with at least fluticasone 250 mcg plus LABA DPI one puff twice daily or its equivalent
- 7. Have peripheral blood eosinophils ≥150 cells/μl obtained at Visit 0 or via another ICAC protocol within 6 months
- 8. Are able to perform spirometry at randomization
- 9. Have documentation of current medical insurance with prescription coverage at randomization
- 10. Have had varicella or the varicella vaccination

## **Exclusion Criteria**

Individuals who meet any of the following criteria are not eligible for enrollment or randomization, if they:

- Are not able or willing to give written informed consent or comply with study protocol
- 2. Have concurrent medical problems that would require systemic corticosteroids or other immunomodulators during the study
- 3. Are currently receiving immunotherapy
- 4. Are currently receiving treatment with omalizumab or have had omalizumab treatment within 6 months prior to randomization
- 5. Are currently requiring greater than fluticasone 500 mcg bid plus LABA one puff twice daily or its equivalent and/or individuals using oral corticosteroids daily or every other day for more than 14 days at the time of Visit 0 (Screening)
- Are currently pregnant or lactating, or plan to become pregnant during the time of study participation. Females of child-bearing potential (post-menarche) must be abstinent or use a medically acceptable birth control method throughout the study (e.g. oral subcutaneous, mechanical, or surgical contraception)
- 7. Have a known, pre-existing clinically important lung condition other than asthma
- 8. Have a current malignancy or previous history of cancer in remission for less than 12 months prior to randomization

| Study Stopping Rules | The occurrence of one death or an unexpected SAE related to the investigational agent. |
|---|---|
| | <ol> <li>Is a current smoker</li> <li>Have a known immunodeficiency disease</li> <li>Have other conditions that could lead to elevated eosinophils such as hypereosinophilic syndromes, including eosinophilic granulomatosis with polyangiitis</li> <li>Have a known, active pre-existing parasitic infestation or undergoing treatment for a parasitic infestation. Once the participant has been successfully treated, the participant may be reevaluated.</li> <li>Use of investigational drugs within 4 weeks of randomization</li> <li>Have past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study</li> <li>Will not allow the study clinician, an asthma specialist, to manage their disease for the duration of the study or who are not willing to change their asthma medications to follow the protocol</li> <li>Have a known history of allergic reaction to previous biologic therapy for asthma</li> <li>Have had a life threatening asthma exacerbation in the last 2 years requiring intubation, mechanical ventilation or resulting in a hypoxic seizure</li> </ol> |
| | 9. Have known, pre-existing, unstable liver disease |

## **Table of Contents**

| 1 | Bac | kground and Rationale | . 15 |
|---|---|---|---|
| | 1.1 | Background and Scientific Rationale | . 15 |
| | 1.2 | Rationale for Selection of Investigational Product or Intervention | . 16 |
| | 1.3 | Preclinical Experience | . 17 |
| | 1.4 | Clinical Studies | . 17 |
| 2 | Stu | dy Hypotheses/Objectives | . 19 |
| | 2.1 | Hypotheses | . 19 |
| | 2.2 | Primary Objective(s) | . 19 |
| | 2.3 | Secondary Objective(s) | . 19 |
| | 2.4 | Exploratory Objective(s) | . 19 |
| 3 | Stu | dy Design | . 20 |
| | 3.1 | Description of Study Design | . 20 |
| | 3.2 | Primary Endpoint | . 21 |
| | 3.3 | Secondary Endpoint(s)/Outcome(s) | . 21 |
| | 3.4 | Exploratory Endpoint(s)/Outcome(s) | . 21 |
| | 3.5 | Stratification, Randomization, and Blinding/Masking | . 22 |
| | 3.5. | 1 Procedure for Unblinding/Unmasking | . 22 |
| 4 | Sele | ection of Participants and Clinical Sites/Laboratories | . 23 |
| | 4.1 | Rationale for Study Population | . 23 |
| | 4.2 | Inclusion Criteria | . 23 |
| | 4.3 | Exclusion Criteria | . 24 |
| 5 | Knc | own and Potential Risks and Benefits to Participants | . 26 |
| | 5.1<br>meno | Risks of Investigational Product or Intervention as Cited in GSK Investigator's Brochure for lizumab | . 26 |
| | 5.2 | Risks of Investigational Product or Intervention Cited in Medical Literature | |
| | 5.3 | Risks of Other Protocol Specified Medications | |
| | 5.3. | 1 Oral Corticosteroids | . 27 |
| | 5.4 | Risks of Study Procedures | . 27 |
| | 5.4. | 1 Allergy Skin Testing | . 27 |
| | 5.4. | 2 Blood Collection | . 27 |
| | 5.4. | 3 Pulmonary Function Testing (Spirometry and Impulse Oscillometry) | . 27 |
| | 5.4. | | |
| _ | | ICAC COLAMARRITO D | 10.4 |

| | 5.4.5<br>5.4.6<br>5.4.7 | | 5 | Nasal Sample Collection | 28 |
|---|---|---|---|---|---|
| | | | ô | Sputum Induction | 29 |
| | | | 7 | Nasal Epithelial Cell Collection | 29 |
| | | 5.4.8 | 3 | Questionnaires | 29 |
| | 5. | 5 | Pote | ntial Benefits | 29 |
| 6 | | Inve | stigat | tional Agent | 29 |
| | 6. | 1 | Inve | stigational Agent: Mepolizumab | 29 |
| | | 6.1.1 | L | Formulation, Packaging, and Labeling | 29 |
| | | 6.1.2 | 2 | Dosage, Preparation, and Administration | 30 |
| | 6. | 2 | Place | ebo | 30 |
| | 6. | 3 | Drug | g Accountability | 30 |
| | 6. | 4 | Asse | ssment of Participant Compliance with Investigational Agent | 30 |
| | 6. | 5 | Toxi | city Prevention and Management | 31 |
| | 6. | 6 | Pren | nature Discontinuation of Study Participation | 31 |
| | 6. | 7 | Pren | nature Discontinuation of Investigational Product | 31 |
| 7 | | Othe | er Me | edications | 31 |
| | 7. | 1 | Cond | comitant Medications | 31 |
| | | 7.1.1 | L | Protocol-mandated | 31 |
| | | 7.1.2 | 2 | Other permitted concomitant medications | 37 |
| | 7. | 2 | Prop | hylactic Medications | 37 |
| | 7. | 3 | Proh | ibited Medications | 37 |
| | 7. | 4 | Resc | ue Medications | 38 |
| | | 7.4.1 | 1 | Definition and Management of Acute Exacerbations | 38 |
| 8 | | Stud | ly Pro | ocedures | 38 |
| | 8. | 1 | Stud | y Procedures | 38 |
| | | 8.1.1 | L | Vital Signs and Growth Parameters | 39 |
| | | 8.1.2 | 2 | Medical History and Physical Examination | 39 |
| | | 8.1.3 | 3 | Aeroallergen Skin Testing | 39 |
| | | 8.1.4 | 1 | Measurement of Fractional Exhaled Nitric Oxide | 40 |
| | | 8.1.5 | 5 | Measurement of Pulmonary Function | 40 |
| | | 8.1.6 | 5 | Questionnaire Assessments | 41 |
| | 8. | 2 | Clini | cal and Research Laboratory Evaluations and Specimen Collection | 41 |
| | | 8.2.1 | 1 | Blood Sample Collection | 41 |

| | 8.2. | 2 N | Nasal Sample Collection | 41 |
|---|---|---|---|---|
| 8.2.3<br>8.2.4 | | 3 ι | Jrine Pregnancy Testing | 42 |
| | | 4 ι | Jrine Cotinine | 42 |
| | 8.2. | 5 I | nduced Sputum | 42 |
| | 8.2. | 6 1 | Nasal Epithelial Cell Collection | 42 |
| | 8.3 | Recru | itment | 42 |
| | 8.4 | Scree | ning/Baseline Visit | 43 |
| | 8.5 | Rando | omization | 44 |
| | 8.6 | Visit 2 | 2 (Week 8) | 45 |
| | 8.7 | Visit 3 | 3 (Week 12) | 45 |
| | 8.8 | Inject | ion Only Visits (Visits 5, 6, 8, 9, 11, 12) | 46 |
| | 8.9 | Asthn | na Evaluation and Management Visits (Visits 4, 7, 10, 13) | 46 |
| | 8.10 | Final | Visit (Visit 14) | 46 |
| | 8.11 | Cold \ | /isits | 47 |
| | 8.12 | Exace | rbation Follow-Up Visits | 47 |
| | 8.13 | Unsch | neduled Visits and Telephone Follow-up | 48 |
| | 8.14 | Visit \ | Vindows | 48 |
| 9 | Med | chanist | ic Assays | 48 |
| 1 | 0 Bi | iospeci | imen Storage | 49 |
| 1 | 1 C | riteria | for Participant and Study Completion and Premature Study Termination | 49 |
| | 11.1 | Partic | ipant Completion | 49 |
| | 11.2 | Partic | ipant Stopping Rules and Withdrawal Criteria | 49 |
| | 11.3 | Partic | ipant Replacement | 50 |
| | 11.4 | Follov | v-up after Early Study Withdrawal | 50 |
| | 11.5 | Study | Stopping Rules | 50 |
| 1 | 2 Sa | afety N | Nonitoring and Reporting | 51 |
| | 12.1 | Overv | riew | 51 |
| | 12.2 | Defini | itions | 51 |
| | 12.2 | 2.1 A | Adverse Event (AE) | 51 |
| | 12.2 | 2.2 l | Jnexpected Adverse Event | 53 |
| | 12.2 | 2.3 | Serious Adverse Event | 53 |
| | 12.3 | Gradi | ng and Attribution of Adverse Events | 54 |
| | 12.3 | 3.1 | Grading Criteria | 54 |

| | 12.3 | 3.2 | Attribution Definitions | 57 |
|---|---|---|---|---|
| | 12.4 | Colle | ection and Recording of Adverse Events | 58 |
| | 12.4 | 4.1 | Collection Period | 58 |
| | 12.4 | 1.2 | Collecting Adverse Events | 58 |
| | 12.4 | 1.3 | Recording Adverse Events | 58 |
| | 12.5 | Rep | orting of Serious Adverse Events and Adverse Events | 58 |
| | 12.5 | 5.1 | Reporting of Serious Adverse Events to the IND Sponsor (DAIT NIAID) | 58 |
| | 12.5 | 5.2 | Reporting to FDA | 59 |
| | 12.5 | 5.3 | Reporting of Adverse Events to IRBs | 60 |
| | 12.6 | Preg | nancy Reporting | 60 |
| | 12.7 | Rep | orting of Other Safety Information | 61 |
| | 12.8 | Revi | ew of Safety Information | 61 |
| | 12.8 | 3.1 | Medical Monitor Review | 61 |
| | 12.8 | 3.2 | DSMB Review | 61 |
| 13 | S | tatisti | ical Considerations and Analytical Plan | 61 |
| | 13.1 | Ove | rview | 62 |
| | 13.2 | End | points/Outcomes | 62 |
| | 13.3 | Mea | sures to Minimize Bias | 62 |
| | 13.4 | Ana | lysis Plan | 63 |
| | 13.4 | 1.1 | Analysis Populations | 63 |
| | 13.4 | 1.2 | Primary Analysis of Primary Endpoint(s)/Outcome(s) | 63 |
| | 13.4 | 1.3 | Supportive Analyses of the Primary Endpoint(s)/Outcome(s) | 63 |
| | 13.4 | 1.4 | Analyses of Secondary and Other Endpoint(s)/Outcome(s) | 64 |
| | 13.4 | 1.5 | Analyses of Exploratory Endpoint(s)/Outcome(s) | 65 |
| | 13.4 | 1.6 | Descriptive Analyses | 65 |
| | 13.5 | Inte | rim Analyses | 65 |
| | 13.5 | 5.1 | Interim Analysis of Efficacy Data | 66 |
| | 13.5 | 5.2 | Interim Analysis of Safety Data | 6e |
| | 13.5 | 5.3 | Futility Analysis | 66 |
| | 13.6 | Stat | istical Hypotheses | 66 |
| | 13.7 | Sam | ple Size Considerations | 66 |
| 14 | · Ic | dentif | ication and Access to Source Data | 67 |
| | 14.1 | Soui | rce Data | 67 |

| 14.2 | Access to So | ource Data | 67 |
|---|---|---|---|
| 15 P | rotocol Devia | ations | 67 |
| 15.1 | Protocol De | eviation Definitions | 67 |
| 15.2 | 1 Protoco | col Deviation | 67 |
| 15.2 | 2 Major l | Protocol Deviation | 68 |
| 15.2 | 3 Non-M | Najor Protocol Deviation | 68 |
| 15.2 | Reporting a | and Managing Protocol Deviations | 68 |
| 16 E | thical Conside | lerations and Compliance with Good Clinical Practice | 68 |
| 16.1 | Quality Cont | ntrol and Quality Assurance | 68 |
| 16.2 | Statement o | of Compliance | 69 |
| 16.3 | Informed Co | onsent Process | 69 |
| 16.4 | Privacy and | l Confidentiality | 69 |
| 17 P | ublication Po | olicy | 69 |
| 18 R | eferences | | 70 |
| Appendi | A: Schedul | le of Procedures/Evaluations | 72 |
| Appendi | k B: Nasal Lav | vage Quality Control Methods | 74 |
| 1 Stud | dy Population | n | 74 |
| 1.1 | Population [ | Description | 74 |
| 1.1. | 1 Inclusio | on Criteria | 74 |
| 1.2 | Requiremen | nts | 74 |
| 1.3 | Procedures . | · | 74 |
| Appendi | c C: Omalizun | mab Dosing Tables | 75 |
| Appendi | CD: Sputum | Induction Quality Control Methods | 77 |
| 1 Stud | dy Population | n | 77 |
| 1.1 | Population [ | Description | 77 |
| 1.1. | 1 Inclusio | on Criteria | 77 |
| 1.2 | Requiremen | nts | 77 |
| 1.3 | Procedures . | | 77 |
| Appendi | κ Ε: Study Re | estrictions Due to COVID-19 | 78 |

## **Glossary of Abbreviations**

| ACT | Asthma Control Test |
|------------------|------------------------------------------------------|
| AE | Adverse Event |
| APIC | Asthma Phenotypes in the Inner City |
| ATS | American Thoracic Society |
| BID | Bis in die (twice a day) |
| ВР | Blood pressure |
| BMI | Body Mass Index |
| CASI | Composite Asthma Severity Index |
| CBC | Complete blood count |
| CFR | Code of Federal Regulations |
| CRF | Case report form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DAIT | Division of Allergy, Immunology, and Transplantation |
| DPI | Dry powder inhaler |
| DSMB | Data Safety Monitoring Board |
| ECP | Eosinophil cationic protein |
| eCRF | Electronic case report form |
| ED | Emergency department |
| E&M | Evaluation and Management |
| EPR-3 | Expert Panel Report 3 |
| FDA | Food and Drug Administration |
| FeNO | Fractional exhaled nitric oxide |
| FEV <sub>1</sub> | Forced expiratory volume in 1 second |
| GCP | Good Clinical Practice |
| GSK | GlaxoSmithKline (GSK) Group Company |

| HIPAA | Health Insurance Portability and Accountability Act |
|-------|-------------------------------------------------------|
| ICAC | Inner City Asthma Consortium |
| ICATA | Inner City Anti-IgE Therapy in Asthma |
| ICH | International Conference on Harmonisation |
| ICS | Inhaled corticosteroid |
| IgE | Immunoglobulin E |
| IgG | Immunoglobulin G |
| IL | Interleukin |
| IND | Investigational New Drug |
| IOS | Impulse oscillometry |
| IRB | Institutional Review Board |
| ІТТ | Intent-to-treat |
| LABA | Long-acting beta agonist |
| МОР | Manual of Procedures |
| NAEPP | National Asthma Education and Prevention Program |
| NCI | National Cancer Institute |
| NIAID | National Institute of Allergy and Infectious Diseases |
| OHRP | Office of Human Research Protections |
| PCP | Primary care provider |
| PEF | Peak expiratory flow |
| PD | Protocol deviation |
| PP | Per Protocol |
| PFT | Pulmonary function tests |
| PHI | Personal health identifiers |
| PI | Principal Investigator |
| RV | Rhinovirus |
| | i . |

| SACCC | Statistical and Clinical Coordinating Center |
|-------|-----------------------------------------------|
| SAE | Serious adverse event |
| SAR | Suspected adverse reaction |
| SQ | Subcutaneous |
| SUSAR | Serious unexpected suspected adverse reaction |
| URECA | The Urban Environment and Childhood Asthma |

## 1 Background and Rationale

## 1.1 Background and Scientific Rationale

Asthma is the most common chronic disease of childhood, and is associated with \$56 billion in health care costs in the United States annually. Episodic exacerbations are the major source of morbidity, mortality, and health care costs due to asthma. These events are particularly common in at risk urban children and adolescents with asthma. Importantly, exacerbations lead to progressive loss of lung function <sup>3,4</sup> which contributes to increasing asthma severity over time. Moreover, it has recently been shown that a significant number of children with mild to moderate asthma at early school age progress to a pattern of fixed obstructive lung disease by early adulthood. <sup>5</sup> Thus, it is a major unmet need to prevent asthma exacerbations, particularly in exacerbation-prone children.

Protocol ICAC-30 MUPPITS-2 clinical trial is designed to determine whether an intervention that is directed towards a phenotype-defined population of urban children and adolescents with difficult-to-control, exacerbation-prone asthma will improve disease management by preventing exacerbations. For a significant number of asthma patients, guidelines-directed treatment does not achieve disease control, suggesting the need, and potential benefit, for treatment(s) that are personalized to the phenotype of these patients. This trial is informed by the DAIT NIAID-sponsored Inner-City Asthma Consortium (ICAC) 2 trial, Protocol ICAC-19, titled "Asthma Phenotypes in the Inner City", <sup>6-8</sup> and based on these observations and others in the literature<sup>9</sup>, the presence of peripheral blood eosinophils in patients with difficult-to-control asthma, despite appropriate guidelines-directed care, is a biomarker for asthma exacerbations and increased morbidity. Therefore, we hypothesize that targeting eosinophils with the addition of the anti-IL-5 monoclonal antibody, mepolizumab, will prevent exacerbations and, as a consequence, reduce overall morbidity, improve asthma control, and quality of life.

To date, phenotype-directed trials using biologic agents have been performed primarily in adults. Protocol ICAC-30 MUPPITS-2 is designed to test whether this approach is effective in urban children and adolescents with difficult-to-control, exacerbation-prone asthma. From a public health perspective, the proposed trial will inform clinical guidelines for care of children at EPR3 Step 4 care and above, where there is currently a paucity of data to guide treatment decisions. The information will not only be useful in the inner-city population but also for the overall management of difficult-to-control, exacerbation-prone asthma in the pediatric age group. This trial will serve as a model for future phenotype-directed protocols for difficult-to-control, exacerbation-prone asthma in at-risk urban youth. Finally, our focus on underlying mechanisms using whole genome transcriptomics of nasal airway and peripheral blood will provide insight to mechanisms by which eosinophils and IL-5 contribute to exacerbations. Furthermore, the transcriptomic characteristics of exacerbations that persist despite anti-IL5 therapy will provide potential new therapeutic targets for the treatment of this difficult-to-control, exacerbation-prone asthma phenotype.

Protocol ICAC-30 MUPPITS-2 is a randomized, double-blind, placebo-controlled, parallel-group, multi-center trial of the efficacy and safety of mepolizumab adjunctive therapy for 12 months in urban asthma patients aged 6-17 years with difficult-to-control, exacerbation-prone asthma with an eosinophilic phenotype (defined by a peripheral blood eosinophil count ≥150 cells/µl).

## 1.2 Rationale for Selection of Investigational Product or Intervention

Nucala<sup>®</sup> <sup>10</sup> is an interleukin-5 antagonist monoclonal antibody (IgG1 kappa) indicated in the United States for add-on maintenance treatment of patients with severe asthma aged 12 years and older, with an eosinophilic phenotype.

Asthma exacerbations are most commonly associated with viral respiratory infections, with human rhinoviruses (RV) the most frequent <sup>11-13</sup>. A number of risk factors for exacerbations with respiratory infections have been identified including underlying allergic disease, allergic inflammation and a T2 sputum cell profile<sup>11</sup>. The mechanisms underlying a reduction in asthma exacerbations associated with mepolizumab treatment <sup>14</sup> are unknown, and a greater understanding of mechanisms responsible for this effect will improve our understanding of the pathogenesis of asthma exacerbations<sup>15</sup>. Because IL-5 is an important survival factor for eosinophils, the reduction in exacerbations is commonly thought to reflect the depletion in airway eosinophils, but this begs the question as to how airway eosinophils predispose to asthma exacerbations. We hypothesize that eosinophil products activate epithelial cell production of chemoattractants for other inflammatory cell types, such as mast cells and CD4+T lymphocytes. Based on this hypothesis, we expect that IL-5 inhibition will have broad effects on cellular inflammation in the airway. In particular, we anticipate that anti-IL-5 treatment will decrease airway mast cells and airway T2 inflammation<sup>16</sup>.

A major unmet need in asthma care is to improve outcomes of disease control in patients with more severe disease that is not responsive to current therapy<sup>17</sup>. We have observed a pattern of treatment response in urban children where, despite intensive efforts to prevent asthma morbidity with asthma counseling<sup>18</sup>, cockroach allergen home mitigation<sup>19</sup>, and optimized guidelines-based asthma management including high-dose inhaled corticosteroids (ICS), long-acting beta-agonists (LABA), and omalizumab<sup>20,21</sup>, exacerbations still occurred frequently and disease control was not always achieved. 48% of 400 ICAC participants who were managed for one year with guidelines-based care (i.e., the control participants in the ICAC Asthma Control Evaluation (ACE)<sup>21</sup> and DAIT NIAID-sponsored clinical trials (IND #100, 210) – Protocol ICAC-08/09, titled "Inner-City Anti-IgE Therapy in Asthma (ICATA)"<sup>20</sup>) had at least one asthma exacerbation requiring a course of systemic corticosteroids, and 24% of the control treated patients in ICATA had at least two exacerbations. Importantly, exacerbations have been associated with progressive loss of lung function over time <sup>3,22</sup>. Given the existing shortcomings in the effectiveness of current treatments for a significant proportion of children and adolescents with asthma, particularly those in urban environments, a new approach for their management is needed to improve disease control and reduce morbidity, focusing on exacerbations.

One consideration in selecting a treatment in high-risk children and adolescents with difficult-to-control asthma is feasibility and a conveniently measurable marker to predict an effective response, i.e. high blood eosinophils. Mepolizumab meets these criteria and can be given monthly in a subcutaneous injection. Moreover, novel immune biologics are not necessarily good candidates for children/adolescents unless they have been well tested in older participants and their efficacy and safety demonstrated. Although a developing array of immune-based therapeutics may also be reasonable candidates for a phenotypic biomarker-directed approach to difficult asthma in at-risk urban youth, they are not sufficiently advanced at this time.

## 1.3 Preclinical Experience

In mice, anti-IL-5 monoclonal antibodies removed eosinophils and virtually eliminated allergic inflammation and pulmonary dysfunction associated with antigen provocation <sup>23</sup>.

#### 1.4 Clinical Studies

The assessment of mepolizumab's effectiveness in asthma in adults has been instructive for the need to identify appropriate patient populations to comprehensively evaluate new therapies, and is applicable to our proposed clinical trials in urban children and adolescents. In an initial clinical trial, Leckie et al <sup>24,25</sup> found mepolizumab significantly reduced peripheral blood and sputum eosinophils, but did not



Figure 4. Mepolizumab reduces asthma exacerbations

block either the late phase response to antigen or the post-challenge increase in airway hyper-responsiveness. These results were a major surprise and raised the possibility that eosinophils, despite their much-recognized relationship to multiple features of asthma, may not have a major pathophysiological role in in this disease. When Flood-Page et al <sup>10</sup> tested mepolizumab in a large population of patients with moderate-to-severe asthma, lung function, symptoms and exacerbations did not improve. There was, however, a trend towards reduced exacerbations in a subpopulation of patients.

At the same time, Green et al <sup>26</sup> compared treatment by British Thoracic Society guidelines to the addition of extra ICS aimed at the reduction of sputum eosinophils. The reduction in sputum eosinophils was associated with a decrease in the frequency of exacerbations. This relationship to the prevention of exacerbations was further confirmed by Haldar et al <sup>25</sup> and Nair et al <sup>27</sup> who evaluated mepolizumab in patients with severe asthma who required high doses of ICS and, in most cases, systemic prednisone, for disease control, but yet had frequent exacerbations and, importantly, persistent sputum and peripheral blood eosinophils. In a one-year treatment with mepolizumab, Haldar et al 25 found the frequency of exacerbations decreased by approximately 50% (Figure 4). Nair et al <sup>27</sup> found similar effects with mepolizumab. No changes in asthma symptoms, need for rescue treatment, or lung function measures were noted in either trial. Pavord et al <sup>14</sup> substantiated these findings with mepolizumab in a large trial. More recently, two additional trials demonstrated similar efficacy for exacerbation prevention using subcutaneous administration of mepolizumab, a more patient friendly route of administration than the intravenous administration in earlier trials <sup>2,28,29</sup>. Therefore, the phenotype-profile in asthma where mepolizumab has been found to be effective is: difficult-to-control asthma with frequent exacerbations and the presence of eosinophils despite ongoing ICS treatment, with the primary outcome being prevention of exacerbations. Since mepolizumab effectively reduces exacerbations and also leads to a reduction in airway area as assessed by high-resolution computerized tomography scans after one year of treatment <sup>26</sup>, it is intriguing to suggest that mepolizumab in school-age children and adolescents, who are exacerbation-prone, has the potential to prevent progressive loss of lung function and disease progression with time.

1. What information can be used to select urban children and adolescents with difficult-to-control asthma for a trial with mepolizumab? A meta-analysis of mepolizumab in adult patients with severe

Protocol ICAC-30 MUPPITS-2

Version 9.0

01/11/21

asthma and persistent eosinophilia revealed significant reductions in the risk for exacerbation across seven trials (OR 0.30 95% CI 0.13 to 0.67, p=0.004)  $^{30}$ . Studies of mepolizumab in adults have identified consistent benefit in exacerbation-prone participants whose peripheral blood eosinophil counts are  $\geq$ 150 cells/ $\mu$ I<sup>2,29</sup>. A post-hoc analysis of the relationship between blood eosinophilia and asthma exacerbations in

the Protocols
ICAC-08/09
ICATA trials
demonstrated
that elevated
peripheral
blood
eosinophils at
randomization
were
significantly
associated with
an increased
risk of

**Table 1.4**. Association between Blood Eosinophils at Randomization and Exacerbations during the Protocols ICAC-08/09 ICATA Double Blind Treatment Phase.

| Blood EOS at | | | | OR | | |
|---|---|---|---|---|---|---|
| Group | Randomization | Size | Exacerbation | Difference | (95% CI) | p-value |
| Both<br>Placebo +<br>Omalizumab | < 340 | 65%<br>(243/373) 33% | 100/ | 2.23 | 0.0003 | |
| | ≥ 340 | 35%<br>(130/373) | 52% | 19% | (1.44, 3.46) | 0.0003 |
| Placebo | < 340 | 64%<br>(116/181) | 41% | 21% | 2.27<br>(1.21, 4.23) | 0.0120 |
| | ≥ 340 | 36%<br>(65/181) | 62% | | | |
| Omalizumab | < 340 | 66%<br>(127/192) | 25% | 18% | 2.25 | 0.0127 |
| | 34%<br>≥ 340 (65/192) | | 43% | | (1.19, 4.24) | 0.0127 |

EOS=eosinophils; OR=odds ratio

exacerbations.

In these analyses, the optimum cut-point for eosinophils was 340 cells/ $\mu$ l (52% vs. 33% over the 12 month treatment period; p=0.0003: **Table 1.4**). Interestingly, and important in the selection of an intervention most likely to be effective in children with uncontrolled asthma, was the finding that exacerbation rates remained high (43%) even in children treated with omalizumab. Thus, even with conventional guidelines-based asthma management, including omalizumab, patients with peripheral blood eosinophilia continue to have frequent exacerbations. These findings suggest that an alternative therapeutic agent than omalizumab may be the best intervention. Given the effect of mepolizumab on exacerbations and its safety profile, mepolizumab is an ideal choice.

Additional analyses of the Protocol ICAC-19 APIC study population characteristics at study screening demonstrate that the typical characteristics utilized in adult mepolizumab trials [eosinophils  $\geq$ 150 cells/ $\mu$ l,  $\geq$ 2 exacerbations in the prior year, and requirement for high level controller therapy (6-11 years: fluticasone DPI 250 mcg BID or equivalent, 12 and above: fluticasone/salmeterol DPI 250/50 mcg BID or equivalent)] identifies urban youth at high risk for exacerbation. Children meeting these characteristics had a 70% risk of exacerbation during the Protocol ICAC-19 APIC 12 month follow up despite guidelines-based care and good adherence with medications.

2. What are potential advantages of mepolizumab in this population? Mepolizumab is administered as a fixed subcutaneous dose of 100 mg every 4 weeks for patients aged 12 years and above; 40 mg every 4 weeks for patients aged 6 to 11 years. These doses are consistent with the approved dosing per the Package Insert (September 2019). The use of mepolizumab will allow us to include children who were not eligible for our previous omalizumab studies (ICAC-08/09/20). For example, in DAIT-Sponsored Protocols ICAC-08/09 ICATA, 35% of children and adolescents identified with exacerbation-prone asthma were ineligible for enrollment due to their weight and/or total serum IgE level. In fact, more

than 50% of Protocol ICAC-19 APIC participants with difficult-to-control, exacerbation prone asthma would have been ineligible for omalizumab therapy based upon weight, total serum IgE level, or lack of aeroallergen sensitization. Of note, a post hoc analysis of the DREAM (Mepolizumab for Severe Eosinophilic Asthma) study suggests that this subgroup of patients with high body mass indices (BMIs) may be particularly responsive to mepolizumab<sup>29</sup>. Further, in the presence of elevated eosinophils, adult patients with and without aeroallergen sensitization responded similarly to mepolizumab<sup>31</sup>. In the same analysis, mepolizumab responses were similar across quartiles of total serum IgE<sup>31</sup>. Thus, it is possible that mepolizumab may be particularly effective in patients who do not fit the current omalizumab dosing paradigm, and have the potential to meet an important unmet need for this group of approximately 50% of urban youth with difficult to control, exacerbation prone asthma.

## 2 Study Hypotheses/Objectives

## 2.1 Hypotheses

The primary research question of this study is whether mepolizumab will lead to a reduced rate of asthma exacerbations in urban children and adolescents (ages 6-17) with difficult-to-control, exacerbation-prone asthma and peripheral blood eosinophils ≥150 cells/µl. We hypothesize that targeting eosinophils with the addition of the anti-IL-5 monoclonal antibody, mepolizumab, will prevent exacerbations and, as a consequence, reduce overall morbidity and improve asthma control. We will also explore the mechanistic hypothesis that IL-5 inhibition will have broad effects on T2 inflammation in the airways.

## 2.2 Primary Objective(s)

The primary objective of this study is to determine whether mepolizumab, in addition to guidelines-based care, will reduce the rate of asthma exacerbations compared to guidelines-based care alone.

## 2.3 Secondary Objective(s)

Secondary objectives are:

- 1. To determine whether mepolizumab will lead to an improved Composite Asthma Severity Index (CASI)<sup>1</sup>
- 2. To determine whether mepolizumab will improve quality of life as assessed by the physicianpatient global assessment<sup>2</sup>
- 3. To determine whether mepolizumab improves lung function as assessed by spirometry and impulse oscillometry
- 4. To determine whether mepolizumab increases the time to first asthma exacerbation
- 5. To separately determine whether mepolizumab reduces the rate of exacerbations in study participants who do not fit the FDA-approved dosing table (see Appendix C) for omalizumab therapy and in study participants who fit the FDA-approved dosing table for omalizumab therapy
- 6. To assess the safety of mepolizumab treatment

### 2.4 Exploratory Objective(s)

Exploratory objectives are:

- 1. To determine whether the following patient characteristics/biomarkers predict response to mepolizumab:
  - BMI percentile
  - Peripheral blood eosinophils
  - Bronchodilator responsiveness at baseline
  - Exacerbation history in year prior to study (2, 3 or 4+)
  - Total serum IgE
  - Fractional exhaled nitric oxide
  - Nasal mucus eosinophil cationic protein (ECP)
- To determine whether mepolizumab improves other important clinical outcomes, including rate
  of virus-induced asthma exacerbations, time to first virus-induced asthma exacerbation, Asthma
  Control Test (ACT) scores, maximum number of asthma symptom days, and bronchodilator
  response
- 3. To use transcriptomics to identify immunologic pathways in the airways and peripheral blood that are characteristic of exacerbations prevented with and persistent despite anti-IL5 therapy.
- 4. To measure levels of antibody to mepolizumab

## 3 Study Design

## 3.1 Description of Study Design

Protocol ICAC-30 MUPPITS-2 is a multicenter, double-blind, placebo-controlled, randomized trial of mepolizumab adjunctive therapy for the prevention of asthma exacerbations in urban children and adolescents 6 to 17 years with exacerbation-prone asthma and peripheral blood eosinophilia. Approximately 290 participants will be randomized 1:1 to one of two study arms: 1) guidelines-based asthma treatment + placebo, or 2) guidelines-based asthma treatment + mepolizumab. All participants will be followed for one year.

There will be a Screening Visit followed by a 4-week run-in period. After the run-in, children who continue to meet eligibility criteria will be randomized to one of the 2 treatment arms and receive their first injection. Participants will receive monthly injections of either 40 mg or 100 mg of mepolizumab/placebo administered subcutaneously, according to their age. Participants 6 to 11 years of age and weighing ≥40 kg who were enrolled in Protocol ICAC-30 under the previous versions of the protocol and initially assigned a 100 mg dose will have their dose reduced to 40 mg. Participants who receive the 40 mg dose at randomization will increase to the 100 mg dose if they become 12 years old during the study. All participants will have Evaluation and Management (E&M) visits every 3 months where their asthma will be assessed and adjustments made to their medications based on asthma guidelines.

Participants will be asked to monitor and report cold symptoms. Participants will come to the clinic at the time of a cold, up to three times, for collection of blood and nasal secretions for associated mechanistic studies.

Participants will also be asked to come into the clinic following an asthma exacerbation for collection of blood and nasal secretions for associated mechanistic studies, assessments of airway physiology, and to collect information for ongoing asthma management.



Figure 3.1. Protocol ICAC-30 MUPPITS-2 Study Design

## 3.2 Primary Endpoint

The primary endpoint is the number of asthma exacerbations during the 12-month treatment period. Exacerbations will be defined as a prescription of a course of systemic corticosteroids by a clinician, initiation of a course of systemic corticosteroids by a participant, or as a hospitalization for asthma. If a participant initiates and completes a course of systemic corticosteroids without clinician involvement, this course will be counted only if the study clinician agrees the treatment was warranted, and it meets the following dosage: the course for prednisone, prednisolone, or methylprednisolone will be at least 20 mg daily dose for 3 of 5 consecutive days. The course for dexamethasone will be at least a 10 mg single daily dose. If a corticosteroid burst for the treatment of an asthma exacerbation is prescribed by a non-ICAC clinician, it will be counted regardless of dose.

### 3.3 Secondary Endpoint(s)/Outcome(s)

- CASI during the treatment period
- 2. Quality of life, as measured by physician-patient global assessment
- 3. Lung function as assessed by spirometry and IOS during the treatment period
- 4. Time to first asthma exacerbation during the treatment period
- 5. Number of reported adverse events and serious adverse events, including their severity and treatment relatedness

### 3.4 Exploratory Endpoint(s)/Outcome(s)

 Time to first respiratory virus-induced exacerbation as measured by an exacerbation associated with a respiratory virus detected using nasal mucus samples obtained at the time of an exacerbation, during the treatment period

- Number of respiratory virus-induced exacerbations as measured by an exacerbation associated with a respiratory virus detected using nasal mucus samples obtained at the time of an exacerbation, during the treatment period
- 3. Childhood ACT/ACT during the treatment period
- 4. Maximum number of asthma symptom days, defined as the highest value among the following three variables over a two-week period: number of days with wheezing, tightness in the chest, or cough; number of nights with disturbed sleep as a result of asthma; and number of days on which the participant had to slow down or discontinue play/physical activities
- 5. Bronchodilator responsiveness at the end of the treatment period
- 6. Gene expression using whole genome transcriptomics of nasal lavage samples during treatment period
- 7. Gene expression using whole genome transcriptomics of whole blood RNA samples during treatment period
- 8. Levels of antibody to mepolizumab during treatment period
- 9. Other biomarkers (banking plasma, banking nasal sample, RNA, DNA)

## 3.5 Stratification, Randomization, and Blinding/Masking

Randomization will be performed using a validated system created by the DAIT Statistical and Clinical Coordinating Center (SACCC) called RhoRAND<sup>TM</sup> that automates the random assignment of treatment groups to study ID numbers. The randomization scheme will be reviewed and approved by a statistician at the DAIT SACCC. Participants will be randomized using a 1:1 ratio of active study drug and control (placebo) participants. A covariate adaptive randomization algorithm developed by Pocock and Simon (1975)  $^{32}$  will be used to maintain a balance between treatment arms with respect to site, number of previous exacerbations (2 or 3+), peripheral blood eosinophils (< or  $\ge$ 400 cells/ $\mu$ l), BMI (< or  $\ge$ 95 th percentile for age), total serum IgE (< or  $\ge$ 540 kUA/L) and treatment dose (40 mg or 100 mg). This strategy was chosen to enhance our ability to balance the distribution of covariates that are known to be highly associated with our primary endpoint (e.g., number of previous exacerbations and peripheral blood eosinophils) as well as covariates that determine if a participant fits the FDA-approved dosing tables for omalizumab therapy (e.g., BMI and total serum IgE), which is related to Secondary Objective 5.

Randomization data will be kept strictly confidential, accessible only to authorized persons, until the time of unblinding. When the study has been completed, the data files verified, and the protocol deviations determined, the investigational agent codes will be broken and made available for data analysis.

The clinical site's research pharmacy will dispense the study drug as per the randomization schedule provided by RhoRAND<sup>TM</sup>. The injections will be administered by trained clinical research staff. Prior to injection, an unblinded site pharmacist will confirm the expiration date, the dose, and randomization assignment. The product will remain blinded to blinded clinical research staff and the participant.

## 3.5.1 Procedure for Unblinding/Unmasking

Unblinding must be approved by the DAIT NIAID Medical Monitor unless an immediate life threatening condition has developed and the Medical Monitor is not accessible. If unblinding is performed through RhoRAND<sup>TM</sup>, a notification will be sent to the protocol chair, the DAIT NIAID Medical Monitor, and the DAIT SACCC team of the unblinding event as soon as unblinding occurs. Otherwise, the site principal

investigator will notify the protocol chair and the DAIT SACCC team of the unblinding event on the next business day. The emergency unblinding will also be reported to the NIAID Allergy and Asthma Data and Safety Monitoring Board (DSMB).

A full account of the event will be recorded, including the date and time of the unblinding, the reason for the decision to unblind, and the name of the individual who made the decision to unblind and the names of the DAIT NIAID Medical Monitor and others who were notified. The reasons for unblinding of a participant's treatment will be included in the final clinical study report.

Unblinding the study due to an approved interim analysis, final analysis, or study termination will require written approval from the DAIT NIAID Medical Monitor.

## 4 Selection of Participants and Clinical Sites/Laboratories

## 4.1 Rationale for Study Population

The population selected for this trial is urban asthma patients aged 6-17 years with difficult-to-control, exacerbation-prone asthma and a peripheral blood eosinophil count ≥150 cells/µl. Previous DAIT NIAID-sponsored inner-city asthma clinical trials have shown that high proportions of children who meet Protocol ICAC-30 MUPPITS-2 inclusion criteria continue to experience exacerbations despite receiving guidelines-based asthma management and maximum levels of treatment with inhaled steroids.<sup>7,8</sup> Omalizumab is an effective add-on treatment, but up to 50% of children and adolescents identified with difficult-to-control, exacerbation-prone asthma may be ineligible for omalizumab due to their high weight, high (or low) total serum IgE level, or lack of aeroallergen sensitization. Given the existing shortcomings in the effectiveness of current treatments for a significant proportion of children and adolescents with asthma, a new approach for their management is needed to improve disease control and reduce morbidity, focusing on exacerbations.

### 4.2 Inclusion Criteria

- 1. Participant and/or parent guardian must be able to understand and provide informed consent and age-appropriate assent
- 2. Are male and female aged 6-17 years, inclusive at randomization
- 3. Have a primary place of residence in one of the pre-selected recruitment census tracts as outlined in the Protocol ICAC-30 Recruitment MOP
  - 3a. Participants who do not live in the pre-selected census tracts but live within the Office of Management and Budget (OMB) defined Metropolitan Statistical Area and have publicly-funded health insurance will qualify for inclusion.
- 4. Have had a diagnosis of asthma made > 1 year prior to recruitment; participants who received an asthma diagnosis by a clinician ≤ 1 year prior to recruitment must report that their respiratory symptoms were present for more than 1 year prior to recruitment
- 5. Have had at least two asthma exacerbations in the prior year (defined as a requirement for systemic corticosteroids and/or hospitalization)
- 6. At Visit 0 (Screening), have the following requirement for asthma controller medication: for participants aged 6 to 11 years, treatments with at least fluticasone 250 mcg dry powder inhaler

- (DPI) one puff twice daily or its equivalent and for participants aged 12 years and older, treatment with at least fluticasone 250 mcg plus LABA DPI one puff twice daily or its equivalent
- 7. Have peripheral blood eosinophils ≥150 cells/µl obtained at Visit 0 or via another ICAC protocol within 6 months
- 8. Are able to perform spirometry at randomization
- 9. Have documentation of current medical insurance with prescription coverage at randomization
- 10. Have had varicella or the varicella vaccination

#### 4.3 Exclusion Criteria

Individuals who meet any of the following criteria are not eligible for enrollment or randomization, if they:

- 1. Are not able or willing to give written informed consent or comply with study protocol
- 2. Have concurrent medical problems that would require systemic corticosteroids or other immunomodulators during the study
- 3. Are currently receiving immunotherapy
- 4. Are currently receiving treatment with omalizumab or have had omalizumab treatment within 6 months prior to randomization
- 5. Are currently requiring greater than fluticasone 500 mcg bid plus LABA one puff twice daily or its equivalent and/or individuals using oral corticosteroids daily or every other day for more than 14 days at the time of Visit 0 (Screening)
- 6. Are currently pregnant or lactating, or plan to become pregnant during the time of study participation. Females of child-bearing potential (post-menarche) must be abstinent or use a medically acceptable birth control method throughout the study (e.g. oral subcutaneous, mechanical, or surgical contraception)
- 7. Have a known, pre-existing clinically important lung condition other than asthma
- 8. Have a current malignancy or previous history of cancer in remission for less than 12 months prior to randomization
- 9. Have known, pre-existing, unstable liver disease
- 10. Is a current smoker
- 11. Have a known immunodeficiency disease
- 12. Have other conditions that could lead to elevated eosinophils such as hypereosinophilic syndromes, including eosinophilic granulomatosis with polyangiitis
- 13. Have a known, active parasitic infestation or undergoing treatment for a parasitic infestation. Once the participant has been successfully treated, the participant may be reevaluated.
- 14. Use of investigational drugs within 4 weeks of randomization
- 15. Have past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the study clinician, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study
- 16. Will not allow the study clinician, an asthma specialist, to manage their disease for the duration of the study or who are not willing to change their asthma medications to follow the protocol
- 17. Have a known history of allergic reaction to previous biologic therapy for asthma

18. Have had a life threatening asthma exacerbation in the last 2 years requiring intubation, mechanical ventilation or resulting in a hypoxic seizure

## 5 Known and Potential Risks and Benefits to Participants

## 5.1 Risks of Investigational Product or Intervention as Cited in GSK Investigator's Brochure for mepolizumab

Hypersensitivity reactions (e.g., anaphylaxis, angioedema, bronchospasm, hypotension, urticaria, rash) have occurred following administration of mepolizumab. These reactions generally occur within hours of administration, but in some instances can have a delayed onset (i.e., days).

In controlled clinical trials, 2 serious adverse reactions of herpes zoster occurred in participants treated with mepolizumab compared with none in placebo. Varicella vaccination or history of varicella is required prior to randomization.

Very common adverse reactions in subjects with severe eosinophilic asthma (incidence greater than or equal 10%) include headache and subcutaneous injection site reaction (such as pain, erythema, swelling, itching or burning sensation). Per the current IB for mepolizumab, the common adverse events are back pain, nasopharyngitis, urinary tract infection, nasal congestion, eczema, and abdominal pain upper. The incidence of AEs was similar for the placebo group as compared to the mepolizumab group regardless of the route of administration (SC or IV) with the exception of a higher rate of injection site reactions with SC administration of mepolizumab (8%) compared with placebo (3%) <sup>33</sup>.

## 5.2 Risks of Investigational Product or Intervention Cited in Medical Literature

Other side effects from Nucala® <sup>10</sup> have been reported. The MENSA trial² was a randomized, double-blind, double-dummy study of 576 patients aged 12-82 years old randomized to 75-mg mepolizumab administered intravenously, 100-mg mepolizumab administered subcutaneously, and placebo. The overall frequency of adverse events was similar across the three treatment groups. The most frequently reported adverse events were nasopharyngitis (24% given mepolizumab intravenously, 17% given mepolizumab subcutaneously, 24% given placebo) and headache (24%, 20%, and 17%). The incidence of adverse events related to a study drug was 17%, 20% and 16%. The incidence of injection-site reactions was more frequent in the subcutaneous-mepolizumab group (9%) than in the intravenous-mepolizumab and placebo groups (3% in both). The incidence of serious adverse events (including asthma-related events) was 7%, 8%, and 14% <sup>2</sup>.

The DREAM study <sup>14</sup> was a multicenter, double-blind, placebo-controlled trial of 621 patients aged 12-74 years old randomized to placebo, 75 mg mepolizumab, 250 mg mepolizumab and 750 mg mepolizumab administered intravenously. The overall frequency of serious adverse events was similar across treatment groups. The most frequently reported adverse events were headache (17% given placebo, 21% given 75 mg mepolizumab, 21% given 250 mg mepolizumab, and 21% given 750 mg mepolizumab) and nasopharyngitis (15%, 22%, 22%, and 19%). The most frequently reported drug-related adverse event was infusion-related reaction (eg, non-allergic reactions), which was reported by 6% given placebo, 5% given 75 mg mepolizumab, 8% given 250 mg mepolizumab, and 12% given 750 mg mepolizumab. Hypersensitivity deemed to be possibly related to investigational product was reported by 2% given placebo, none given 75 mg mepolizumab, <1% given 250 mg mepolizumab, and 1% given 750 mg mepolizumab <sup>14</sup>.

## 5.3 Risks of Other Protocol Specified Medications

### 5.3.1 Oral Corticosteroids

Oral prednisone will be dispensed to each participant at the beginning of the study for treatment of asthma exacerbations as per the participant's Asthma Action Plan (see Section 7.1.1.4). Oral corticosteroids can cause hoarseness, sore throat, and yeast infection of the mouth or throat if taken in high doses for lengthy periods of time. In addition, they can cause weight gain, growth delay, bruising of the skin, cataracts, and glucose intolerance. These effects are more likely if the medicine is taken at very high doses for extended periods of time. These side effects are not anticipated in this study because of the length of time (4 days on any occasion) that oral corticosteroids will be taken.

## **5.4 Risks of Study Procedures**

#### 5.4.1 Allergy Skin Testing

Allergy skin testing is routinely performed in the management of asthma and allergic diseases. Skin testing will be completed by clinical research staff trained and certified to perform the procedure in accordance with the Protocol ICAC-30 MOP to maximize safety. If a participant is allergic to any of the allergens, redness, swelling, and itching of the skin may occur and last for 1 to 2 hours. These symptoms could occur up to 1 or 2 days after the skin test. A study clinician may provide a topical corticosteroid or oral antihistamine to treat these symptoms. There is also a very rare chance that the participant may have asthma symptoms or faint during the test. A medical provider trained in treating anaphylaxis will be available to provide immediate treatment in the event that a participant experiences a systemic allergic reaction. Stopping antihistamines before skin testing may make allergy (but not asthma) symptoms worse. Participants will be told they can take their medications if they need them, but the test will need to be rescheduled.

To date, aeroallergen skin prick test procedures, conducted according to our MOP by trained and certified clinical research staff on thousands of children, have NEVER resulted in a systemic adverse reaction. Further, performance of such allergen evaluation is consistent with national asthma guidelines and provides direct benefits to both children and their families/caretakers. The results of the skin tests are provided to families, as well as relevant educational materials for environmental control.

## 5.4.2 Blood Collection

The risks associated with a blood draw include possible pain from the stick, as well as bleeding, bruising, and infection of the skin. Lightheadedness and fainting rarely occur. To minimize these risks, a clinical staff member who is trained to draw blood from children will collect the samples. Additionally, clinical staff may apply a topical anesthetic to the skin before the blood draw to reduce the discomfort of the stick. Side effects from topical anesthetics include erythema, burning, paleness at the skin site, edema, and alterations in temperature. Reactions are mild and transient. There is a potential for cutaneous allergic reactions to topical anesthetics. Topical anesthetics are routinely used for usual care venipunctures to minimize discomfort. The amount of blood to be collected is within the NIH pediatric guidelines.

## 5.4.3 Pulmonary Function Testing (Spirometry and Impulse Oscillometry)

Pulmonary function measurements will be performed by trained and certified clinical research staff according to American Thoracic Society standards as performed routinely in usual care as part of subspecialist management of asthma.

Pulmonary function tests can cause coughing or lightheadedness, which will go away shortly after the test is finished.

Participants may be asked to withhold their asthma medications for 8-24 hours before the procedures depending on the medication. Withholding of asthma medications before testing may cause a worsening of asthma symptoms. These medications and withholding instructions are specified in the Protocol ICAC-30 MOP. Participants will be informed that they can take their asthma medications if needed. If participants do take their medications, the procedure will only be rescheduled as described in the Protocol ICAC-30 MOP.

The albuterol that is given during reversibility testing can cause increased heart rate and blood pressure, nausea, headache, and a jittery or nervous feeling. These symptoms usually resolve in less than an hour.

#### 5.4.4 Exhaled Nitric Oxide Measurement

Trained and certified clinical research staff will measure exhaled nitric oxide. This test is minimal risk and well tolerated. Rarely, dizziness may occur, which goes away as soon as the test is finished.

## 5.4.5 Nasal Sample Collection

Trained and certified clinical research staff will obtain nasal mucus and nasal lavage samples from participants according to the Protocol ICAC-30 MOP. There are no known risks to collecting a nasal mucus sample.

If a participant is unable to come to a cold visit (Section 8.11) or an exacerbation visit (Section 8.12), he/she will be asked to collect a nasal swab sample at home. The nasal swab collection may cause localized discomfort. Rarely, mild epistaxis may occur. There is a risk of irritation if the liquid reagent in the nasal swab collection tube comes in contact with the skin. It is unknown whether the collection of the nasal swabs will increase the risk of infection to household members. Because we do not know if there is an increased risk of infection transmission, the study will provide gloves and masks for each participant as a protection to those assisting with nasal swab collection at home.

Nasal lavage may be associated with some transient discomfort due to the <10 second breath hold and the feeling of fluid in the nares. A very rare potential complication of nasal lavage is acute bacterial sinusitis (sinus infection). The nasal lavage procedure is considered minimal risk, and is often referred to as a nasal wash or nasal irrigation. A variety of over-the-counter products (such as the neti-pot filled with a saline solution) have been widely available for home use to safely flush out nasal passages and alleviate both nasal congestion and even sinusitis symptoms. In fact, the American Academy of Otolaryngology-Head and Neck Surgery Foundation has just issued new national guidelines recommending home irrigation of the nose with such saline solutions (as an alternative to antibiotic use), due to its ability to thin the mucus in the nose, promote drainage, and reduce inflammation as an effective intervention for both acute and chronic sinusitis. We are proposing to conduct this minimal risk procedure in the clinic, but to save and process this nasal drainage for analysis.

The study clinician may use their discretion as to whether to administer a nasal decongestant prior to the nasal collections. The nasal decongestant may be associated with temporary discomfort such as burning, stinging, sneezing, or an increase in nasal discharge.

The nasosorption procedure may produce mild discomfort such as a tickle and/or tearing of the eyes. If a participant is unable to come to a cold visit (Section 8.11) or an exacerbation visit (Section 8.12), he/she will be asked to perform the nasosorption procedure at home. It is unknown whether the nasosorption procedure will increase the risk of infection to household members. Because we do not know if there is an increased risk of infection transmission, the study will provide gloves and masks for each participant as a protection to those assisting with the nasosorption procedure at home.

## 5.4.6 Sputum Induction

Sputum induction may result in wheezing, coughing or chest tightness. Participants will be premedicated with albuterol to minimize this risk.

## 5.4.7 Nasal Epithelial Cell Collection

The risks associated with the nasal cell collection procedure include discomfort or pain, transient nosebleed, sneezing, tearing of the eyes, runny nose, and postnasal drip.

#### 5.4.8 Questionnaires

There is a possibility that participants and caretakers may find the questions too personal. Participants and caretakers may refuse to answer any questions that make them feel uncomfortable.

## 5.5 Potential Benefits

Whereas the participant's asthma may or may not improve while in this study, participants may directly benefit from study participation by receiving study-based asthma assessments and care from an asthma specialist. Participants will receive information about their spirometry and allergy skin testing and relevant asthma education consistent with recommendations in the national asthma guidelines for patients with asthma. Furthermore, these participants will receive close monitoring and direct management of asthma exacerbations on a 24/7 basis throughout the study. Participant families will receive contact numbers for the study site and a tailored asthma action plan and education. A supply of prednisone will be provided in concert with this management.

## 6 Investigational Agent

### 6.1 Investigational Agent: Mepolizumab

Mepolizumab (SB-240563) is the investigational agent and will be provided to the clinical research sites by the IND Sponsor (DAIT NIAID). Mepolizumab will be obtained by the IND Sponsor free of charge from the manufacturer (The Glaxo-Smith Kline Research and Development Ltd., Brentford, Middlesex, UK).

## 6.1.1 Formulation, Packaging, and Labeling

Mepolizumab is a humanized monoclonal antibody (IgG1, kappa) that blocks interleukin-5 (IL-5) from binding to the IL-5 receptor complex expressed on the eosinophil cell surface and thus inhibits signaling, resulting in the reduction in production and survival of eosinophils.

Mepolizumab for injection (100 mg/vial) is supplied as a sterile, white to off-white, preservative-free, lyophilized powder. Mepolizumab is presented in a 10 mL Type I clear glass, stoppered, single-use vial. The drug product must be stored in a refrigerator at a temperature of 2°C to 8°C (36°F to 46°F), protected from light.

## 6.1.2 Dosage, Preparation, and Administration

Mepolizumab is licensed for add-on maintenance treatment for severe eosinophilic asthma at a dose of 100 mg every 4 weeks and is available as a powder for solution for subcutaneous (SC) injection. In the United States, the approved dose of Nucala® for children age 12 years and above is 100 mg administered once every 4 weeks by subcutaneous injection into the upper arm, thigh, or abdomen <sup>34</sup>. For children between 6 and 11 years of age, the approved dose is 40 mg every 4 weeks.

Mepolizumab for injection (100 mg/vial) is reconstituted in the vial with 1.2 mL Sterile Water for Injection, USP, preferably using a 2- or 3-mL syringe and a 21-G needle. The reconstituted solution will contain a concentration of approximately 100 mg/mL mepolizumab. Participants assigned to the 100 mg treatment group will receive 1.0 mL of reconstituted mepolizumab. Participants assigned to the 40 mg treatment group will receive 0.4 mL of reconstituted mepolizumab.

The reconstituted solution should be kept at refrigerated or controlled room temperature (up to 25°C). It should be used as soon as possible and any unused solution remaining after 8 hours should be discarded. Complete reconstitution instructions are available in the GSK Investigator's Brochure for mepolizumab.

#### 6.2 Placebo

Placebo for mepolizumab will be 0.9% sodium chloride (normal saline) for injection. Supplies of normal saline for injection will be obtained locally by the clinical site research pharmacists.

## 6.3 Drug Accountability

Under Title 21 of the Code of Federal Regulations (21CFR §312.62), the investigator will maintain adequate records of the disposition of the investigational agent, including the date and quantity of the drug received, to whom the drug was dispensed (participant-by-participant accounting), and a detailed accounting of any drug accidentally or deliberately destroyed.

Records for receipt, storage, use, and disposition will be maintained by the study site. A drug-dispensing log will be kept current for each participant. This log will contain the identification of each participant and the date and quantity of drug dispensed.

All remaining unused investigational product will be returned to the sponsor (DAIT, NIAID) or sponsor's representative after study termination, or destroyed with the permission of the sponsor in accordance with applicable law and study site procedures. If investigational product is to be destroyed locally, the investigator will provide documentation in accordance with sponsor's specifications.

All records regarding disposition of the investigational product will be available for inspection by the clinical trial monitor.

## 6.4 Assessment of Participant Compliance with Investigational Agent

As participants will receive their mepolizumab/placebo injections in the clinic, compliance will be monitored by assessing the number of completed and missed clinic visits.

## **6.5 Toxicity Prevention and Management**

Mepolizumab/placebo doses will not be modified. Protocol Section 8.5 describes safety measures to monitor potential signs and symptoms post injection.

## 6.6 Premature Discontinuation of Study Participation

Study participation may be prematurely discontinued for any participant for any of the reasons identified in Section 11.2 Participant Stopping Rules and Withdrawal Criteria. Participants who are prematurely discontinued will follow end of study procedures as described in Section 11.4 Follow-up After Early Study Withdrawal.

Study participation may also be prematurely discontinued for any participant if the study clinician believes that the study treatment is no longer in the best interest of the participant.

## 6.7 Premature Discontinuation of Investigational Product

Participants who are discontinued from investigational product for any reason after receiving at least one injection, and who agree to remain in the study, will have an altered visit schedule. These participants will be seen in clinic every 3 months for asthma management and evaluation of protocol defined outcomes and endpoints (i.e. Visits 3, 4, 7, 10, 13 and 14 and cold and exacerbation visits). The participants will not attend the monthly protocol defined injection visits which do not involve outcome evaluation and asthma management. These participants will not receive any injections of the investigational product during the visits they do attend. During the visits the participant attends, they will undergo all other scheduled procedures, evaluations, and blood draws.

## 7 Other Medications

#### 7.1 Concomitant Medications

## 7.1.1 Protocol-mandated

All participants will receive asthma step care according to the Guidelines for the Diagnosis and Management of Asthma (Expert Panel Report 3 [EPR-3], National Asthma Education and Prevention Program [NAEPP], 2007). Treatment will be supervised by a study clinician. The study clinician will prescribe initial appropriate concomitant asthma therapies (see Section 7.1.1.1) and will provide a written Asthma Action Plan for the participant at Visits 0, 1, 4, 7, 10 and 13 (see Section 7.1.1.4). The regimen will then be adjusted as necessary at those visits throughout the duration of the trial based on the principles of the EPR-3 guidelines (see Table 7.1.1.2a, below).

The study clinician will prescribe the appropriate step controller therapy according to the participant's insurance/health maintenance organization guidelines. The preferred controller steps and alternate equivalent medications may be modified or updated based on changes in standard clinical practice, discontinuation of current medications, or the introduction of new medications. For the standardized treatment of asthma exacerbations, the clinical research staff will provide oral prednisone and written instructions for use. Montelukast may be prescribed by study clinicians if the participant was already

taking the medication prior to study enrollment. Montelukast will not affect the algorithm for prescribing asthma treatment.

All participants are required to have medical insurance at randomization that will cover, at least in part, the costs of their asthma medications. It is likely, however, that some participants may lose this coverage during the time that they are in the study. To maintain participant safety and avoid a loss of these participants to the study, Protocol ICAC-30 MUPPITS-2 will fund the cost of these participants' asthma medications during the remainder of the study or until the participant regains insurance coverage during the study. Medications will be prescribed in the same manner using the same algorithms as all insured participants. Each research site will develop plans to use local pharmacies in a cost efficient and timely manner. This design is in place to mimic the support typical insured participants receive, i.e. they receive a prescription and have to fill it at a pharmacy. To limit the time that Protocol ICAC-30 MUPPITS-2 is required to fund the cost of asthma medications for a participant who has lost coverage, each research site will develop a plan for evaluation of insurance options and referral to appropriate support systems to obtain coverage for medication costs. In addition to addressing potential insurance from employers and governmental sources, this may include free clinics and support programs available through pharmaceutical firms.

## 7.1.1.1 Initial Regimen

During Visit 0, the study clinician will determine the appropriate asthma control regimen that will be prescribed for the participant. Along with the participant's medical history and physical examination results, the medication regimen is determined by the participant's symptoms, number of systemic corticosteroid bursts in the past 6 months, percent-predicted forced expiratory volume in 1 second (FEV<sub>1</sub>), and current level of asthma controller therapy.

First, the study clinician will determine the highest "control level" of the participant's morbidity across the 4 categories in Table 7.1.1.1a. For example, if the participant has 8 days with symptoms (control level 2), 1 night with symptoms (control level 1), is at 75% predicted FEV<sub>1</sub> (control level 3), and has 0 systemic steroid bursts, (control level 1), then the participant is at control level 3 because that is the highest of these 4 categories.

Table 7.1.1.1a Asthma Symptoms for Determining Run-in Asthma Medication Regimen

| Control Level | Maximum of 1) # days<br>with asthma<br>symptoms/ two weeks<br>and 2) # days with<br>rescue albuterol or<br>levalbuterol use/ two<br>weeks* | Maximum of 1) # nights of sleep disruption due to asthma/ 2 weeks and 2) # nights use of albuterol or levalbuterol for awakening / 2 weeks* | FEV <sub>1</sub><br>(% pred)** | Courses of<br>systemic steroids<br>in the last 6<br>months*** |
|---|---|---|---|---|
| 1 | 0-3 days | 0-1 night | ≥ 85 | 0 |
| 2 | 4-9 days | 2 nights | 80 - < 85 | 1 |
| 3 | 10-13 days | 3-4 nights | 70 - < 80 | 2 |
| 4 | 14 days | 5-14 nights | < 70 | >2 |

 $FEV_1$  = forced expiratory volume in 1 second; pred = predicted

\* Determined from participant recall, based on the 2-week interval directly preceding the study visit.

\*\*Predicted references are provided in the Protocol ICAC-30 MOP.

\*\*\* Defined as a prescription of a course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant to prevent a serious asthma outcome. If a participant initiates and completes a course of systemic steroids without clinician involvement, this course will be counted only if it meets the following dosage: the course for prednisone, prednisolone, or methylprednisolone will be at least 20 mg daily dose for 3 of 5 consecutive days. The course for dexamethasone will be at least a 10 mg single daily dose. If a corticosteroid burst for the treatment of an asthma exacerbation is prescribed by a non-ICAC clinician, it will be counted regardless of dose.

Next, the study clinician will determine the current level of controller therapy that the participant is using. Table 7.1.1.1b shows the asthma regimens that will be used during the treatment phase of Protocol ICAC-30 MUPPITS-2. If the participant is currently on one of the therapies below, then the step level of that therapy will be noted. Otherwise, the study clinician must refer to the Protocol ICAC-30 MOP for equivalency tables for other asthma therapies. From the information in the Protocol ICAC-30 MOP, the study clinician will determine the corresponding step level of therapy that the participant is currently using. For example, if the participant is currently taking Flovent® Diskus® 250 mcg twice per day (bid), then he/she is receiving Step 3 therapy.

Table 7.1.1.1b Asthma Regimen by Step Level of Therapy

| Step | Medication Equivalent* |
|------|---------------------------------------------------------|
| 0 | No controller medication; albuterol or levalbuterol prn |
| 1 | fluticasone 50 mcg bid |
| 2 | fluticasone 100 mcg bid |
| 3 | fluticasone 250 mcg bid |
| 4 | fluticasone 250 mcg bid plus LABA |
| 5 | fluticasone 500 mcg bid plus LABA |

bid = twice per day; LABA = long-acting beta agonist

Based on the participant's current control level (from Table 7.1.1.1a) and the participant's current step level of therapy (from Table 7.1.1.1b and the Protocol ICAC-30 MOP), the study clinician will find the corresponding row in Table 7.1.1.1c below that includes both the current regimen and the current control level. The last column of that row gives the corresponding regimen as a step level, which refers back to Table 7.1.1.1b. The study clinician will prescribe this regimen. Study eligibility in terms of treatment step level will be as follows:

- For participants ages 6 to 11 years, who have a requirement for at least Step Level 3 (defined in Table 7.1.1.1b) at Visit 0
- For participants ages 12 years and older, who have a requirement for at least Step Level 4 (defined in Table 7.1.1.1b) at Visit 0

<sup>\*</sup>Equivalent medication covered by participant's insurance formulary – see Protocol ICAC-30 MOP.

Continuing the example from above, since the participant is taking Step 3 therapy and is at control level 3, the regimen assigned would be Step 4 (fluticasone 250 mcg bid with LABA from Table 5.2b).

Table 7.1.1.1c Algorithm for Prescribing Treatment Regimen at Visit 0

| Current Regimen | <b>Current Control Level</b> | Regimen Assigned |
|---|---|---|
| Regimen equivalent to Step 0<br>(or 1-3 days/week of a regimen<br>equivalent to Step 1) | Control level 1<br>Control level 2<br>Control level 3<br>Control level 4 | Step 2<br>Step 2<br>Step 2<br>Step 2 (and may also need prednisone<br>burst) |
| Regimen equivalent to Step 1<br>(or 1-3 days/week of a regimen<br>equivalent to Step 2) | Control level 1<br>Control level 2<br>Control level 3<br>Control level 4 | Step 2 Step 2 Step 2 Step 2 Step 3 (and may also need prednisone burst) |
| Regimen equivalent to Step 2<br>(or 1-3 days/week of a regimen<br>equivalent to Step 3) | Control level 1<br>Control level 2<br>Control level 3<br>Control level 4 | Step 2 Step 3 Step 3 Step 3 Step 4 (and may also need prednisone burst) |
| Regimen equivalent to Step 3<br>(or 1-3 days/week of a regimen<br>equivalent to Step 4) | Control level 1<br>Control level 2<br>Control level 3<br>Control level 4 | Step 3 Step 4 Step 4 Step 4 Step 5 (and may also need prednisone burst) |
| Regimen equivalent to Step 4 (or 1-3 days/week of a regimen equivalent to Step 5) | Control level 1<br>Control level 2<br>Control level 3<br>Control level 4 | Step 4 Step 5 Step 5 Step 5 Step 5 (and may also need prednisone burst) |
| Regimen equivalent to Step 5 | Control level 1<br>Control level 2<br>Control level 3<br>Control level 4 | Step 5 Step 5 Step 5 Step 5 (and may also need prednisone burst) Step 5 (and may also need prednisone burst) |

Note: Shading in the table corresponds to the example described in the text.

In addition to the controller regimen assigned above, all participants will be prescribed albuterol by metered-dose inhaler beta-agonist or nebulizer (per clinician discretion) to be used as needed and will be provided oral prednisone to be used as per protocol – see Section 7.4 and the Protocol ICAC-30 MOP. The study clinician will prescribe enough medication to last until the next E&M visit. If a participant is not eligible to continue, the study clinician may prescribe an appropriate treatment regimen based on clinical judgment.

## 7.1.1.2 Study Period Treatment Regimen (Visits 1, 4, 7, 10 and 13)

At Visits 1, 4, 7, 10 and 13 participants' asthma medication regimen will be adjusted based on symptoms, albuterol/levalbuterol use,  $FEV_1$ , recent exacerbations, and their current level of therapy.

Except at Visit 1, participants will be stepped down from controller medications at each visit for which their control level is equal to 1. At Visit 1, it is not appropriate to step down a participant's treatment

after 4 weeks of observation during the assumption care. As such, participants will not be stepped down at Visit 1. At Visit 1, a participant may be stepped up as per the protocol algorithm.

Participants will undergo pre-bronchodilator spirometry and an assessment of symptoms, rescue bronchodilator usage, recent exacerbations and medication adherence. Bronchodilator use as a preventive measure prior to exercise will not count toward the assessment of rescue bronchodilator use. Based on these data, a study clinician will determine the participant's current control level from Table 7.1.1.2a below. The control levels originated from the published national guidelines, Guidelines for the Diagnosis and Management of Asthma (EPR-3, NAEPP, 2007).

For all participants, the highest control level for days with symptoms or albuterol/levalbuterol use, nights with symptoms or albuterol/levalbuterol use, percent personal best FEV<sub>1</sub>, and exacerbation history will be determined by the study clinician. The day and night symptoms, albuterol/levalbuterol use, adherence to prescribed asthma controller medications by self-report, and exacerbation history will be determined from questionnaires. The FEV<sub>1</sub> personal best is defined in the Protocol ICAC-30 MOP. If the quality of the spirometry maneuver at the current visit is unacceptable according to the technician's judgment, FEV<sub>1</sub> in Table 7.1.1.2a will not be used, and the control level will be based on day and night symptoms, albuterol/levalbuterol use, and exacerbation history. For example, if a participant has 0 days with symptoms (control level 1), 4 nights with symptoms (control level 3), FEV<sub>1</sub> at 85% of personal best (control level 1), and 1 exacerbation (control level 2), then the participant's overall control level is 3 because that is the maximum value of control levels 1, 3, 1, and 2.

Table 7.1.1.2a Control Levels of Symptoms, Bronchodilator Usage, FEV<sub>1</sub> (% personal best), and Exacerbations

| Control<br>Level | Maximum of 1) # days with asthma symptoms/ 2 weeks and 2) # days with rescue albuterol/levalbuterol use/ 2 weeks* | Maximum of 1) # nights of sleep<br>disruption due to asthma/ 2<br>weeks and 2) # nights use of<br>albuterol/levalbuterol for<br>awakening/ 2 weeks* | FEV <sub>1</sub><br>(% personal<br>best) | Courses of Systemic Steroids since the Last Medication Management Visit** |
|---|---|---|---|---|
| 1 | 0-3 days | 0-1 night | ≥ 85 | 0 |
| 2 | 4-9 days | 2 nights | 80-84 | 1 |
| 3 | 10-13 days | 3-4 nights | 70-79 | - |
| 4 | 14 days | 5-14 nights | < 70 | - |

FEV<sub>1</sub> = forced expiratory volume in 1 second

<sup>\*</sup> Determined from participant recall, based on the 2-week interval directly preceding the study visit.

<sup>\*\*</sup>Defined as a prescription of a course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant to prevent a serious asthma outcome. If a participant initiates and completes a course of systemic steroids without clinician involvement, this course will be counted only if it meets the following dosage: the course for prednisone, prednisolone, or methylprednisolone will be at least 20 mg daily dose for 3 of 5 consecutive days. The course for dexamethasone will be at least a 10 mg single daily dose. If a corticosteroid burst for the treatment of an asthma exacerbation is prescribed by a non-ICAC clinician, it will be counted regardless of dose.

Note: Shading in the table corresponds to the example described in the text above.

Based on the overall control level and the participant's estimated level of adherence, the study clinician will use Table 7.1.1.2bb below to determine how the participant's current therapy should be modified. At E&M Visits, the participant will be considered to have acceptable adherence if he/she reports having taken 50% or more of the prescribed doses in the last 2 weeks. Participants with unacceptable adherence will not be stepped up in the same way as those with acceptable adherence. Continuing with the same example, since this participant is at control level 3 and assuming he/she has acceptable adherence, the study clinician would recommend a 2-step increase in therapy (or an increase to Step 5 if on Step 4 or maintenance on Step 5 if already on Step 5). In all cases, consideration will be given to a burst of prednisone according to the suggestions in the table.

Table 7.1.1.2b Treatment Adjustment Based on Control Levels and Adherence

Inner-City Asthma Consortium

| Control<br>Level | Treatment Algorithm for Participants with Unacceptable Adherence | Treatment Algorithm for Participants with Acceptable Adherence |
|---|---|---|
| 1 | Continue same controller regimen | If on Step 0, maintain at Step 0 If on Steps 1-5, decrease controller regimen by 1 step ** Do not decrease controller regimen if at Visit 1 |
| 2 | Continue same controller regimen or place on Step 2 therapy, whichever is higher | Increase controller regimen by 1 step, or continue Step 5 therapy if already on Step 5 |
| 3 | Continue same controller regimen or place on Step 2 therapy, whichever is higher | No systemic steroids since the Last Medication Management visit* If on Steps 0-4 increase controller regimen by 1 step If on Step 5 continue Step 5 or treat with Step 5 and a 4 day burst of prednisone or equivalent; ≥1 course(s) of systemic steroids since the last E&M visit* If on steps 0-3 increase controller regimen by 2 steps If on treatment Step 4 increase controller regimen to Step 5 or treat with Step 5 and a 4 day burst of prednisone or equivalent If on treatment Step 5 continue Step 5 or treat with Step 5 and a 4 day burst of prednisone or equivalent |
| 4 | Continue same controller regimen or place on Step 3 therapy, whichever is higher OR Treat with 4-day prednisone burst and continue same controller regimen or place on Step 3 therapy, whichever is higher | If on Steps 0-3 increase controller regimen by 2 steps If on Step 4, increase to Step 5 <b>or</b> treat with Step 5 <u>and</u> a 4-day prednisone burst or equivalent If already on Step 5, continue on Step 5 <b>or</b> treat with Step 5 <u>and</u> a 4-day burst of prednisone or equivalent |

<sup>\*</sup>Defined as a prescription of a course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant to prevent a serious asthma outcome. If a participant initiates and completes a course of systemic steroids without clinician involvement, this course will be counted only if it meets the following dosage: the course for prednisone, prednisolone, or methylprednisolone will be at least 20 mg daily dose for 3 of 5 consecutive days. The course for dexamethasone will be at least a 10 mg single daily dose. If a corticosteroid burst for the treatment of an asthma exacerbation is prescribed by a non-ICAC clinician, it will be counted regardless of dose. Note: Shading in the table corresponds to the example described in the text above.

Based on the participant's step level assigned at the last E&M visit and the change in steps determined above, the new regimen will be prescribed according to Table 7.1.1.2b above. In the example above, if
the participant were currently on Step 2 and having no problems with adherence, then the recommended new treatment step based on symptoms, albuterol/levalbuterol use, FEV<sub>1</sub>, and exacerbations is Step 4.

#### 7.1.1.3 Final Study Visit

At the final study visit (Visit 14), the final treatment regimen prescribed will be based on the protocol-based medications management algorithm or the discretion of the study clinician who examines the participant. He/she will base the treatment on factors such as symptoms, albuterol use, spirometry, adherence, and the participant's current level of therapy; however, the participant's treatment will not be stepped down at Visit 14. The participant's care will then be transferred back to their primary care provider (PCP) and/or asthma specialist.

#### 7.1.1.4 Asthma Action Plan

Clinical research staff will provide a written Asthma Action Plan consistent with NAEPP guidelines for the participant at Visits 0, 1, 4, 7, 10, 13, and 14. This plan describes a Green, Yellow, and Red Zone for the participant based on his/her symptoms. In the Green Zone, the participant has no symptoms of an asthma episode and is directed to use his/her usual asthma medications. In the Yellow Zone, the participant is experiencing asthma, allergy, or cold symptoms, and is directed to increase rescue medication use until the symptoms have been resolved. In the Red Zone, the participant is having persistent symptoms that cannot be controlled. The participant is instructed to contact a study clinician OR go to the emergency department (ED) if unable to contact a study clinician.

#### 7.1.1.5 Asthma Education

As part of the meeting at Visits 0, 1, 4, 7, 10, 13, and 14 with a clinical research staff member for asthma education, participants will be educated on topics related to asthma. These topics include background on asthma as a disease, use of the Asthma Action Plan (see Section 5.5), adherence to medications, using medications at school (when applicable), and allergen and irritant avoidance. Handouts will be provided and the education content will be tailored to each participant. For example, the allergen avoidance education will be based on the participant's aeroallergen skin test/serum IgE results. The participant will receive education about the allergens to which he/she is sensitive. The information contained in the handouts will be based on the EPR-3: Guidelines for the Diagnosis and Management of Asthma and on experience from previous ICAC clinical trials. The involvement of the caretaker in these sessions depends on the age and maturity of the participant.

## 7.1.2 Other permitted concomitant medications

During the study, maintenance medications, aside from those excluded in Section 4.3, Exclusion Criteria, will be permitted.

#### 7.2 Prophylactic Medications

Not applicable.

#### 7.3 Prohibited Medications

- 1. Allergen immunotherapy (sublingual or subcutaneous)
- 2. Anti-IgE therapy
- 3. Any investigational drug
- 4. Additional medications listed in the Protocol ICAC-30 MUPPITS-2 MOP

#### 7.4 Rescue Medications

Inner-City Asthma Consortium

Use of albuterol by participants and study clinicians will be guided by each participant's Asthma Action Plan (see Section 7.1.1.4), which will be updated and provided at Visits 0, 1, 4, 7, 10 and 13. To achieve as much uniformity in approach as possible across clinical sites, these plans will be pre-printed with specific albuterol dosing for the Yellow and Red zones.

## **Definition and Management of Acute Exacerbations**

Consistent with NAEPP 2007 guidelines, study clinicians caring for participants in the Protocol ICAC-30 MUPPITS-2 study will start a course of corticosteroids for severe and/or unresponsive exacerbations of asthma. For the purposes of the proposed analyses, an asthma exacerbation is defined as a prescription of a course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant or a hospitalization to prevent a serious asthma outcome. If a participant initiates and completes a course of systemic steroids without clinician involvement, this course will be counted only if the study clinician agrees the treatment was warranted and it meets the following dosage: the course for prednisone, prednisolone, or methylprednisolone will be at least 20mg daily for 3 of 5 consecutive days. The course for dexamethasone will be at least a 10 mg single daily dose. Study clinicians will strongly consider initiation of corticosteroids if:

- Albuterol is needed by inhaler (with or without a spacer) or by nebulization for more than 6 individual treatments in 24 hours; or
- Moderate-severe wheeze, cough, shortness of breath, and/or chest tightness or pain occurs for at least 5 of the preceding 7 days; or
- Symptoms of wheeze, cough, shortness of breath, and/or chest tightness or pain severe enough to place a participant in his or her "Red Zone" on their Asthma Action Plan (see Section 7.1.1.4) do not significantly improve after 3 doses of albuterol. (In such situations, in addition to the initiation of oral corticosteroids, the study clinician should consider directing the participant to the nearest ED.); or
- There is an unscheduled visit for acute asthma care requiring repeated doses of albuterol (clinician office, urgent care, ED); or
- Hospitalization is needed for asthma.

Permissible drugs for systemic corticosteroid treatment of asthma exacerbations include: prednisone, prednisolone, methylprednisolone, and dexamethasone. The course for prednisone, prednisolone, or methylprednisolone will be 2 mg/kg/day as a single daily dose for 4 days with a maximum dose of 60 mg per day. The course for dexamethasone will be 0.3 to 0.6 mg/kg/day as a single daily dose for 2 days with a maximum dose of 16 mg per day. Failure to respond to initial treatment will result in additional evaluation and possible hospitalization for further management. This management approach has been applied to previous ICAC clinical trials and is consistent with asthma specialist usual care practices.

## 8 Study Procedures

## 8.1 Study Procedures

#### 8.1.1 Vital Signs and Growth Parameters

Height (using a calibrated stadiometer) will be measured at clinic visits as part of spirometry. Respiratory rate and temperature, along with a chest auscultation will be obtained at clinic visits as part of the targeted pulmonary exam.

The following vital signs and growth parameters will be collected at asthma evaluation and management visits (Visits 0, 1, 4, 7, 10, 13 and 14) unless otherwise noted:

- Weight in kilograms
- Pulse rate
- Blood pressure

#### 8.1.2 Medical History and Physical Examination

The participant's medical history will be obtained, and a study clinician will perform a physical examination at Visit 0. The study clinician will perform a targeted pulmonary examination and current asthma symptom assessment at the other evaluation and management study visits. Additional examinations may be completed at the remainder of the visits at the study clinician's discretion.

Significant findings that are present prior to the start of the study must be included on the appropriate case report form (CRF). Significant findings that meet the definition of an adverse event (AE) must also be recorded on the AE form.

If the participant is currently having an asthma exacerbation or other symptoms that the study nurse or study clinician feel may compromise the participant's ability to complete the study procedures safely, a physical exam may be performed and the study visit may be rescheduled. If the study clinician observes any AEs during the study visit, a targeted physical exam may be performed. Additional details regarding AE assessment are outlined in Section 12, Safety Monitoring and Reporting.

#### 8.1.3 Aeroallergen Skin Testing

The participant's atopic status will be assessed with skin prick tests to assess allergy to dust mites, cockroaches and various other aeroallergens. The allergens chosen include those that are likely to cause sensitization in people living in urban environments. Participants will be asked to stop taking antihistamines for 5 days prior to the visit at which the skin test is performed to limit interference with the results of the skin test.

Skin testing will be done by the prick technique using the Greer Pick system (Greer; Lenoir, NC). Testing will be performed by certified clinical research staff according to the instructions in the Protocol ICAC-30 MOP. Tests will be read after 15 minutes by measuring the wheal for each antigen and for the controls.

Acceptable skin testing completed as part of a participant's participation in other ICAC protocols within 12 months will meet the requirement for this procedure. In this situation, the skin testing results documentation from the previous study will be added to the participant's study file, and the skin testing procedure will not be repeated.

The national asthma guidelines have emphasized that exposure of patients who have asthma to allergens to which they are sensitive has been shown to increase asthma symptoms and precipitate asthma exacerbations. They further state that the clinician should evaluate the potential role of

allergens, particularly indoor inhalant allergens via medical history and skin testing, and then assess the significance of positive tests in the context of the patient's medical history. Patients who have asthma at any level of severity should: reduce, if possible, exposure to allergens to which the patient is sensitized and exposed; know that effective allergen avoidance requires a comprehensive approach; and (3) be provided with relevant educational materials for control of environmental factors. For over 20 years, study clinicians with the DAIT NIAID-sponsored National Cooperative Inner-City Study (1991-1997), the DAIT NIAID-sponsored Inner-City Asthma Study (1994-2001), the DAIT NIAID-sponsored Inner-City Asthma Consoritium1 (ICAC1) (2002-2009), ICAC2 (2009-2014), and now ICAC3 as of 2015, have applied the recommendations from the asthma guidelines as best practices and "usual care" for children with asthma, especially as relevant to children residing in our inner-cities. These asthma specialists believe that participants and their families who enroll in our studies can receive direct benefit from the conduct of environmental histories, aeroallergen skin tests, and provision of education about personal allergen triggers and measures to avoid them. Seminal publications from the first study in 1997 reported that the enrolled study children who were both allergic to cockroach allergen and highly exposed had significantly higher rates of asthma hospitalization and asthma morbidity. Subsequent research has confirmed these observations and extended our knowledge on the extent of allergen sensitization in the inner-city environment, risks to these children, and successful interventions to mitigate these risks. For example, in the Protocol ICAC-07 Urban Environment and Childhood Asthma birth cohort study (URECA), children were aeroallergen skin prick tested as per the procedures we describe for Protocol ICAC-30 MUPPITS-2. By age 3, 44% of the Protocol ICAC-07 URECA cohort (n=418) were sensitized, primarily to cockroach, mouse, dog, dust mite, and cat. There were statistically significant odds ratios of the relationship between allergic sensitization and recurrent wheeze. Each of the ICAC1, ICAC2, and now ICAC3 trials have incorporated aeroallergen skin prick testing procedures as an evaluation that provides direct value to both children and their families. Feedback from parents and caretakers consistently confirm this value. These standardized procedures, performed by trained and certified clinical research staff, have now been safely performed in thousands of participating children in all inner-city studies with no reports of systemic adverse events.

#### 8.1.4 Measurement of Fractional Exhaled Nitric Oxide

Measurement of FeNO will be obtained (if location of visit allows) prior to spirometry. Exhaled nitric oxide will be measured following American Thoracic Society guidelines for FeNO assessment.<sup>27</sup> This procedure is detailed in the Protocol ICAC-30 MOP.

#### 8.1.5 Measurement of Pulmonary Function

Spirometry and impulse oscillation spirometry will be conducted following the ATS and European Respiratory Society guidelines. For children under 8 years of age, ATS Preschool Guidelines will be used for spirometry acceptance evaluation. This procedure has been successfully implemented in previous DAIT NIAID-sponsored ICAC trials. Details regarding pulmonary function testing (PFT) are provided in the Protocol ICAC-30 MOP. All PFTs will be performed by certified clinical research staff.

Participants may be asked to stop taking some asthma medications 8-24 hours before the visit (depending on the type of medication) to limit their interference with the results of the pulmonary function testing. These medications and withholding instructions are specified in the Protocol ICAC-30 MOP.

#### 8.1.6 Questionnaire Assessments

Questionnaires administered by site staff will collect inclusion/exclusion criteria information, participant contact information, demographic characteristics, asthma and allergy history and medication use, asthma exacerbation history, asthma symptoms and health care utilization, cold symptoms, concomitant medications, AE information, and primary care provider (PCP) contact information.

#### 8.2 Clinical and Research Laboratory Evaluations and Specimen Collection

## 8.2.1 Blood Sample Collection

Blood will be collected by peripheral venipuncture for transcriptomics, to preserve DNA/RNA, to assess a complete blood count (CBC) and differential and blood chemistry, as well as total and allergen-specific serum IgE. With the participant's consent, blood will be stored for use in the future for unplanned tests. Blood volume will be indicated in the informed consent document along with any possibility for a repeat blood draw, if needed. An eosinophil value obtained as part of a participant's participation in another ICAC protocol within 6 months of the screening visit will determine the requirement for Protocol ICAC-30 MUPPITS-2 eligibility.

| Table 8.2.1 CBC and Blood | Chemistry | / Components |
|---------------------------|-----------|--------------|
|---------------------------|-----------|--------------|

| CBC (and differential) | Blood Chemistry |
|------------------------|----------------------------|
| Platelets | BUN |
| Hematocrit | CO2 |
| Hemoglobin | Creatinine |
| Erythrocytes | Glucose |
| Leukocytes | Serum chloride |
| Monocytes | Serum potassium |
| Eosinophils | Serum sodium |
| Basophils | Bilirubin |
| Neutrophils | Aspartate aminotransferase |
| Lymphocytes | Alanine aminotransferase |

#### 8.2.2 Nasal Sample Collection

Nasal mucus samples will be collected as per the Protocol ICAC-30 MOP for respiratory virus/bacteria assessment. If a participant is unable to come to an exacerbation visit (Section 8.12), he/she will be asked to collect the nasal mucus sample at home. Training and supplies will be provided to the participant by the site staff.

If a participant is unable to come to a cold visit (Section 8.11) or exacerbation visit (Section 8.12), he/she will be asked to collect a nasal swab sample at home. Training and supplies will be provided to the participant by the site staff as per the Protocol ICAC-30 MOP.

As per the Protocol ICAC-30 MOP, nasal lavage samples will be collected by instilling preservative-free buffered saline into the nostrils and allowing fluid to return passively into collection specimens. If the nostrils are occluded, a nasal decongestant may be administered at the discretion of the study clinician. Samples will be split and processed for both cell differentials and RNA extraction. Site clinical research staff who are trained, study-authorized, and certified will perform the nasal lavage and processing procedure as specified in the Protocol ICAC-30 MOP.

Nasosorption is a non-invasive technique for sampling of undisturbed mucosal lining fluid from the upper airways through which quantification of in situ levels of immune mediators, such as cytokines and chemokines, will be performed. The sample will be obtained using the size-appropriate single use Nasosorption™ FX·i device (Hunt Developments, UK) consisting of a synthetic absorptive matrix strip (SAM) attached to an applicator handle. Details of the nasosorption sample collection and processing procedures are described in the Protocol ICAC-30 MOP. If a participant is unable to come to a cold visit (Section 8.11) or an exacerbation visit (Section 8.12), he/she will be asked to perform the nasosorption procedure at home. Training and supplies will be provided to the participant by the site staff.

## 8.2.3 Urine Pregnancy Testing

All females who have reached menarche will be required to have a urine pregnancy test before completing study activities. If the result is positive, the participant will not undergo any procedures. Results of all pregnancy tests will be given to the participant or caretaker as per site-specific guidelines and relevant state laws.

## 8.2.4 Urine Cotinine

Urinary cotinine (a metabolite of nicotine) will be measured to determine exposure to environmental tobacco smoke. A urine sample will be collected following procedures described in the Protocol ICAC-30 MOP. The urine sample will be stored long-term for future research in the field of asthma. Participants will be asked to give permission for long-term storage and future use during the consent process.

### 8.2.5 Induced Sputum

Sputum will be induced by inhalation of hypertonic saline solution using the method that was used in the Asthma Clinical Research Network (ACRN)<sup>35</sup>. Safety monitoring per spirometry and symptom report will be performed during and after sputum induction. Slides will be read at a central site for cellular determinations. Sputum cells will be processed for CyTOF analysis and RNA and DNA isolation for expression and epigenetic studies. Sputum supernatants will be collected, aliquoted, and stored pending further analysis. This procedure will be performed in a subset of children ≥10 years of age.

#### 8.2.6 Nasal Epithelial Cell Collection

Nasal epithelial cell samples will be obtained by using a cytology brush. A trained study clinician will conduct the procedure. The inferior turbinate of one nasal passage will be sampled to obtain an adequate number of epithelial cells for mRNA and DNA isolation. The sampled area will be observed for hemostasis. Procedural details and instructions for processing the samples are included in the Protocol ICAC-30 MOP. This procedure will be performed in a subset of children ≥10 years of age.

## 8.3 Recruitment

The research site may use any Institutional Review Board (IRB)-approved means to identify potential participants. Examples include hospital, clinic, or emergency department admission records; study clinicians' specialty clinic records; and advertising (in public locations and on the radio). Potential participants will be screened and recruited using a standardized questionnaire that collects contact information and inclusion/exclusion criteria information. Participants may be recruited by phone or in person.

Retention methods involve a number of different approaches. We will use an appointment reminder system that consists of phone calls several days and one day prior to scheduled appointments for Protocol ICAC-30 MUPPITS-2 Version 9.0 01/11/21

confirmation. To facilitate telephone contact with participants whose phone service may change during the study, up to three telephone contact numbers (relatives, neighbors, friends) will be collected for each participant. This has proven to be an effective strategy in previous DAIT NIAID-sponsored ICAC trials. Those who have no obvious characteristics making them ineligible and who are interested will be invited to the clinic for a Screening Visit.

## 8.4 Screening/Baseline Visit

This research study will be explained in lay terms to the parent/legal guardian of each potential participant. Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization will be obtained from all parents/legal guardians at the beginning of this visit and before the child undergoes any screening study procedures. Children age 12 years and older will sign a written assent form. When the informed consent has been signed, the participant is considered enrolled in the study and will be assigned a unique participant number. Study procedures will be stopped, and the participant will be deemed ineligible for the study at any point during the Screening Visit if and when he/she fails to meet eligibility criteria.

The purpose of the screening period is to confirm eligibility to continue in the study. After the consent (and assent, if applicable) is signed, participants will undergo screening study procedures as listed below:

- Vital signs (see Section 8.1.1)
- Urine collection for pregnancy test for female participants who have reached menarche (see Section 8.2.3)
- Medical history and a physical examination by study clinician (see Section 8.1.2)
- Concomitant medication assessment (see Sections 8.1.6 and 7.1)
- Questionnaires (see Section 8.1.6)
- Weight and height measurement, using a calibrated stadiometer (see Section 8.1.1)
- Spirometry (see Section 8.1.5)
- Assignment of asthma medication regimen by study clinician (see Section 7.1.1)
- Blood sample collection (see Section 8.2.1.1)
  - o CBC with differential
  - Blood chemistry
  - Total and allergen-specific IgE
- Asthma counseling (see Section 7.1.1) (not completed if participant is a screen fail)
- AE assessment (see Section 12)

Participants will also undergo skin prick tests (see Section 8.1.3) to a panel of allergens detailed in the Protocol ICAC-30 MOP to characterize the study population. Participants who have valid skin test results within the previous year under another ICAC protocol will not need to be re-tested. Clinical research staff may choose to perform the skin prick tests at Visits 2, 3, or 4 instead of Screening.

Participants may be re-screened per study clinician discretion. Participants who meet any of the following criteria are not eligible for re-screening:

- Have a known, pre-existing clinically important lung condition other than asthma
- Have known, pre-existing, unstable liver disease

- Have a known immunodeficiency disease
- Have other conditions that could lead to elevated eosinophils such as hypereosinophilic syndromes, including eosinophilic granulomatosis with polyangiitis
- Will not allow the study clinician, an asthma specialist, to manage their disease for the duration of the study or who are not willing to change their asthma medications to follow the protocol
- Have a known history of allergic reaction to previous biologic therapy for asthma

If total eosinophil counts were measured as a part of a CBC with differential in a previous ICAC protocol, total eosinophil results will be used to determine eligibility if drawn within 6 months of the Screening Visit. If values are not available from a previous ICAC protocol, total eosinophil counts obtained at Visit 0 will be used to determine eligibility. If a participant fails eligibility due to total eosinophil count only, the study clinician may choose to redraw total eosinophil counts one additional time for re-screening.

#### 8.5 Randomization

At this study visit, participants will be re-assessed to confirm they continue to meet study eligibility criteria.

The study clinician will adjust the participant's asthma medications as necessary according to the treatment algorithm (see Section 7.1.1.2), write an appropriate prescription, and provide a new asthma action plan (see Section 7.1.1.4). At Visit 1, it is not appropriate to step down a participant's treatment after 4 weeks of observation during the assumption of care. As such, participants will not be stepped down at Visit 1. At Visit 1, a participant may be stepped up as per the protocol algorithm. Participants will receive basic asthma education (see Section 7.1.1.5).

Other assessments completed at this visit include:

- Targeted pulmonary exam (see Section 8.1.2)
- Spirometry and IOS with reversibility (see Section 8.1.4),
- Exhaled nitric oxide (see Section 8.1.4)
- Urine cotinine (see Section 8.2.4)
- Urine pregnancy test, where indicated (see Section 8.2.3)
- Nasal mucus sample collection (see Section 8.2.2)
- Nasal lavage (see Section 8.2.2)
- Blood sample collection (see Section 8.2.1)
  - CBC with differential
  - Blood markers (plasma/DNA/RNA)
  - Antibody to drug
- Questionnaires (see Section 8.1.6)
- Assignment of asthma medication regimen by study clinician (see Section 7.1.1)
- Asthma education/counseling (see Section 7.1.1.5)

After they have been found eligible for randomization, participants will be randomized (see Section 13.3) and receive their first injection of mepolizumab/placebo.

Before each injection, participants will be screened for evidence of an ongoing allergic reaction or worsening of asthma. If a participant is unable to receive the study drug injection that day, the injection will be rescheduled. Injections must be at least 14 days apart.

The injection will be administered by trained clinical research staff. Clinical research staff may apply a topical anesthetic to the skin before the injection to reduce the discomfort of the stick.

During all dosing visits, a medical provider trained in treating anaphylaxis will be available to provide immediate treatment in the event that a participant experiences an allergic reaction. Participants will remain at the clinic for observation for at least 60 minutes after the first 3 injections, after which a 30 minute wait period will be required.

#### 8.6 Visit 2 (Week 8)

At this visit, the following procedures and assessments will be performed:

- Urine pregnancy test, where indicated (see Section 8.2.3)
- Vital signs (see Section 8.1.1)
- Lungs assessment
- Study drug administration
- AE assessment (see Section 12)
- Concomitant medication assessment (see Sections 8.1.6 and 7.1.2)
- Nasal mucus sample collection (see Section 8.2.2)
- Allergen skin testing (see Section 8.1.3) if not performed at a previous study visit or in another ICAC protocol within 12 months

## 8.7 Visit 3 (Week 12)

At this visit, the following procedures and assessments will be performed:

- Urine cotinine (see Section 8.2.4)
- Urine pregnancy test, where indicated (see Section 8.2.3)
- Vital signs (see Section 8.1.1)
- Lungs assessment
- Study drug administration
- AE assessment (see Section 12)
- Concomitant medication assessment (see Sections 8.1.6 and 7.1.2)
- Nasal mucus sample collection (see Section 8.2.2)
- Nasal lavage (see Section 8.2.2)
- Blood sample collection (see Section 8.2.1)
  - o CBC with differential
  - Blood chemistry
  - Blood markers (plasma/DNA/RNA)
  - Antibody to drug
- Exhaled nitric oxide (see Section 8.1.4)
- Allergen skin testing (see Section 8.1.3) if not performed at a previous study visit or in another ICAC protocol within 12 months

## 8.8 Injection Only Visits (Visits 5, 6, 8, 9, 11, 12)

At these visits, the following procedures and assessments will be performed:

- Urine pregnancy test, where indicated (see Section 8.2.3)
- Vital signs (see Section 8.1.1)
- Lungs assessment
- Study drug administration
- AE assessment (see Section 12)
- Concomitant medication assessment (see Sections 8.1.6 and 7.1.2)
- Nasal mucus sample collection (see Section 8.2.2)

#### 8.9 Asthma Evaluation and Management Visits (Visits 4, 7, 10, 13)

At these visits, the following procedures and assessments will be performed:

- Urine pregnancy test, where indicated (see Section 8.2.3)
- Study drug administration
- AE assessment (see Section 12)
- Concomitant medication assessment (see Sections 8.1.6 and 7.1.2)
- Questionnaires (see Section 8.1.6)
- Vital signs (see Section 8.1.1)
- Spirometry (see Section 8.1.5)
- Nasal mucus sample collection (see Section 8.2.2)
- Targeted pulmonary examination by study clinician (see Section 8.1.2)
- Assignment of asthma medication regimen by study clinician (see Section 7.1.1)
- Asthma education/counseling (see Section 7.1.1.5)

At Visits 4 and 13 only, spirometry and IOS with reversibility will be performed.

Visits 7 and 10 will include measurement of exhaled nitric oxide (see Section 8.1.4).

Visit 10 will include blood collection for CBC and differential (total eosinophil count) (see Section 8.2.1).

#### 8.10 Final Visit (Visit 14)

At the final visit, the following procedures and assessments will be performed:

- Urine cotinine (see Section 8.2.4)
- Urine pregnancy test, where indicated (see Section 8.2.3)
- Questionnaires (see Section 8.1.6)
- AE assessment (see Section 12)
- Concomitant medication assessment (see Sections 8.1.6 and 7.1.2)
- Vital signs (see Section 8.1.1)
- Spirometry (see Section 8.1.5)
- Targeted pulmonary examination by study clinician (see Section 8.1.2)
- Assignment of asthma medication regimen by study clinician (see Section 7.1.1)
- Asthma education/counseling (see Section 7.1.1.5)

- Exhaled nitric oxide (see Section 8.1.4)
- Nasal mucus sample collection (see Section 8.2.2)
- Nasal lavage (see Section 8.2.2)
- Nasosorption (see Section 8.2.2)
- Blood sample collection (see Section 8.2.1)
  - CBC with differential
  - Blood chemistry
  - Total and allergen-specific IgE
  - Blood markers (plasma/DNA/RNA)
  - Antibody to drug
- Sputum induction for a subset of children ≥10 years of age
- Nasal epithelial cell collection for a subset of children ≥10 years of age

#### 8.11 Cold Visits

Participants will be asked to report cold symptoms and come to the clinic at the start of up to three colds over the course of the 12-month follow-up. At this visit, the following activities will take place:

- Urine cotinine (see Section 8.2.4)
- Vital signs (see Section 8.1.1)
- Questionnaires (see Section 8.1.6)
- AE assessment (see Section 12)
- Concomitant medication assessment (see Sections 8.1.6 and 7.1.2)
- Spirometry and IOS (see Section 8.1.4)
- Targeted pulmonary exam (see Section 8.1.2)
- Exhaled nitric oxide (see Section 8.1.4)
- Nasal swab sample collection (see Section 8.2.2)
- Nasal lavage (see Section 8.2.2)
- Nasosorption (see Section 8.2.2)
- Blood sample collection (see Section 8.2.1)
  - o CBC with differential
  - Blood markers (plasma/DNA/RNA)

## 8.12 Exacerbation Follow-Up Visits

Over the course of the 12-month follow-up, participants who exacerbate will be asked to come in for a follow-up visit approximately 7 days following the start of systemic corticosteroids. As described in Section 3.2, exacerbations will be defined as a prescription of a course of systemic corticosteroids by a clinician, initiation of a course of systemic corticosteroids by a participant, or as a hospitalization for asthma. This visit will include:

- Urine cotinine (see Section 8.2.4)
- Vital signs (see Section 8.1.1)
- Questionnaires (see Section 8.1.6)
- AE assessment (see Section 12)
- Concomitant medication assessment (see Sections 8.1.6 and 7.1.2)

- Spirometry and IOS (see Section 8.1.4)
- Targeted pulmonary exam (see Section 8.1.2)
- Nasal swab sample collection (see Section 8.2.2)
- Nasal lavage (see Section 8.2.2)
- Nasosorption (see Section 8.2.2)
- Blood sample collection (see Section 8.2.1)
  - o CBC with differential
  - Blood markers (plasma/DNA/RNA)

## 8.13 Unscheduled Visits and Telephone Follow-up

Participants who experience asthma-related problems or concerns between scheduled study visits will be seen by a study clinician as warranted by the situation. If the site staff are notified by the participant, his/her family, an ED, a hospital, or clinic that the participant was seen for an unscheduled visit elsewhere, the site staff will contact the participant within 2 weeks of discharge to obtain an update on the participant's clinical status. A follow-up visit at the study center will be scheduled if needed. For details on the management plan, please refer to Section 7.1 and the Protocol ICAC-30 MOP.

Participants who are at Control Level 4 at a study visit will either be seen in the clinic or will receive a follow-up phone call within 1-2 weeks of the visit to check the status of their symptoms. Participants prescribed systemic corticosteroids who do not have an exacerbation study visit will receive a follow-up phone call within 1-2 weeks of the visit to check the status of their symptoms. If systemic corticosteroids were prescribed by a non-ICAC clinician and the participant does not come in for a study exacerbation visit, the participant will be seen in the clinic or will receive a follow-up phone call within 1-2 weeks to check the status of their symptoms. If this prescribing is uncovered more than two weeks after initiation of the corticosteroids, and the participant is doing well at the time of notification, then no follow up phone call is required.

Participants who have 2 exacerbations within a 1-month period must be seen in a face-to-face visit to determine if continuation in the study is in the best interest of the participant.

## 8.14 Visit Windows

Mepolizumab/placebo injections should be scheduled as close as possible to the every 4 week target date. See the Protocol ICAC-30 MOP for details regarding visit scheduling.

## 9 Mechanistic Assays

To identify the inflammatory pathways affected by mepolizumab treatment, we will examine airway gene expression using whole genome transcriptomics of nasal lavage and peripheral blood. Blood and nasal lavage samples for these studies will be collected pre-treatment (V1), early in the treatment period (V3), at the end of the study (V14), as well as during cold visits as described in Section 8.11 and exacerbation visits as described in Section 8.12. The quality of nasal lavage samples will be monitored regularly throughout the course of the study. Specifically, RNA will be extracted from samples for assessment of RNA concentration as well as integrity.

## 10 Biospecimen Storage

Unused samples of biological specimens collected during the course of the study will be stored (described in the Protocol ICAC-30 MOP) for future use for tests that may or may not be planned. These tests may or may not be related to the study of asthma and allergy. Participants will be asked to give permission for long-term storage and future use during the consent process. With the participant's approval and as approved by the Central IRB, de-identified biological samples will be stored indefinitely at the central repository.

## 11 Criteria for Participant and Study Completion and Premature Study Termination

## 11.1 Participant Completion

Participants are considered to have completed the study once they have completed the Final Study Visit.

## 11.2 Participant Stopping Rules and Withdrawal Criteria

Participants may be prematurely terminated from the study for the following reasons:

- 1. The participant elects to withdraw consent from all future study activities, including follow-up.
- 2. The participant is "lost to follow-up" as defined in the Protocol ICAC-30 MOP.
- 3. The participant dies.
- 4. Development of any serious medical illness whose natural history, sequela, or treatment would be worsened or impaired by continuation in the protocol.
- 5. The study clinician no longer believes participation is in the best interest of the participant.
- 6. The participant has an SAE related to investigational agent.
- 7. The participant becomes pregnant.
- 8. The participant has a need for > 3 bursts of systemic corticosteroids for asthma exacerbations during the treatment period OR has a need for > 2 bursts of systemic corticosteroids for asthma exacerbations within 6 months during the treatment period. If prescribed by an ICAC study clinician, a burst is defined as a course for prednisone, prednisolone, or methylprednisolone will be 2 mg/kg/day as a single daily dose for 4 days with a maximum dose of 60 mg per day. The course for dexamethasone will be 0.3 to 0.6 mg/kg/day as a single daily dose for 2 days with a maximum dose of 16 mg per day. If a corticosteroid burst for the treatment of an asthma exacerbation is prescribed by a non-ICAC clinician, it will be counted regardless of dose. If a participant initiates and completes a course of systemic corticosteroids without clinician involvement, this course will be counted only if the study clinician agrees the treatment was warranted, and it meets the following dosage: the course for prednisone, prednisolone, or methylprednisolone will be at least 20 mg daily dose for 3 of 5 consecutive days. The course for dexamethasone will be at least a 10 mg single daily dose.
- The participant has a need for > 14 days of prednisone (or prednisolone or methylprednisolone; defined as a minimum of 5 mg/day) over a 21 day period from Visit 1 through Visit 14.
- 10. The participant has a hypoxic seizure due to asthma.
- 11. The participant requires intubation due to asthma.
- 12. The participant has intolerable adverse experiences.

- 13. There is a major violation of the clinical trial protocol (defined as any variation from the protocol-directed conduct of the study that affects the safety of a participant or the ability of the trial to evaluate efficacy of the study agent).
- 14. The participant begins immunotherapy during the study period.
- 15. The participant has a new diagnosis of malignancy.
- 16. The participant has a new diagnosis requiring regular treatment with systemic corticosteroids, immunosuppressives, or any other drug that would interfere with participation in the study.
- 17. The participant has a serious parasitic infection and does not respond to treatment.

**Note:** If investigational product is discontinued by a study clinician, participants may continue on-study if agreed upon by the participant and study clinician (see Section 8.13).

#### 11.3 Participant Replacement

Participants who are discontinued prior to completing the 12-month follow up will not be replaced. All reasons for withdrawal will be captured on the appropriate electronic case report form (eCRF).

## 11.4 Follow-up after Early Study Withdrawal

Participants who withdraw or are dropped from the study between visits will be contacted by phone and will be invited to the study center for a final assessment. This assessment will include:

- Urine pregnancy test, where indicated (see Section 8.2.3)
- Questionnaires (see Section 8.1.6)
- AE assessment (see Section 12)
- Concomitant medication assessment (see Sections 8.1.6 and 7.1.2)
- Vital signs (see Section 8.1.1)
- Spirometry (see Section 8.1.5)
- Targeted pulmonary exam (see Section 8.1.2)
- Assignment of asthma medication regimen by study clinician (see Section 7.1.1)
- Asthma education/counseling (see Section 7.1.1.5)
- Blood sample collection (see Section 8.2.1)
  - o CBC with differential
  - Blood chemistry

Procedures contraindicated by the medical condition of the participant will not be conducted at the discretion of the study clinician. For participants who refuse to come to the clinic, the final clinical assessment as described above may be conducted over the phone. Besides this visit, no further follow-up will be made, except for participants who are discontinued due to pregnancy or SAEs. These participants will be contacted to determine the outcome of the pregnancy or the SAE. Refer to Section 12.6 for more information on AE reporting for pregnancy.

## 11.5 Study Stopping Rules

Study enrollment will be temporarily suspended pending expedited review of all pertinent data after the occurrence of one death or SAE which is unexpected and related to the investigational agent.

If the study enrollment is stopped due to meeting the above criteria, it may not be resumed until all pertinent information is discussed with the IND Sponsor (DAIT NIAID), NIAID Asthma and Allergy DSMB, and the Central IRB, and all parties concur with the resumption of the study. The FDA will be notified if stopping rules are met and also on resumption of the study.

The study may be terminated by the IND sponsor (DAIT NIAID) or the NIAID Allergy and Asthma DSMB upon review of any observations, events, or new information that merits such action.

## 12 Safety Monitoring and Reporting

#### 12.1 Overview

This section defines the types of safety data that will be collected under this protocol and outlines the procedures for appropriately collecting, grading, recording, and reporting those data. Adverse events that are classified as serious according to the definition of Health Authorities must be reported promptly (per Section 12.5, Reporting of Serious Adverse Events and Adverse Events) to the IND sponsor (DAIT NIAID). Appropriate notifications will also be made to site Principal Investigators, Institutional Review Boards (IRBs), and appropriate Health Authorities.

Information in this section complies with ICH Guideline E2A: Clinical Safety Data Management: Definitions and Standards for Expedited Reporting, ICH Guideline E-6: Guideline for Good Clinical Practice, 21CFR Parts 312 and 320, and applies the standards set forth in the National Cancer Institute, Common Terminology Criteria for Adverse Events (CTCAE), Version [enter 4.0 or correct version applicable to trial]: <a href="http://ctep.cancer.gov/reporting/ctc.html">http://ctep.cancer.gov/reporting/ctc.html</a>.

## 12.2 Definitions

#### 12.2.1 Adverse Event (AE)

Any untoward or unfavorable medical occurrence, or worsening of an undesirable or unintended sign, symptom, laboratory finding or disease that occurs during participation in the trial, whether or not considered related to the participant's participation in the research (modified from the definition of adverse events in the 1996 International Conference on Harmonisation E-6 Guidelines for Good Clinical Practice) (from OHRP "Guidance on Reviewing and Reporting Unanticipated Problems Involving Risks to Subjects or Others and Adverse Events (1/15/07)" http://www.hhs.gov/ohrp/policy/advevntguid.html#Q2)

AEs that occur due to a study procedure will be collected and recorded. The following clinical situations, when associated with study procedures, are defined as adverse events and will be recorded on the AE CRF. These situations do not limit the Principal Investigator from reporting to the Study Sponsor (DAIT NIAID) any other events, associated or not with these procedures, as AEs.

- Study therapy regimen: mepolizumab administered by the subcutaneous route
- **Study mandated procedures**: AEs that occur due to a study procedure will be collected and recorded. The following clinical situations, when associated with study procedures, are defined as adverse events and will be recorded on the AE eCRF. These situations do not limit the

Principal Investigator from reporting to the Study Sponsor any other events, associated or not with these procedures, as AEs.

## **Allergen Skin Testing**

- Prolonged (>24 hours) itching at test site
- Swelling (> 10 cm) at site of test lasting more than 24 hours
- Nasal allergic symptoms within 30 minutes of the procedure
- Fainting/Vasovagal event within 30 minutes of the procedure
- Anaphylaxis

#### **Blood Draws**

- Fainting/Vasovagal events
- Bruising at puncture site larger than 2 cm diameter
- Bleeding from puncture site lasting more than 30 minutes
- Swelling at puncture site larger than 2 cm

## **Pulmonary Function Testing**

- Wheezing or bronchoconstriction requiring treatment with bronchodilators within 30 minutes from the procedure
- Coughing requiring treatment with bronchodilators within 30 minutes from the procedure

## **Sputum Induction**

- Wheezing or bronchoconstriction requiring treatment with bronchodilators within 30 minutes from the procedure
- Coughing requiring treatment with bronchodilators within 30 minutes from the procedure

## **Nasal Lavage**

 Acute sinusitis diagnosed by study clinician or based upon assessment of outside health records within 72 hours after the procedure

## Nasal Blow / Nasal Mucus Sample Collection

 Acute sinusitis diagnosed by study clinician or based upon assessment of outside health records within 72 hours after the procedure

## **Nasal Epithelial Cell Collection**

Epistaxis within 24 hours of the procedure

#### **Nasal Swab Sample Collection**

- Epistaxis within 24 hours of the procedure
- Headache, earache or rhinorrhea lasting longer than 24 hours

## 12.2.1.1 Suspected Adverse Reaction

Any adverse event for which there is a reasonable possibility that the investigational drug [or investigational study therapy regimen] caused the adverse event. For the purposes of safety reporting, 'reasonable possibility' means there is evidence to suggest a causal relationship between the drug and the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug (21 CFR 312.32(a)).

## 12.2.2 Unexpected Adverse Event

An adverse event or suspected adverse reaction is considered "unexpected" when its nature (specificity), or severity, or rate of occurrence is not consistent with applicable product information as described in the safety information provided in the current GSK Investigator's Brochure for mepolizumab.

"Unexpected" also refers to adverse events or suspected adverse reactions that are mentioned in the current GSK Investigator's Brochure for mepolizumab as occurring with a class of drugs or as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with the particular drug under investigation (21 CFR 312.32(a)).

#### 12.2.3 Serious Adverse Event

An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or the IND sponsor (DAIT NIAID), it results in any of the following outcomes (21 CFR 312.32(a)):

- 1. Death.
- 2. A life-threatening event: An AE or SAR is considered "life-threatening" if, in the view of either the Principal Investigator or IND Sponsor, its occurrence places the participant at immediate risk of death. It does not include an AE or SAR that, had it occurred in a more severe form, might have caused death.
- 3. Inpatient hospitalization or prolongation of existing hospitalization.
- 4. Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- 5. Congenital anomaly or birth defect.
- 6. Important medical events that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above.

Elective hospitalizations, hospitalizations for pre-existing conditions that do not worsen during the course of the trial, or hospital admissions for the purpose of conduct of protocol mandated procedures are not to be reported as an SAE unless hospitalization is prolonged due to complications.

Exacerbations of asthma are ordinary, anticipated complications of asthma observed in patients receiving standard of care. An asthma exacerbation that requires hospitalization and is determined to be a SAR (Section 12.2.1.1) will be considered a SAE. All other asthma hospitalizations will not be considered SAEs and will be entered only on the appropriate CRFs. The date of onset of the asthma exacerbation SAE will be the date of hospital admission and the date of resolution will be the discharge date. The underlying condition will be followed as per protocol.

#### 12.3 Grading and Attribution of Adverse Events

Information in this section complies with *ICH Guideline E-6: Guidelines for Good Clinical Practice* and applies the following standards:

- Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (published September 2007) for local reactions to study procedures.
- Grading System of Severity of Anaphylaxis adapted, from the grading scale of Brown et al. (<sup>36</sup>) for anaphylaxis and systemic reactions to study procedures.
- National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (published June 14, 2010) for all other reactions. (This document is referred to herein as the "NCI-CTCAE manual.")

## 12.3.1 Grading Criteria

# **12.3.1.1** Adverse Events Related to Skin Testing and Injection Site Reactions Skin Testing

Excessive local reactions to skin testing not associated with systemic signs or symptoms will be graded according to Table 12.3.1.1a below. All AEs should be recorded on the eCRF.

| Grade | 1 (Mild) | 2 (Moderate) | (Severe) |
|---|---|---|---|
| Skin testing | Meets the minimum criteria listed in section 12.2.1, but requiring no medication other than topical corticosteroids or antihistamines. | Interfering with usual daily activities or sleep and requiring oral steroids. | Requiring a visit<br>to a health care<br>provider for<br>treatment |

**Table 12.3.1.1a Grading of Local Reactions to Study Procedures** 

#### **Anaphylaxis**

Criteria from <sup>37</sup>Sampson, et al. will be used to determine whether systemic allergic reactions constitute anaphylaxis (see Table 12.3.1.1b Clinical Criteria for Diagnosing Anaphylaxis). To be considered anaphylaxis, the event must involve at least two organ systems (e.g. not be simply a skin reaction). All anaphylaxis events, regardless of severity grade, will be recorded as Adverse Events and will be graded according to Table 12.3.1c Grading System of Severity of Anaphylaxis, adapted from the grading scale of <sup>36</sup>Brown et al.

## Table 12.3.1.1b Clinical Criteria for Diagnosing Anaphylaxis

## Anaphylaxis is highly likely when any one of the following 3 criteria are fulfilled:

- 1) Acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (e.g., generalized hives, pruritus or flushing, swollen lips-tongue-uvula) AND AT LEAST ONE OF THE FOLLOWING:
  - a) Respiratory compromise (e.g., dyspnea, wheeze-bronchospasm, stridor, reducted PEF, hypoxemia
  - Reduced BP or associated symptoms of end-organ dysfunction (e.g., hypotonia [collapse], syncope, incontinence)
- 2) Two or more of the following that occur rapidly after exposure to a <u>likely</u> allergen for that patient (minutes to several hours):
  - a) Involvement of the skin-mucosal tissue (e.g., generalized hives, itch-flush, swollen lips-tongue-uvula)
  - b) Respiratory compromise (e.g., dyspnea, wheeze-bronchospasm, stridor, reducted PEF, hypoxemia)
  - c) Reduced BP or associated symptoms (e.g., hypotonia [collapse], syncope, incontinence)
  - d) Persistent gastrointestinal symptoms (e.g., crampy abdominal pain, vomiting)
- 3) Reduced BP after exposure to known allergen for that patient (minutes or several hours):
  - a) Infants and children: low systolic BP (age specific) or greater than 30% decrease in systolic BP\*
  - b) Adults: systolic BP of less than 90 mm Hg or greater than 30% decrease from that person's baseline

PEF, Peak expiratory flow; BP, blood pressure.

\*Low systolic blood pressure for children is defined as less than 70 mm Hg from 1 month to 1 year, less than (70 mm Hg + [2 x age]) from 1 to 10 years, and less than 90 mm Hg from 11 to 17 years.

**Table 12.3.1.1c Grading System of Severity of Anaphylaxis** 

| Grade | Defined By |
|---|---|
| Mild (skin & subcutaneous tissues, GI, &/or mild respiratory) | Flushing, urticaria, periorbital or facial angioedema; mild dyspnea, wheeze or upper respiratory symptoms; mild abdominal pain and/or emesis |
| 2. Moderate (mild symptoms + features suggesting moderate respiratory, cardiovascular or GI symptoms) | Marked dysphagia, hoarseness, and/or stridor; shortness of breath, wheezing & retractions; crampy abdominal pain, recurrent vomiting and/or diarrhea; and/or mild dizziness |
| 3. Severe (hypoxia, hypotension, or neurological compromise) | Cyanosis or SpO2 ≤ 92% at any stage, hypotension, confusion, collapse, loss of consciousness; or incontinence |

## **Injection Site Reactions (ISRs)**

This study will grade injection site reactions as defined by the following table, from the Guidance for Industry – Toxicity Grading Scale for healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials, Food and Drug Administration, September 2007<sup>38</sup>.

Table 12.3.1.1d Grading System of Severity of Injection Site Reactions

| Local Reaction to<br>Injectable Product | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially<br>Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Pain | Does not interfere with activity | Repeated use of<br>non-narcotic pain<br>reliever >24 hours<br>or interferes with<br>activity | Any use of narcotic pain reliever or prevents daily activity | Emergency<br>room (ER) visit<br>or<br>hospitalization |
| Tenderness | Mild discomfort<br>to touch | Discomfort with movement | Significant discomfort at rest | ER visit or hospitalization |
| Erythema/Redness* | 2.5 – 5 cm | 5.1 – 10 cm | >10 cm | Necrosis or exfoliative dermatitis |
| Induration/Swelling** | 2.5 – 5 cm and<br>does not<br>interfere with<br>activity | 5.1 – 10 cm or interferes with activity | >10 cm or<br>prevents daily<br>activity | Necrosis |

<sup>\*</sup>In addition to grading the measured local reaction at the greatest single diameter, the measurement should be recorded as a continuous variable.

<sup>\*\*</sup>Induration/swelling should be evaluated and graded using the functional scale as well as the actual measurement.

#### 12.3.1.2 Grading and Attribution of All Other Adverse Events

The study site will grade the severity of adverse events experienced by the study participants according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 with the exception of anaphylaxis and injection site reactions (Section 12.3.1.1). This document (referred to herein as the NCI-CTCAE manual) provides a common language to describe levels of severity, to analyze and interpret data, and to articulate the clinical significance of all adverse events. The NCI-CTCAE has been reviewed by the Principal Investigators and has been deemed appropriate for the participant population to be studied in this protocol.

Adverse events will be graded on a scale from 1 to 5 according to the following standards in the NCI-CTCAE manual:

Grade 1 = mild adverse event

Grade 2 = moderate adverse event

Grade 3 = severe and undesirable adverse event

Grade 4 = life-threatening or disabling adverse event

Grade 5 = death

Events Grade 1 or higher will be recorded on the appropriate AE electronic case report form for this study.

For grading an abnormal value or result of a clinical or laboratory evaluation (including, but not limited to, a radiograph, an ultrasound, an electrocardiogram etc.), a treatment-emergent adverse event will rely on clinical judgment of the study clinician to determine if the value is an adverse event.

For additional information and a printable version of the NCI-CTCAE manual, consult the NCI-CTCAE web site: http://ctep.cancer.gov/reporting/ctc.html.

## 12.3.2 Attribution Definitions

The relationship, or attribution, of an adverse event to the study therapy regimen or study procedure(s) will initially be determined by the study clinician and recorded on the appropriate AE/SAE eCRF. Final determination of attribution for safety reporting will be determined by DAIT NIAID. The relationship of an adverse event to study therapy regimen or procedures will be determined using the descriptors and definitions provided in Table 12.3.2.

For additional information and a printable version of the NCI-CTCAE manual, consult the NCI-CTCAE web site: http://ctep.cancer.gov/reporting/ctc.html.

Descriptor Relationship (to primary investigational product Code and/or other concurrent mandated study therapy or study procedure) **UNRELATED CATEGORY** The adverse event is clearly not related; there is 1 Unrelated insufficient evidence to suggest a causal relationship. **RELATED CATEGORIES** The adverse event has a reasonable possibility to be Possible related; there is evidence to suggest a causal relationship. 3 Definite The adverse event is clearly related.

**Table 12.3.2 Attribution of Adverse Events** 

## 12.4 Collection and Recording of Adverse Events

#### 12.4.1 Collection Period

Inner-City Asthma Consortium

Adverse events will be collected from the time of consent until a participant completes study participation or until 30 days after he/she prematurely withdraws (without withdrawing consent) or is withdrawn from the study.

#### 12.4.2 Collecting Adverse Events

Adverse events (including SAEs) may be discovered through any of these methods:

- Observing the participant
- Interviewing the participant
- Receiving an unsolicited complaint from the participant
- In addition, an abnormal value or result from a clinical or laboratory evaluation can also indicate an adverse event, as defined in Section 12.3, Grading and Attribution of Adverse **Events**

## 12.4.3 Recording Adverse Events

Throughout the study, the study clinician will record adverse events and serious adverse events as described previously (Section 12.2, Definitions) on the appropriate AE/SAE eCRF regardless of the relationship to study therapy regimen or study procedure.

Once recorded, an AE/SAE will be followed until it resolves with or without seguelae, or until the end of study participation, or until 30 days after the participant prematurely withdraws (without withdrawing consent)/or is withdrawn from the study, whichever occurs first. The DAIT NIAID Medical Officer may request continued follow-up of an adverse event beyond the stated timeframe if deemed clinically important.

#### 12.5 Reporting of Serious Adverse Events and Adverse Events

## 12.5.1 Reporting of Serious Adverse Events to the IND Sponsor (DAIT NIAID)

This section describes the responsibilities of the Principal Investigator to report serious adverse events to the IND sponsor via SAE eCRF. Timely reporting of adverse events is required by 21 CFR and ICH E6 guidelines.

Principal Investigators will report all serious adverse events (see Section 12.2.3, Serious Adverse Event), regardless of relationship or expectedness within 24 hours of discovering the event.

For serious adverse events, all requested information on the AE/SAE eCRF will be provided. The following minimal criteria must be included in the initial SAE eCRF:

- AE Term
- Study Drug Treatment
- Relationship to study drug
- Reason why the event is serious

However, unavailable details of the event will not delay submission of the known information. As additional details become available, the AE/SAE eCRF will be updated and submitted.

#### 12.5.2 Reporting to FDA

After an adverse event requiring 24 hour reporting (per Section 12.5.1, Reporting of Serious Adverse Events to Sponsor) is submitted by the Principal Investigator and assessed by the IND sponsor (DAIT NIAID), there are two options for DAIT NIAID to report the adverse event to the FDA: annual reporting and expedited safety reporting.

#### 12.5.2.1 IND Annual Reporting

DAIT NIAID will include in the IND Annual Report to the FDA all adverse events classified as:

- Serious, expected, suspected adverse reactions (see Section 12.2.1.1, Suspected Adverse Reaction, and Section 12.2.2, Unexpected Adverse Event).
- Serious and not a suspected adverse reaction (see Section 12.2.1.1, Suspected Adverse Reaction).
- Pregnancies.

Note that all adverse events (not just those requiring 24-hour reporting) will be reported in the IND Annual Report.

#### 12.5.2.2 Expedited Safety Reporting

This option, with 2 possible categories, applies if the adverse event is classified as one of the following:

**Category 1: Serious and unexpected suspected adverse reaction [SUSAR]** (see Section 12.2.1.1, Suspected Adverse Reaction and Section 12.2.2, Unexpected Adverse Event and 21 CFR 312.32(c)i).

The sponsor shall report any suspected adverse reaction that is both serious and unexpected. The sponsor shall report an adverse event as a suspected adverse reaction only if there is evidence to suggest a causal relationship between the study drug and the adverse event, such as:

1. A single occurrence of an event that is uncommon and known to be strongly associated with drug exposure (e.g., angioedema, hepatic injury, or Stevens-Johnson Syndrome)

- One or more occurrences of an event that is not commonly associated with drug exposure, but is otherwise uncommon in the population exposed to the drug (e.g., tendon rupture)
- An aggregate analysis of specific events observed in a clinical trial (such as known consequences of the underlying disease or condition under investigation or other events that commonly occur in the study population independent of drug therapy) that indicates those events occur more frequently in the drug treatment group than in a concurrent or historical control group

## Category 2: Any findings from studies that suggests a significant human risk

The sponsor shall report any findings from other epidemiological studies, analyses of adverse events within the current study or pooled analysis across clinical studies or animal or in vitro testing (e.g. mutagenicity, teratogenicity, carcinogenicity) that suggest a significant risk in humans exposed to the drug that would result in a safety-related change in the protocol, informed consent, investigator brochure, or other aspects of the overall conduct of the study.

DAIT NIAID must notify the FDA and all participating Principal Investigators of expedited Safety Reports within 15 calendar days; unexpected fatal or immediately life-threatening suspected adverse reaction(s) shall be reported as soon as possible or within 7 calendar days.

#### 12.5.3 Reporting of Adverse Events to IRBs

All Principal Investigators must report adverse events, including expedited reports, in a timely fashion to the Central IRB in accordance with applicable regulations and guidelines. All IND Safety Reports to the FDA shall be distributed by the IND sponsor (DAIT NIAID) or designee to all participating institutions for Central IRB submission.

#### 12.6 Pregnancy Reporting

The Principal Investigator shall be informed immediately of any pregnancy in a study participant occurring from time of consent through 30 days after the participant completes study participation. A pregnant participant shall be instructed to stop taking study medication. The investigator shall counsel the participant and discuss the risks of continuing with the pregnancy and the possible effects on the fetus. Monitoring of the pregnant participant shall continue until the conclusion of the pregnancy.

The investigator shall report to the DAIT SACCC and the IND sponsor (DAIT NIAID) all pregnancies within 1 business day of becoming aware of the event using the Pregnancy eCRF. All pregnancies identified during the study shall be followed to conclusion and the outcome of each must be reported. The Pregnancy eCRF shall be updated and submitted to the DAIT SACCC when details about the outcome are available.

Information requested about the delivery shall include:

- Gestational age at delivery
- Birth weight, length, and head circumference
- Gender

- Appearance, pulse, grimace, activity, and respiration (APGAR) score at 1 minute, 5 minutes, and 24 hours after birth, if available
- Any abnormalities

All pregnancy complications that result in a congenital abnormality, birth defect, miscarriage, and medically indicated abortion - an SAE shall be submitted to the DAIT SACCC and the IND sponsor (DAIT NIAID) using the SAE reporting procedures described above.

#### 12.7 Reporting of Other Safety Information

A Principal Investigator shall promptly notify the Central IRB as well as the DAIT SACCC and the IND sponsor (DAIT NIAID) via email when an "unanticipated problem involving risks to subjects or others" is identified, which is not otherwise reportable as an adverse event.

#### 12.8 Review of Safety Information

#### 12.8.1 Medical Monitor Review

The DAIT NIAID Medical Monitor shall receive monthly reports from the DAIT SACCC compiling new and accumulating information on AEs, SAEs, and pregnancies recorded by the study site(s) on appropriate eCRFs.

In addition, the DAIT NIAID Medical Monitor shall review and make decisions on the disposition of the SAE and pregnancy reports received by the DAIT SACCC (See Sections 12.5 and 12.6).

#### 12.8.2 DSMB Review

## 12.8.2.1 Planned DSMB Reviews

The NIAID Allergy and Asthma Data and Safety Monitoring Board (DSMB) shall review safety data at least yearly during planned DSMB Data Review Meetings. Data for the planned safety reviews will include, at a minimum, a listing of all reported AEs and SAEs.

The DSMB will be informed of an Expedited Safety Report as determined by the DAIT NIAID Medical Monitor. An SAE which the DAIT NIAID Medical Monitor determines to be an unexpected safety risk will be sent to the DSMB immediately.

#### 12.8.2.2 Ad hoc DSMB Reviews

In addition to the pre-scheduled data reviews and planned safety monitoring, the DSMB may be called upon for *ad hoc* reviews. The DSMB will review any event that potentially impacts safety at the request of the protocol chair or the IND sponsor (DAIT NIAID). In addition, occurrences described in Section 11.5 Study Stopping Rules will trigger an ad hoc comprehensive DSMB Safety Review.

After review of the data, the DSMB will make recommendations regarding study conduct and/or continuation.

A temporary halt in enrollment and study treatment will be implemented if an ad hoc DSMB safety review is required.

## 13 Statistical Considerations and Analytical Plan

#### 13.1 Overview

The primary research question of this study is whether mepolizumab will lead to a reduced rate of asthma exacerbations in urban children and adolescents with difficult-to-control, exacerbation-prone asthma and peripheral blood eosinophils ≥150 cells/µl. This objective will be addressed using a multicenter, double-blind, placebo-controlled, randomized trial of mepolizumab adjunctive therapy for the prevention of asthma exacerbations in urban children and adolescents ages 6 to 17 years with difficult-to-control, exacerbation-prone asthma and peripheral blood eosinophilia.

#### 13.2 Endpoints/Outcomes

The primary endpoint is the number of asthma exacerbations between randomization and the end of participant follow-up or 12 months since randomization, whichever comes first. Exacerbations will be defined as a prescription of a course of systemic corticosteroids by a clinician, initiation of a course of systemic corticosteroids by a participant, or as a hospitalization for asthma. If a participant initiates and completes a course of systemic corticosteroids without clinician involvement, this course will be counted only if the study clinician agrees the treatment was warranted, and it meets the following dosage: the course for prednisone, prednisolone, or methylprednisolone will be at least 20 mg daily dose for 3 of 5 consecutive days. The course for dexamethasone will be at least a 10 mg single daily dose. If a corticosteroid burst for the treatment of an asthma exacerbation is prescribed by a non-ICAC clinician, it will be counted regardless of dose.

Key secondary endpoints include:

- 1. Asthma burden, as measured by a composite score (CASI) of asthma symptoms, medication usage, and exacerbation risk measured at Visits V1, V4, V7, V10, V13 and V14.
- 2. Patient reported outcomes, as measured by physician-patient global assessment tool measured at Visit V14.
- 3. Lung function, as assessed by spirometry measured at Visit V1, V4, V7, V10, V13, and V14 and IOS measured at Visit V1, V4, and V13.
- 4. Time between randomization and first asthma exacerbation or the end of participant followup, whichever comes first. Participants that do not have an asthma exacerbation will be rightcensored at the end of follow-up.

## 13.3 Measures to Minimize Bias

To minimize bias, randomization will be performed using a validated system created by the DAIT SACCC that automates the random assignment of treatment groups to study ID numbers. The randomization scheme will be reviewed by a statistician at the DAIT SACCC and locked after approval. Participants will be randomized using a 1:1 ratio of active and control (placebo) participants. A covariate adaptive randomization algorithm developed by Pocock and Simon  $(1975)^{32}$  will be used to maintain a balance between treatment arms with respect to study site, number of previous exacerbations (2 or 3+), peripheral blood eosinophils (< or  $\ge$ 400 cells/ $\mu$ l), BMI (< or  $\ge$ 95<sup>th</sup> percentile for age), total serum IgE (< or  $\ge$ 540 kUA/L) and treatment dose (40 mg or 100 mg). This strategy was chosen to enhance our ability to balance the distribution of covariates that are known to be highly associated with our primary endpoint (e.g., number of previous exacerbations and peripheral blood eosinophils) as well as covariates that determine if a participant fits the FDA-approved dosing tables for omalizumab therapy (e.g., BMI and total serum IgE), which is related to Secondary Objective 5.

#### 13.4 Analysis Plan

## 13.4.1 Analysis Populations

The following groups of participants will define samples for endpoint analysis:

- Modified Intent-to-treat (ITT) sample: All participants who are randomized and receive at least one dose of study treatment. Participants will be analyzed according to the treatment arm to which they were randomized, regardless of the medication they actually received.
- Safety sample: All participants who are randomized and receive at least one dose of study treatment. Participants will be analyzed according to the medication they actually received, regardless of the treatment arm to which they were randomized. Non-treatment emergent adverse events (e.g., any adverse event that occurs before the first injection) will be summarized in all participants who are enrolled, while treatment emergent adverse events (e.g., any adverse event that occurs on or after the first injection) will be summarized in the safety sample.
- Per-protocol (PP) sample: All participants who are randomized, received the correct medication and dosage to which they were randomized, do not have a major protocol deviation and cannot have missed 3 or more consecutive injections or 4 or more scheduled injections.

## 13.4.2 Primary Analysis of Primary Endpoint(s)/Outcome(s)

The primary analysis will compare the rate of exacerbations during the treatment period using a negative binomial model applied to the modified intent-to-treat sample. The model will include an offset term to account for differential follow-up among participants. To account for adaptive randomization, the model will also be adjusted for study site, number of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils (< or  $\ge$ 400 cells/ $\mu$ l), BMI (< or  $\ge$ 95th percentile for age), total serum IgE (< or  $\ge$ 540 kUA/L) and treatment dose (40 mg or 100 mg). Such a model will allow us to estimate the adjusted relative rate and corresponding 95% CI between the mepolizumab and placebo arms. A two-sided significance level of 0.05 will be used for this analysis. The reduction of the dose of mepolizumab from 100 mg to 40 mg in children 6 to 11 years of age and >40 kg will not affect the primary outcome as data from the GSK-sponsored pediatric trial 200363, NCT02377427 is therapeutically equivalent.

#### 13.4.3 Supportive Analyses of the Primary Endpoint(s)/Outcome(s)

Analyses for the primary endpoint may be supported by several analyses.

One disadvantage of a covariate adaptive randomization strategy is that Type I error may be inflated in certain circumstances (e.g., time trends). Consequently, rather than adjusting the model for the variables used in the adaptive randomization as discussed in Section 13.4.2, a permutation test will be used for inference instead as it involves fewer assumptions. Under a permutation model, the observed relative rate between the mepolizumab and placebo arms will be assessed with reference to all possible permutations that the treatment arms could have been assigned to participants.

Rather than adjusting the model for the variables used in the adaptive randomization, the model will instead adjust for study site (as a random or fixed effect), number of exacerbations in year prior to study (2, 3 or 4+), BMI percentile (treated as a continuous variable), total serum IgE (treated as a continuous variable and log-transformed, if appropriate) peripheral blood eosinophils (treated as a continuous variable and log-transformed, if appropriate), and treatment dose (40 or 100 mg).

To test if the effect of mepolizumab on the rate of asthma exacerbations during the treatment period is modified by particular sub-groups, separate negative binomial models of the rate of asthma exacerbations during the treatment period will be developed to test the two-way interaction between treatment arm and:

- Indicator for whether or not a participant fits the FDA-approved dosing table for omalizumab therapy
- BMI percentile at baseline (continuous or categorical)
- Peripheral blood eosinophils at baseline (continuous or categorical and log-transformed, if appropriate)
- Bronchodilator responsiveness at baseline (continuous or categorical)
- Number of exacerbations in year prior to study (2, 3 or 4+)
- Total serum IgE at baseline (continuous or categorical and log-transformed, if appropriate)
- Dose at baseline (40 mg or 100 mg)
- FeNO (continuous or categorical) at baseline
- Nasal ECP at baseline

To test if the effect of mepolizumab on the rate of asthma exacerbations during the treatment period is modified by both number of exacerbations in year prior to study as well as peripheral blood eosinophils, a separate negative binomial model of the rate of asthma exacerbations during the treatment period will be developed to test the three-way interaction between treatment arm, peripheral blood eosinophils (treated as either a piecewise linear spline or non-linear spline and log-transformed, if appropriate) and number of exacerbations in year prior to study (2, 3 or 4+).

## 13.4.4 Analyses of Secondary and Other Endpoint(s)/Outcome(s)

Generalized linear mixed models will be used to model CASI and lung function during the treatment period. A generalized logit model will be used to analyze the physician-patient global assessment at Visit 14. Kaplan-Meier curves and a Cox PH model will also be used to model the time to first asthma exacerbation during the treatment period.

As with the primary analyses, generalized linear mixed models, the generalized logit model, as well as the Cox PH model will include treatment arm as the primary exposure but will also adjust for study site, number of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils (above or below 400 cells/ $\mu$ l), BMI (above or below 95th percentile for age) and total serum IgE (above or below 540 kUA/L) to account for adaptive randomization.

To determine if mepolizumab reduces the rate of asthma exacerbation in participants who do not fit the FDA-approved dosing table for omalizumab therapy or alternatively, if mepolizumab reduces the rate of asthma exacerbation in participants who fit the FDA-approved dosing table, a separate negative

binomial model similar to that used for the primary analysis will be applied to all participants in the modified intent-to-treat sample in each of the 2 sub-groups. Because the goal of this objective is to estimate the effect of mepolizumab on the rate of asthma exacerbation in each sub-group, rather than compare these two effects using an interaction test, these effects will be reported regardless of the results obtained from the interaction test, which will be performed as part of the supportive analyses for the primary endpoint (see Section 13.4.3).

Safety will be summarized by arm in the safety sample by the number and percentage of serious and non-serious adverse events stratified by grade and relationship to treatment as well as the number and percentage of participants who have a serious and non-serious adverse event stratified by grade and relationship to treatment. Levels of antibody to mepolizumab will be analyzed in the safety sample using generalized linear mixed models as stated above in the mepolizumab arm only.

#### 13.4.5 Analyses of Exploratory Endpoint(s)/Outcome(s)

To determine whether mepolizumab improves other important clinical outcomes, including rate of virus-induced asthma exacerbations, ACT/cACT scores, maximum number of asthma symptom days or bronchodilator response, negative binomial models, generalized linear mixed models, generalized logit models, Kaplan-Meier curves and Cox PH models will be applied as appropriate to each endpoint in a manner similar to that described in Sections 13.4.2 to 13.4.4.

To identify immunologic pathways in the airways and peripheral blood that are characteristic of exacerbations prevented with and persistent despite anti-IL5 therapy, general linear models appropriate for RNA-sequencing count data will be used. Between group comparisons will be treated as a two independent group comparison and within group comparisons will use a mixed effect model with individual as a random effect. For comparisons where we are testing whether the two groups behave differently with a cold, an exacerbation, or over time, a general linear model will be created adding in these variables as main effects in the model and interaction terms between each effect. The general linear models will be expanded to include cell enumeration data as additional variables. Similarly, other salient variables (eg virus PCR data, collection site, collection time) that explain heterogeneity seen in the gene expression pattern, will be added to the model as appropriate. When relevant, predefined genes and gene sets of interest identified through Protocol ICAC-29 MUPPITS-1 results or previously published data will be tested separately without stringent multiple testing correction. Gene expression differences will be assigned to specific cell types using gene expression deconvolution algorithms appropriate for bulk cell population expression data. Predefined subgroups including PCR virus results, age, sex, race/ethnicity, obesity, timing of onset of asthma exacerbation relative to onset of cold symptoms, systemic corticosteroid use, season, nasal corticosteroid use, tobacco smoke exposure, and eNO will also be compared.

#### 13.4.6 Descriptive Analyses

Descriptive analyses will be reported separately for mepolizumab and placebo arms. Continuous baseline measures will be reported 1) means (or geometric means) with 95% confidence intervals, or 2) median with first and third quartiles, as appropriate. Categorical baseline and demographic characteristics and study disposition will be reported as frequencies and proportions.

#### 13.5 Interim Analyses

## 13.5.1 Interim Analysis of Efficacy Data

No formal interim analysis of efficacy data will be performed for this study.

## 13.5.2 Interim Analysis of Safety Data

The DSMB will receive periodic safety reports on enrolled participants. However, no formal interim analysis of safety data will be conducted.

#### 13.5.3 Futility Analysis

No formal futility analysis will be performed for this study.

## 13.6 Statistical Hypotheses

All primary and secondary objectives will be based on two-sided superiority tests. For instance, the null and alternative hypotheses for the primary objective are:

H0: The rate of asthma exacerbations during the treatment period in the mepolizumab arm is equal to the rate of asthma exacerbations during the treatment period in the placebo arm.

Ha: The rate of asthma exacerbations during the treatment period in the mepolizumab arm is not equal to the rate of asthma exacerbations during the treatment period in the placebo arm.

Additionally, Secondary Objective 5 will separately determine whether mepolizumab reduces the rate of asthma exacerbations in the sub-group of study participants who do not fit the FDA-approved dosing table for omalizumab therapy and in study participants who fit the FDA-approved dosing table for omalizumab therapy. In this case, the null and alternative hypotheses for this objective are:

H0: The rate of asthma exacerbations during the treatment period in the mepolizumab arm is equal to the rate of asthma exacerbations during the treatment period in the placebo arm in study participants who do not fit the FDA-approved dosing table for omalizumab therapy.

Ha: The rate of asthma exacerbations during the treatment period in the mepolizumab arm is not equal to the rate of asthma exacerbations during the treatment period in the placebo arm in study participants who do not fit the FDA-approved dosing table for omalizumab therapy.

H0: The rate of asthma exacerbations during the treatment period in the mepolizumab arm is equal to the rate of asthma exacerbations during the treatment period in the placebo arm in study participants who fit the FDA-approved dosing table for omalizumab therapy.

Ha: The rate of asthma exacerbations during the treatment period in the mepolizumab arm is not equal to the rate of asthma exacerbations during the treatment period in the placebo arm in study participants who fit the FDA-approved dosing table for omalizumab therapy.

#### 13.7 Sample Size Considerations

Based on Pavord et al,<sup>14</sup> the estimated relative rate of clinically significant asthma exacerbations between 75 mg, 250 mg, and 750 mg Mepolizumab arms and the Placebo arm was 0.52, 0.61, and 0.48 respectively. In Protocol ICAC-19 APIC, we found that among 94 enrolled participants that were difficult-to-treat at screening, had at least 2 exacerbations in the previous year at screening and peripheral blood eosinophils  $\geq$ 150 cells/µl, the rate of asthma exacerbations per patient –year was approximately 1.43

with an associated dispersion parameter of 0.47. Assuming that we will observe a relative rate similar to that seen in Pavord et al (2012) of 0.60 and that the event rate in the placebo arm is assumed to be 1.20 asthma exacerbations per patient-year with corresponding dispersion parameter of 0.50 in both arms, a total sample size of 256 participants (128 participants per arm) is required to detect such a relative rate with 90% power, based on a two-sided significance level of 0.05 and the work outlined in Zhu & Lakkis, <sup>39</sup> using maximum likelihood (method 3) for estimating the variance under the null hypothesis. Assuming approximately 20% of randomized participants do not meet criteria for modified intent-to-treat and are not replaced, we originally proposed to enroll 320 participants (160 participants per arm). However, our observed post-randomization dropout rate has been lower than expected (11%), and therefore the sample size was revised to 290.

Secondary Objective 5 will also determine if mepolizumab reduces the rate of asthma exacerbation in participants who do not fit the FDA-approved dosing table for omalizumab therapy and in participants who fit the FDA-approved dosing table for omalizumab therapy. In Protocol ICAC-19 APIC participants meeting Protocol ICAC-30 MUPPITS-2 eligible criteria, approximately 50% of participants did not fit the FDA-approved dosing table for omalizumab therapy and so we would expect approximately 128 participants (64 participants per arm) in each of these sub-groups in Protocol ICAC-30 MUPPITS-2. Assuming an event rate in the placebo arm of 1.20 and dispersion parameter of 0.50 in both arms, such a sample size would allow us to detect a relative rate between arms of 0.53 with 80% power.

#### 14 Identification and Access to Source Data

#### 14.1 Source Data

Source documents and source data are considered to be the original documentation where participant information, visits consultations, examinations and other information are recorded. Documentation of source data is necessary for the reconstruction, evaluation and validation of clinical findings, observations and other activities during a clinical trial. All clinical site laboratory reports, spirometry reports, and any paper and electronic CRFs will be maintained as source data.

#### 14.2 Access to Source Data

The Principal Investigators and site staff will make all source data available to the IND sponsor (DAIT NIAID), as well as to the FDA. Authorized representatives as noted above are bound to maintain the strict confidentiality of medical and research information that may be linked to identified individuals.

## 15 Protocol Deviations

#### 15.1 Protocol Deviation Definitions

#### 15.1.1 Protocol Deviation

The Principal Investigators and site staff will conduct the study in accordance to the protocol; no deviations from the protocol are permitted. Any change, divergence, or departure from the study design or procedures constitutes a protocol deviation. As a result of any deviation, corrective actions will be developed by the site and implemented promptly.

#### 15.1.2 Major Protocol Deviation

A protocol violation is a deviation from the IRB-approved protocol that may affect the participant's rights, safety, or well-being and/or the completeness, accuracy and reliability of the study data. In addition, protocol violations include willful or knowing breaches of human subject protection regulations, or policies, any action that is inconsistent with the NIH Human Research Protection Program's research, medical, and ethical principles, and a serious or continuing noncompliance with federal, state, local or institutional human subject protection regulations, policies, or procedures.

#### 15.1.3 Non-Major Protocol Deviation

A non-major protocol deviation is any change, divergence, or departure from the study design or procedures of a research protocol that does not have a major impact on the participant's rights, safety or well-being, or the completeness, accuracy and reliability of the study data.

#### 15.2 Reporting and Managing Protocol Deviations

The Principal Investigator has the responsibility to identify, document and report major and non-major protocol deviations as directed by the study Sponsor. However, major and non-major protocol deviations may also be identified during site monitoring visits or during other forms of study conduct review.

Upon determination that a protocol deviation (major or minor) has occurred, the study staff will a) notify the Principal Investigator (PI), b) notify the DAIT SACCC, and c) complete the Protocol Deviation form. The Protocol Deviation form will document at a minimum the date the protocol deviation (PD) occurred, the date PD identified, a description of event, whether the deviation resulted in SAE/AE, the signature of PI, report to Central IRB, and documentation of a corrective action plan. The DAIT SACCC and the IND sponsor (DAIT NIAID) may request discussion with the PI to determine the effect of the protocol deviation on the study participant and his/her further study participation, the effect of the protocol deviation on the overall study, and corrective actions. The PI will complete and sign the Protocol Deviation form and submit it to the DAIT SACCC and to the Central IRB, per IRB regulations. Major protocol deviations will be reported to the DSMB by the DAIT NIAID Medical Monitor at the Medical Monitor's discretion.

## 16 Ethical Considerations and Compliance with Good Clinical Practice

## 16.1 Quality Control and Quality Assurance

The Principal Investigator is required to keep accurate records to ensure that the conduct of the study is fully documented. The Principal Investigator is required to ensure that all CRFs are completed for every participant entered in the trial.

The sponsor is responsible for regular inspection of the conduct of the trial, for verifying adherence to the protocol, and for confirming the completeness, consistency, and accuracy of all documented data.

The CRFs will be completed online via a web-based electronic data capture (EDC) system that has been validated and is compliant with Part 11 Title 21 of the Code of Federal Regulations. Study staff at the site will enter information into the electronic CRFs, and the data will be stored remotely at a central database. Data quality will be ensured through the EDC system's continuous monitoring of data and real-time detection and correction of errors. All elements of data entry (i.e., time, date, verbatim text, Protocol ICAC-30 MUPPITS-2 Version 9.0 01/11/21

and the name of the person performing the data entry) will be recorded in an electronic audit trail to allow all changes in the database to be monitored and maintained in accordance with federal regulations.

## 16.2 Statement of Compliance

This clinical study will be conducted using good clinical practice (GCP), as delineated in *Guidance for Industry: E6 Good Clinical Practice Consolidated Guidance*, and according to the criteria specified in this study protocol. Before study initiation, the protocol and the informed consent documents will be reviewed and approved by the Central IRB. Any amendments to the protocol or to the consent materials will also be approved by the Central IRB before they are implemented.

The Principal Investigator will ensure that this study is conducted in full conformity with Regulations for the Protection of Human Subjects of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, and/or the ICH E6.

#### 16.3 Informed Consent Process

The consent process will provide information about the study to a prospective participant and parent(s)/legal guardian(s) and will allow adequate time for review and discussion prior to his/her decision. The Principal Investigator or designee listed on the FDA 1572 will review the consent and answer questions. The consent designee must be listed on the delegation log and have knowledge of the study. The prospective participant and parent(s)/legal guardian(s) will be told that being in the trial is voluntary and that he or she may withdraw from the study at any time, for any reason. All participants (or their legally acceptable representative) and parent(s)/legal guardian(s) will read, sign, and date a consent form before undergoing any study procedures. Assent will be obtained as per instruction by the Central IRB. Consent materials will be presented in participants' primary language. A copy of the signed consent form will be given to the participant.

The consent process will be ongoing. The consent form will be revised when important new safety information is available, the protocol is amended, and/or new information becomes available that may affect participation in the study.

#### 16.4 Privacy and Confidentiality

A participant's privacy and confidentiality will be respected throughout the trial. Each participant will be assigned a unique identification number and these numbers rather than names will be used to collect, store, and report participant information. Site personnel will not transmit documents containing personal health identifiers (PHI) to the study sponsor or their representatives.

#### 17 Publication Policy

Presentations and publication of the results of this trial will be governed by the ICAC Publication Policy.

#### 18 References

- 1. Wildfire JJ, Gergen PJ, Sorkness CA, et al. Development and validation of the Composite Asthma Severity Index--an outcome measure for use in children and adolescents. J Allergy Clin Immunol 2012;129:694-701.
- 2. Ortega HG, Liu MC, Pavord ID, et al. Mepolizumab Treatment in Patients with Severe Eosinophilic Asthma. The New England journal of medicine 2014.
- 3. O'Byrne PM, Pedersen S, Lamm CJ, Tan WC, Busse WW, Group SI. Severe exacerbations and decline in lung function in asthma. American journal of respiratory and critical care medicine 2009;179:19-24.
- 4. O'Brian AL, Lemanske RF, Jr., Evans MD, Gangnon RE, Gern JE, Jackson DJ. Recurrent severe exacerbations in early life and reduced lung function at school age. J Allergy Clin Immunol 2012:129:1162-4.
- 5. McGeachie MJ, Yates KP, Zhou X, et al. Patterns of Growth and Decline in Lung Function in Persistent Childhood Asthma. The New England journal of medicine 2016;374:1842-52.
- 6. Liu AH, Babineau DC, Krouse RZ, et al. Pathways through which asthma risk factors contribute to asthma severity in inner-city children. J Aller Clin Immunol 2016;138:1042-50.
- 7. Pongracic JA, Krouse RZ, Babineau DC, et al. Distinguishing Characteristics of Difficult-to-Control Asthma in Inner-City Children and Adolescents. J Aller Clin Immunol 2016;138:1030-41.
- 8. Zoratti EM, Krouse RZ, Babineau DC, et al. Asthma phenotypes in inner-city children. J Aller Clin Immunol 2016;138:1016-29.
- 9. Price DB, Rigazio A, Campbell JD, et al. Blood eosinophil count and prospective annual asthma disease burden: a UK cohort study. The lancet Respiratory medicine 2015;3:849-58.
- 10. Flood-Page P, Swenson C, Faiferman I, et al. A study to evaluate safety and efficacy of mepolizumab in patients with moderate persistent asthma. American journal of respiratory and critical care medicine 2007;176:1062-71.
- 11. Busse WW, Lemanske RF, Jr., Gern JE. Role of viral respiratory infections in asthma and asthma exacerbations. Lancet 2010;376:826-34.
- 12. Johnston SL, Pattemore PK, Sanderson G, et al. Community study of role of viral infections in exacerbations of asthma in 9-11 year old children. Bmj 1995;310:1225-9.
- 13. Kloepfer KM, Gern JE. Virus/allergen interactions and exacerbations of asthma. Immunology and allergy clinics of North America 2010;30:553-63, vii.
- 14. Pavord ID, Korn S, Howarth P, et al. Mepolizumab for severe eosinophilic asthma (DREAM): a multicentre, double-blind, placebo-controlled trial. Lancet 2012;380:651-9.
- 15. Pavord ID, Bafadhel M. Exhaled nitric oxide and blood eosinophilia: independent markers of preventable risk. J Allergy Clin Immunol 2013;132:828-9.
- 16. Robinson DS. The role of the mast cell in asthma: induction of airway hyperresponsiveness by interaction with smooth muscle? J Allergy Clin Immunol 2004;114:58-65.
- 17. Busse WW. Asthma diagnosis and treatment: filling in the information gaps. J Allergy Clin Immunol 2011;128:740-50.
- 18. Evans R, 3rd, Gergen PJ, Mitchell H, et al. A randomized clinical trial to reduce asthma morbidity among inner-city children: results of the National Cooperative Inner-City Asthma Study. The Journal of pediatrics 1999;135:332-8.
- 19. Morgan WJ, Crain EF, Gruchalla RS, et al. Results of a home-based environmental intervention among urban children with asthma. The New England journal of medicine 2004;351:1068-80.
- 20. Busse WW, Morgan WJ, Gergen PJ, et al. Randomized trial of omalizumab (anti-IgE) for asthma in inner-city children. The New England journal of medicine 2011;364:1005-15.

- 21. Szefler SJ, Mitchell H, Sorkness CA, et al. Management of asthma based on exhaled nitric oxide in addition to guideline-based treatment for inner-city adolescents and young adults: a randomised controlled trial. Lancet 2008;372:1065-72.
- 22. Bai TR, Vonk JM, Postma DS, Boezen HM. Severe exacerbations predict excess lung function decline in asthma. Eur Respir J 2007;30:452-6.
- 23. Bochner BS, Gleich GJ. What targeting eosinophils has taught us about their role in diseases. J Allergy Clin Immunol 2010;126:16-25; quiz 6-7.
- 24. Leckie MJ, ten Brinke A, Khan J, et al. Effects of interleukin-5 blocking monoclonal antibody on eosinophils, airway hyperresponsiveness and the late asthmatic response. Lancet 2000;(in press).
- 25. Haldar P, Brightling CE, Hargadon B, et al. Mepolizumab and exacerbations of refractory eosinophilic asthma. The New England journal of medicine 2009;360:973-84.
- 26. Green RH, Brightling CE, McKenna S, et al. Asthma exacerbations and sputum eosinophil counts: a randomised controlled trial. Lancet 2002;360:1715-21.
- 27. Nair P, Pizzichini MM, Kjarsgaard M, et al. Mepolizumab for prednisone-dependent asthma with sputum eosinophilia. The New England journal of medicine 2009;360:985-93.
- 28. Bel EH, Wenzel SE, Thompson PJ, et al. Oral Glucocorticoid-Sparing Effect of Mepolizumab in Eosinophilic Asthma. The New England journal of medicine 2014.
- 29. Ortega H, Li H, Suruki R, Albers F, Gordon D, Yancey S. Cluster analysis and characterization of response to mepolizumab: A step closer to personalized medicine for patients with severe asthma. Annals of the American Thoracic Society 2014.
- 30. Liu Y, Zhang S, Li DW, Jiang SJ. Efficacy of anti-interleukin-5 therapy with mepolizumab in patients with asthma: a meta-analysis of randomized placebo-controlled trials. PloS one 2013;8:e59872.
- 31. Ortega H, Chupp G, Bardin P, et al. The role of mepolizumab in atopic and nonatopic severe asthma with persistent eosinophilia. Eur Respir J 2014;44:239-41.
- 32. Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics 1975;31:103-15.
- 33. Mepolizumab (SB-240563) Investigator's Brochure. 05Nov2016.
- 34. NUCALA Prescribing Information. 2017. (Accessed 21 Apr, 2017, at https://www.gsksource.com/pharma/content/dam/GlaxoSmithKline/US/en/Prescribing\_Information/Nucala/pdf/NUCALA-PI-PIL.PDF.)
- 35. Fahy JV, Boushey HA, Lazarus SC, et al. Safety and reproducibility of sputum induction in asthmatic subjects in a multicenter study. American journal of respiratory and critical care medicine 2001;163:1470-5.
- 36. Brown SG. Clinical features and severity grading of anaphylaxis. J Allergy Clin Immunol 2004;114:371-6.
- 37. Sampson HA M-FA, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol 2006;117:7.
- 38. Guidance for Industry Toxixity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. 2007. (Accessed 21 Apr, 2017, at https://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/Vaccines/ucm091977.pdf.)
- 39. Zhu H, Lakkis H. Sample size calculation for comparing two negative binomial rates. Statistics in medicine 2014;33:376-87.

## Appendix A: Schedule of Procedures/Evaluations

| | Scree-<br>ning | Rand<br>omiz<br>ation | | | | | | Tr | eatment | : Phase ( | (12 mon | ths) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Asthma Management | | | | | | | | | | | | | | | |
| Week | 0 | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | PRN | PRN |
| Visit | V0 | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12 | V13 | V14 | Cold+ | EX# |
| Consent/Assent | + | | | | | | | | | | | | | | | | |
| Medical history | + | | | | | | | | | | | | | | | | |
| Asthma Eval & Mgt | + | + | | | + | | | + | | | + | | | + | + | | |
| Asthma Counseling | + | + | | | + | | | + | | | + | | | + | + | | |
| Spirometry | + | + | | | + | | | + | | | + | | | + | + | + | + |
| IOS | | + | | | + | | | | | | | | | + | | + | + |
| Bronchodilator<br>reversibility (Spiro &<br>IOS) | | + | | | + | | | | | | | | | + | | | |
| CASI | + | + | | | + | | | + | | | + | | | + | + | | |
| ACT/c-ACT | + | + | | | + | | | + | | | + | | | + | + | | |
| Physician-patient global assessment tool | | | | | | | | | | | | | | | + | | |
| Physical Exam | + | | | | | | | | | | | | | | | | |
| Targeted pulmonary exam | | + | | | + | | | + | | | + | | | + | + | + | + |
| Lungs assessment | | | + | + | | + | + | | + | + | | + | + | | | | |
| FeNO | | + | | + | | | | + | | | + | | | | + | + | |
| SQ study drug/placebo | | + | + | + | + | + | + | + | + | + | + | + | + | + | | | |
| Pregnancy test | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | | |
| Urinary cotinine | | + | | + | | | | | | | | | | | + | + | + |
| Blood collection | + | + | | + | | | | | | | + | | | | + | + | + |
| CBC with differential | + * | + | | + | | | | | | | + | | | | + | + | + |
| Blood chemistry | + | | | + | | | | | | | | | | | + | | |
| Serum total IgE & specific IgE | + | | | | | | | | | | | | | | + | | |
| Blood markers<br>(plasma/RNA/DNA) | | + | | + | | | | | | | | | | | + | + | + |
| Antibodies to drug | | + | | + | | | | | | | | | | | + | | |
| Skin Testing | +* | | +* | +* | +* | | | | | | | | | | | | |
| Nasal lavage | | + | | + | | | | | | | | | | | + | + | + |
| Nasosorption | | | | | | | | | | | | | | | + | + | + |

Protocol ICAC-30 MUPPITS-2

Version 9.0
| Г | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Nasal blow | | + | + | + | + | + | + | + | + | + | + | + | + | + | + | | |
| Nasal resp virus | | + | + | + | + | + | + | + | + | + | + | + | + | + | + | | |
| Nasal ECP | | + | + | + | + | | | + | | | | | | | + | | |
| Nasal swab collection^ | | | | | | | | | | | | | | | | + | + |
| Nasal epithelial cell collection | | | | | | | | | | | | | | | +** | | |
| Sputum Induction | | | | | | | | | | | | | | | +** | | |
| Vital signs and growth parameters | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + |
| Adverse event assessment | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + |
| Concomitant medication assessment | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + |

<sup>\*</sup> may use CBC results collected in another ICAC protocol if within past 6 months and allergen skin tests performed in another ICAC protocol if within past 12 months – skin tests can be performed at V0, V2, V3 or V4 if not previously obtained in past 12 months

<sup>+</sup> up to two with an optional third cold visit will occur for each participant

<sup>#</sup> as needed exacerbation visits to occur 7 days after start of systemic corticosteroids

<sup>\*\*</sup> to be performed in participants 10 years and older

<sup>^</sup>Nasal swab collection replaced the nasal blow procedure at cold and exacerbation visits in Protocol Version 8.0

#### **Appendix B: Nasal Lavage Quality Control Methods**

#### 1 Study Population

#### 1.1 Population Description

Clinical research staff performing nasal lavage will be required to demonstrate proficiency in performing the procedure within Protocol ICAC-30 MUPPITS-2. The proficiency testing will be conducted by collecting and processing nasal lavage samples from individuals that have signed a consent specific to this procedure. Up to 200 participants may be enrolled across the research sites to ensure all study staff members are trained.

#### 1.1.1 Inclusion Criteria

Participants to be included in this training are those:

- 1. who are male or female age 6-17, inclusive
- 2. have a history of asthma
- 3. who are willing and able to provide informed consent
- 4. who are willing and able to provide assent, if applicable

#### 1.2 Requirements

All clinical research staff performing the nasal lavage collection and processing must perform at least two proficiency tests. After collection and processing, the site staff will send the samples to a central lab for review. The central lab will determine whether the samples are sufficient. If a sample is deemed not sufficient, then the staff member may be required to repeat the proficiency testing.

#### 1.3 Procedures

The nasal lavage collection and processing procedures are detailed in the Protocol ICAC-30 MOP; however, the study clinician will not have the option to use a nasal decongestant prior to performing the nasal lavage for the quality control procedure (as described in Section 8.2.2).

#### **Appendix C: Omalizumab Dosing Tables**

Table 1. Subcutaneous Xolair Doses Every 4 Weeks for Patients 12 Years of Age and Older with Asthma

| Pre-treatment | Body Weight | | | |
|---|---|---|---|---|
| Serum IgE | 30-60 kg | > 60-70 kg | > 70–90 kg | > 90-150 kg |
| ≥ 30-100 IU/mL | 150 mg | 150 mg | 150 mg | 300 mg |
| > 100-200 IU/mL | 300 mg | 300 mg | 300 mg | |
| > 200-300 IU/mL | 300 mg | | | |
| > 300-400 IU/mL | | SEE TA | ABLE 2 | |
| > 400-500 IU/mL | | | | |
| > 500-600 IU/mL | | | | |

Table 2. Subcutaneous Xolair Doses Every 2 Weeks for Patients 12 Years of Age and Older with Asthma

| Pre-treatment | Body Weight | | | |
|---|---|---|---|---|
| Serum IgE | 30-60 kg | > 60-70 kg | > 70-90 kg | > 90-150 kg |
| ≥ 30-100 IU/mL | SEE TABLE 1 | | | |
| > 100-200 IU/mL | | SEE 17 | 225 mg | |
| > 200-300 IU/mL | | 225 mg | 225 mg | 300 mg |
| > 300-400 IU/mL | 225 mg | 225 mg | 300 mg | |
| > 400-500 IU/mL | 300 mg | 300 mg | 375mg | |
| > 500-600 IU/mL | 300 mg | 375 mg | DO NOT DOSE | |
| > 600-700 IU/mL | 375 mg | | | |

Pediatric patients 6 to <12 years of age: Initiate dosing according to Table 3.

Table 3. Subcutaneous Xolair Doses Every 2 or 4 Weeks\* for Pediatric Patients with Asthma Who Begin Xolair Between the Ages of 6 to <12 Years

| Pre-treatment | Dosing | Body Weight | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Serum IgE<br>(IU/mL) | Freq. | 20-25 | >25-30 | >30-40 | >40-50 | >50-60 | >60-70 | >70-80 | >80-90 | >90-125 | >125-150 |
| (TO/IIIL) | | kg | kg | kg | kg | kg | kg | kg | kg | kg | kg |
| | | | | | | Do | se (mg) | | | | |
| 30-100 | | 75 | 75 | 75 | 150 | 150 | 150 | 150 | 150 | 300 | 300 |
| >100-200 | | 150 | 150 | 150 | 300 | 300 | 300 | 300 | 300 | 225 | 300 |
| >200-300 | | 150 | 150 | 225 | 300 | 300 | 225 | 225 | 225 | 300 | 375 |
| >300-400 | Every | 225 | 225 | 300 | 225 | 225 | 225 | 300 | 300 | | |
| >400-500 | 4 | 225 | 300 | 225 | 225 | 300 | 300 | 375 | 375 | | |
| >500-600 | weeks | 300 | 300 | 225 | 300 | 300 | 375 | | | | |
| >600-700 | | 300 | 225 | 225 | 300 | 375 | | | | | |
| >700-800 | | 225 | 225 | 300 | 375 | | | | | | |
| >800-900 | Ever | 225 | 225 | 300 | 375 | | | DO NO | OT DOS | E | |
| >900-1000 | Every<br>2 | 225 | 300 | 375 | | | | | | | |
| >1000-1100 | weeks | 225 | 300 | 375 | | | | | | | |
| >1100-1200 | | 300 | 300 | | | | | | | | |
| >1200-1300 | | 300 | 375 | | | | | | | | |

#### \*Dosing frequency:

☐ Subcutaneous doses to be administered every 4 weeks ☐ Subcutaneous doses to be administered every 2 weeks

#### **Appendix D: Sputum Induction Quality Control Methods**

#### 1 Study Population

#### 1.1 Population Description

Clinical research staff performing sputum induction will be required to demonstrate proficiency in performing the procedure within Protocol ICAC-30 MUPPITS-2. The proficiency testing will be conducted by collecting and processing sputum samples from individuals who have signed a consent specific to this procedure. Up to 100 participants may be enrolled across a subset of clinical research sites to ensure all study staff members are trained.

#### 1.1.1 Inclusion Criteria

Participants to be included in this procedure are those who:

- 1. Are male and female age 10-17, inclusive
- 2. Have a history of asthma
- 3. Are willing and able to provide informed consent
- 4. Are willing and able to provide assent

#### 1.2 Requirements

All clinical research staff performing the sputum induction processing must perform at least two proficiency tests. After collection and processing, the site staff will send the samples to a central lab for review. The central lab will determine whether the samples are sufficient. If a sample is deemed not sufficient, then the staff member may be required to repeat the proficiency testing.

#### 1.3 Procedures

The sputum induction collection and processing procedures are detailed in the Protocol ICAC-30 MUPPITS-2 MOP.

#### Appendix E: Study Restrictions Due to COVID-19

In the event of institutional or ICAC-wide restrictions on certain types of procedures or certain classes of research due to COVID-19, some study procedures may be suspended. This may include certain in-person study visits or specific inhalation or nasal procedures, such as:

- Spirometry
- Impulse Oscillometry
- Exhaled nitric oxide
- Sputum Induction
- Nasal lavage sampling
- Nasal blow sampling
- Nasal epithelial cell collection

If in-person visits are suspended, study staff will continue to make contact with study participants and will conduct visits over the phone. Prescriptions for asthma management medications can be sent to local pharmacies and additional prednisone, if needed, can be mailed to the participant.

### STATISTICAL ANALYSIS PLAN

## MECHANISMS UNDERLYING ASTHMA EXACERBATIONS PREVENTED AND PERSISTENT WITH IMMUNE-BASED THERAPY:

#### A SYSTEMS APPROACH PHASE 2

#### **PROTOCOLICAC-30**

SHORT TITLE: MUPPITS-2

NCT#:

COMPOUND #:

SPONSOR: The Division of Allergy, Immunology, and Transplantation (DAIT), The

National Institute of Allergy and Infectious Diseases (NIAID)

REGULATORY

AGENCY IDENTIFIER NUMBER(S):

IND #: 136355 PREPARED BY: Rho

> 2635 E NC Hwy 54 Durham, NC 27713

Telephone: (919) 408-8000

Fax: (919) 408-0999

This document is confidential and proprietary to the National Institute of Allergy and Infectious Diseases. This study is being conducted in compliance with good clinical practice, including the archiving of essential documents. Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be reproduced, published, or otherwise disclosed without the prior written approval of National Institute of Allergy and Infectious Diseases, except that this document may be disclosed to appropriate Institutional Review Boards under the condition that they keep the information confidential.

## ACKNOWLEDGEMENT AND SIGNATURE SHEET


| Approved: | DROTOCOL CO CILAIR | Date: |
|-----------|----------------------------------------------|-------|
| | PROTOCOL CO-CHAIR -<br>DANIEL J. JACKSON, MD | |
| Approved: | PROTOCOL CO-CHAIR -<br>WILLIAM W. BUSSE, MD | Date: |
| Approved: | MEDICAL MONITOR -<br>PETER GERGEN, MD, MPH | Date: |
| Approved: | RESEARCH SCIENTIST – CYNTHIA VISNESS, PHD | Date: |
| Approved: | BIOSTATISTICIAN –<br>MIGUEL VILLARREAL | Date: |

## **VERSION HISTORY**

| SAP Version | Version Date | Comments/Changes |
|-------------|--------------|------------------|
| 0.1 | 16 DEC 2020 | Initial Version |
| 1.0 | 01 APR 2021 | Version 1.0 |

## TABLE OF CONTENTS

| 1. | LIST OF ABBREVIATIONS | 7 |
|--------|------------------------------------------------|----|
| 2. | PURPOSE OF THE ANALYSES | 9 |
| 3. | PROTOCOL SUMMARY | 10 |
| 4. | GENERAL ANALYSIS AND REPORTING CONVENTIONS | 15 |
| 5. | ANALYSIS SAMPLES | 16 |
| 6. | STUDY SUBJECTS | 17 |
| 6.1. | Disposition of Subjects | 17 |
| 6.2. | Demographic and Other Baseline Characteristics | 18 |
| 6.3. | Prior and Concomitant Medications | 18 |
| 7. | STUDY OPERATIONS | 19 |
| 7.1. | Protocol Deviations | 19 |
| 7.2. | Randomization | 19 |
| 7.3. | Measures of Treatment Adherence | 19 |
| 8. | ENDPOINT EVALUATION | 20 |
| 8.1. | Overview of Efficacy Analysis Methods. | 20 |
| 8.1.1. | Multicenter Studies. | 20 |
| 8.1.2. | Assessment Time Windows | 20 |
| 8.1.3. | Multiple Comparisons/Multiplicity | 20 |
| 8.2. | Primary Endpoint | 20 |
| 8.2.1. | Computation of the Primary Endpoint | 20 |
| 8.2.2. | Primary Analysis of the Primary Endpoint | 21 |
| 8.2.3. | Sensitivity Analyses of the Primary Analysis | 21 |
| 8.2.4. | Secondary Analyses of the Primary Endpoint | 21 |
| 8.3. | Secondary Endpoints | 22 |
| 8.3.1. | Endpoint 1 | 22 |
| 8.3.2. | Endpoint 2 | 22 |
| 8.3.3. | Endpoint 3 | 23 |
| 8.3.4. | Endpoint 4. | 23 |
| 8.3.5. | Endpoint 5 | 23 |
| 8.3.6. | Endpoint 6 | 23 |

| * | • | |
|---|---|---|
| 8.4. | Other Endpoints | 23 |
| 8.4.1. | Exploratory Analysis of the Primary Endpoint | 23 |
| 8.4.2. | Exploratory Endpoints | 24 |
| 9. | SAFETY EVALUATION | 25 |
| 9.1. | Overview of Safety Analysis Methods | 25 |
| 9.2. | Adverse Events | 26 |
| 9.3. | Deaths, Serious Adverse Events | 27 |
| 9.4. | Clinical Laboratory Evaluation | 27 |
| 9.5. | Vital Signs and Growth Parameters, Physical Findings, and Targeted Pulmonary Exam Results | 27 |
| 9.5.1. | Vital Signs and Growth Parameters | 27 |
| 9.5.2. | Physical Examinations | 28 |
| 9.5.3. | Targeted Pulmonary Exam | 28 |
| 10. | OTHER ANALYSES | 29 |
| 11. | INTERIM ANALYSES AND DATA MONITORING | 30 |
| 12. | CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL | 31 |
| 13. | REFERENCES | 32 |
| 14. | APPENDIX | 33 |
| 14.1. | Study Flow Chart | 33 |
| 14.2. | Schedule of Events | 33 |

| ICAC<br>{Statistical | Analysis Plan - Protocol #} |
|----------------------|-----------------------------|
| | LIST OF TABLES |
| Table 1: | List of Abbreviations |

## 1. LIST OF ABBREVIATIONS

**Table 1: List of Abbreviations** 

| Abbreviation | Term |
|--------------|------------------------------------------------------|
| ACT | Asthma Control Test |
| AE | Adverse Event |
| BP | Blood Pressure |
| BMI | Body Mass Index |
| cACT | Childhood Asthma Control Test |
| CASI | Composite Asthma Severity Index |
| CI | Confidence Interval |
| COVID-19 | Coronavirus Disease 2019 |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DAIT | Division of Allergy, Immunology, and Transplantation |
| DSMB | Data Safety Monitoring Board |
| ECP | Eosinophil Cationic Protein |
| eCRF | Electronic Case Report Form |
| FeNO | Fractional Exhaled Nitric Oxide |
| FEV1 | Forced Expiratory Volume in 1 Second |
| GCP | Good Clinical Practice |
| GSK | GlaxoSmithKline (GSK) Group Company |
| IB | Investigator's Brochure |
| ICAC | Inner City Asthma Consortium |
| ICH | International Conference on Harmonization |
| ID | Participant Study Identifier |
| IgE | Immunoglobulin E |
| IgG | Immunoglobulin G |
| IL | Interleukin |
| IND | Investigational New Drug |
| IOS | Impulse Oscillometry |
| IRB | Institutional review Board |

| NIAID | National Institute of Allergy and Infectious Diseases |
|--------|-------------------------------------------------------|
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intent-to-Treat |
| PD | Protocol Deviation |
| PT | Preferred Term |
| SACCC | Statistical and Clinical Coordinating Center |
| SD | Standard Deviation |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SAR | Suspected Adverse Reaction |
| SOC | System Organ Class |
| TEAE | Treatment-Emergent Adverse Event |

#### 2. PURPOSE OF THE ANALYSES

The purpose of this statistical analysis plan (SAP) is to describe the planned analyses and data displays to be included in the Clinical Study Report (CSR) for Protocol ICAC-30 MUPPITS-2. This document provides details on study populations, how the variables will be derived, how missing data will be handled and details on statistical methods to be used to analyze the safety and efficacy data.

The statistical analysis plan (SAP) is based on ICH guidelines E3 and E9 (Statistical Principles for Clinical Trials).

The document may evolve over time, for example, to reflect the requirements of protocol amendments or regulatory requests. However, the final SAP must be finalized, approved by the Sponsor, and placed on file before database is locked. Deviations from the final approved plan will be noted in the clinical study report.

## 3. PROTOCOL SUMMARY

| Title | Mechanisms Underlying Asthma Exacerbations Prevented and<br>Persistent with Immune-Based Therapy: A Systems Approach<br>Phase 2 |
|---|---|
| Short Title | Protocol ICAC-30 MUPPITS-2 |
| Clinical Phase | II |
| Number of Sites | Multiple |
| IND Sponsor/Number | IND sponsor: DAIT NIAD<br>IND#: 136355 |
| Primary Hypothesis | The primary research question of this study is whether mepolizumab will lead to a reduced rate of asthma exacerbations in urban children and adolescents (ages 6-17) with difficult-to-control, exacerbation-prone asthma and peripheral blood eosinophils ≥150 cells/µl. We hypothesize that targeting eosinophils with the addition of the anti-IL-5 monoclonal antibody, mepolizumab, will prevent exacerbations and, as a consequence, reduce overall morbidity and improve asthma control. |
| Study Objectives | The primary objective of the study is to determine if phenotype-directed use of mepolizumab reduces the rate of asthma exacerbations as defined by the need for systemic corticosteroid treatment in urban children and adolescents (ages 6-17) with difficult-to-control exacerbation-prone asthma and peripheral blood eosinophils ≥150 cells/µl. |
| | <ol> <li>Secondary objectives are: <ol> <li>To determine whether mepolizumab will lead to an improved Composite Asthma Severity Index (CASI)<sup>1</sup></li> <li>To determine whether mepolizumab will improve quality of life as assessed by the physician-patient global assessment<sup>2</sup></li> <li>To determine whether mepolizumab improves lung function as assessed by spirometry and impulse oscillometry</li> </ol> </li> <li>To determine whether mepolizumab increases the time to first asthma exacerbation</li> <li>To separately determine whether mepolizumab reduces the rate of asthma exacerbations in study participants who do not fit the</li> </ol> |


| Study Design | FDA-approved dosing table for omalizumab therapy and in study participants who fit the FDA-approved dosing table for omalizumab therapy 6. To assess the safety of mepolizumab treatment Protocol ICAC-30 MUPPITS-2 is a multicenter, double-blind, placebo-controlled, randomized trial of mepolizumab adjunctive therapy for the prevention of asthma exacerbations in urban children and adolescents with difficult-to-control exacerbation- |
|---|---|
| Primary Endpoint(s) | prone asthma and peripheral blood eosinophils ≥150 cells/μl. The primary endpoint is the number of asthma exacerbations during the treatment period. |
| Secondary Endpoint(s) | <ol> <li>CASI during the treatment period</li> <li>Quality of life as measured by the physician-patient global assessment</li> <li>Lung function as assessed by spirometry and IOS during the treatment period</li> <li>Time to first asthma exacerbation during the treatment period</li> <li>Number of reported adverse events and serious adverse events, including their severity and treatment relatedness</li> </ol> |
| Accrual Objective | 290 |
| Study Duration | 27 months recruitment + 12 months treatment |
| Agent/Treatment<br>Description | <ul> <li>Mepolizumab (anti-IL-5 antagonist monoclonal antibody) by subcutaneous injection every 4 weeks at the following doses:</li> <li>Age 12 years and above: 100 mg</li> <li>Age 6-11 years: 40 mg Participants 6 to 11 years of age and weighing ≥40 kg who were enrolled in Protocol ICAC-30 MUPPITS-2 under the previous versions of the protocol and initially assigned a 100 mg dose will have their dose reduced to 40 mg. Participants age 11 years will increase to the 100 mg dose if they become age 12 years during the study. </li> </ul> |
| Inclusion Criteria | <ol> <li>Participant and/or parent guardian must be able to understand<br/>and provide informed consent and age-appropriate assent</li> <li>Are male and female aged 6-17 years, inclusive at<br/>randomization</li> </ol> |

## 

| | <ol> <li>Have a primary place of residence in one of the pre-selected recruitment census tracts as outlined in the Protocol ICAC-30 Recruitment Manual of Operations <ul> <li>3a. Participants who do not live in the pre-selected census tracts but live within the Office of Management and Budget (OMB) defined Metropolitan Statistical Area and have publicly-funded health insurance will qualify for inclusion.</li> </ul> </li> <li>Have had a diagnosis of asthma made &gt; 1 year prior to recruitment; participants who received an asthma diagnosis by a clinician ≤ 1 year prior to recruitment must report that their respiratory symptoms were present for more than 1 year prior to recruitment</li> <li>Have had at least two asthma exacerbations in the prior year (defined as a requirement for systemic corticosteroids and/or hospitalization)</li> <li>At Visit 0 (Screening), have the following requirement for asthma controller medication: for participants aged 6 to 11 years, treatments with at least fluticasone 250 mcg dry powder inhaler (DPI) one puff twice daily or its equivalent and for participants aged 12 years and older, treatment with at least fluticasone 250 mcg plus LABA DPI one puff twice daily or its equivalent</li> <li>Have peripheral blood eosinophils ≥150 cells/μl obtained at Visit 0 or via another ICAC protocol within 6 months</li> <li>Are able to perform spirometry at randomization</li> <li>Have documentation of current medical insurance with prescription coverage at randomization</li> <li>Have had varicella or the varicella vaccination</li> </ol> |
|---|---|
| Exclusion Criteria | Individuals who meet any of the following criteria are not eligible for enrollment or randomization, if they: |
| | <ol> <li>Are not able or willing to give written informed consent or comply with study protocol</li> <li>Have concurrent medical problems that would require systemic</li> </ol> |
| | <ul> <li>corticosteroids or other immunomodulators during the study</li> <li>Are currently receiving immunotherapy</li> <li>Are currently receiving treatment with omalizumab or have had omalizumab treatment within 6 months prior to randomization</li> </ul> |


- 5. Are currently requiring greater than fluticasone 500 mcg bid plus LABA one puff twice daily or its equivalent and/or individuals using oral corticosteroids daily or every other day for more than 14 days at the time of Visit 0 (Screening)
- 6. Are currently pregnant or lactating, or plan to become pregnant during the time of study participation. Females of child-bearing potential (post-menarche) must be abstinent or use a medically acceptable birth control method throughout the study (e.g. oral subcutaneous, mechanical, or surgical contraception)
- 7. Have a known, pre-existing clinically important lung condition other than asthma
- 8. Have a current malignancy or previous history of cancer in remission for less than 12 months prior to randomization
- 9. Have known, pre-existing, unstable liver disease
- 10. Is a current smoker
- 11. Have a known immunodeficiency disease
- 12. Have other conditions that could lead to elevated eosinophils such as hypereosinophilic syndromes, including eosinophilic granulomatosis with polyangiitis
- 13. Have a known, active pre-existing parasitic infestation or undergoing treatment for a parasitic infestation. Once the participant has been successfully treated, the participant may be reevaluated.
- 14. Use of investigational drugs within 4 weeks of randomization
- 15. Have past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study
- 16. Will not allow the study clinician, an asthma specialist, to manage their disease for the duration of the study or who are not willing to change their asthma medications to follow the protocol
- 17. Have a known history of allergic reaction to previous biologic therapy for asthma

| | 18. Have had a life threatening asthma exacerbation in the last 2 years requiring intubation, mechanical ventilation or resulting in a hypoxic seizure |
|---|---|
| Study Stopping Rules | The occurrence of one death or an unexpected SAE related to the investigational agent. |

#### 4. GENERAL ANALYSIS AND REPORTING CONVENTIONS

The following analyses and reporting conventions will be used:

Categorical variables will be summarized using counts (n) and percentages (%) and will be presented in the form "n (%)." Percentages will be rounded to one decimal place. If a count is 0, 0% will be shown for the percentage.

Continuous variables will be summarized using sample size (n), mean, standard deviation (SD), median, first and third quartiles, minimum (min), and maximum (max), as appropriate. The mean will be reported at one more significant digit than the precision of the data, the standard deviation will be reported at two more significant digits than the precision of the data, and first and third quartiles, minimum, maximum, and median will be reported at the same precision as the data. The median will be reported as the average of the two middle numbers if the dataset contains an even number of observations.

Test statistics including t, z, and  $\chi$ 2 test statistics will be reported to two decimal places.

P-values will be reported to three decimal places if greater than or equal to 0.001. If less than 0.001, the value will be reported as "<0.001." A p-value can be reported as "1.000" only if it is exactly 1.000 without rounding. A p-value can be reported as "0.000" only if it is exactly 0.000 without rounding.

Each data listing will be sorted by treatment arm and subject identifier (ID) unless otherwise noted.

If departures from these general conventions are present in the specific evaluations section of this SAP, then those conventions will take precedence over these general conventions.

#### 5. ANALYSIS SAMPLES

The following groups of participants will define samples for endpoint analysis:

- Modified Intent-to-treat (ITT) sample: All participants who are randomized and receive at least one dose of study treatment. Participants will be analyzed according to the treatment arm to which they were randomized, regardless of the medication they actually received.
- Safety sample: All participants who are randomized and receive at least one dose of study treatment. Participants will be analyzed according to the medication they actually received, regardless of the treatment arm to which they were randomized. Non-treatment emergent adverse events (e.g., any adverse event that occurs before the first injection) will be summarized in all participants who are enrolled, while treatment emergent adverse events (e.g., any adverse event that occurs on or after the first injection) will be summarized in the safety sample.
- Per-protocol (PP) sample: All participants who are randomized, received the correct medication and dosage to which they were randomized, do not have a major protocol deviation and cannot have missed 3 or more consecutive injections or 4 or more scheduled injections.

#### 6. STUDY SUBJECTS

### 6.1. Disposition of Subjects

The disposition of all enrolled participants, defined as those who consented/assented, will be summarized in a table and listed. The following disposition information will be included in the table:

- The number of participants who had a screening visit (Visit 0)
- Among screened participants:
  - o The number and percentage of participants who were deemed ineligible
- Among randomized participants:
  - o The number and percentage of participants in the mITT population.
  - o The number and percentage of participants in the safety population.
  - o The number and percentage of participants in the PP population.
- Among participants in the mITT population and grouped by treatment arm:
  - o The number and percentage of participants in the safety population.
  - o The number and percentage of participants in the PP population.
  - o The number and percentage of participants who withdrew during the study due to:
    - Withdrawal of consent/assent
    - Major protocol violation
    - Pregnancy
    - Investigator decision
    - Started exclusionary medication
    - Started immunotherapy
    - Intubation due to asthma
    - Hypoxic seizure due to asthma
    - Developed exclusionary condition
    - Development of serious medical illness
    - >14 days of prednisone over a 21-day period
    - Exacerbation stopping rules
    - Death
    - SAE related to injection
    - Intolerable adverse event
    - Lost to follow-up
    - Did not meet randomization criteria
    - Withdrawal of consent/assent due to positive diagnosis of Coronavirus Disease 2019 (COVID-19)
    - Coronavirus Disease restrictions


- Other
- The number and percentage of participants who discontinued study treatment and primary reason for discontinuation.

A data listing of participant disposition will be provided for the mITT population, sorted by treatment arm and ID.

#### 6.2. Demographic and Other Baseline Characteristics

Descriptive statistics for demographic and baseline characteristics will be summarized for the mITT population grouped by randomized treatment arm and overall.

Demographic data will include age at randomization, sex, race, ethnicity, and clinical study site.

Baseline will be defined as the last measurement prior to or on the day of randomization. Baseline characteristics will include:

- Weight
- Height
- Body Mass Index (BMI) percentile, BMI categorical variable (< or ≥95% for age)
- Number of previous exacerbations (2 or 3+)
- Peripheral blood eosinophils (< or >=400 cells/ul)
- Total serum IgE (< or >=540 kUA/L)
- Treatment dose (40 mg or 100 mg)

A data listing of demographics, baseline characteristics, and medical history will be provided for the mITT population. A data listing of all participants who had visits that were remote or missed due to COVID-19 will be provided for the mITT population and will include the number of visits that were remote or missed due to COVID-19 for each participant

#### 6.3. Prior and Concomitant Medications

Prior and concomitant medications will be listed for the mITT population by treatment arm and ID.

#### 7. STUDY OPERATIONS

#### 7.1. Protocol Deviations

Protocol deviations will be recorded on the protocol deviation electronic case report form (eCRF) page. Major protocol deviations will be identified by the DAIT Medical Monitor and study team prior to unblinding of treatment assignment and database lock.

Protocol deviations will be summarized in tabular format by treatment arm and by type of deviation (including major deviations). A data listing of all protocol deviations sorted by treatment arm and participant ID.

#### 7.2. Randomization

Randomization was performed using a validated system created by the DAIT SACCC that automated the random assignment of treatment groups to study ID numbers. Participants were randomized using a 1:1 ratio of active and control (placebo) participants. A covariate adaptive randomization algorithm developed by Pocock and Simon (1975)⁴ was used to maintain a balance between treatment arms with respect to study site, number of previous exacerbations (2 or 3+), peripheral blood eosinophils (< or ≥400 cells/µl), BMI (< or ≥95th percentile for age), total serum IgE (< or ≥540 kUA/L) and treatment dose (40 mg or 100 mg). This strategy was chosen to enhance the ability to balance the distribution of covariates that are known to be highly associated with our primary endpoint (e.g., number of previous exacerbations and peripheral blood eosinophils) as well as covariates that determine if a participant fits the FDA-approved dosing tables for omalizumab therapy (e.g., BMI and total serum IgE).

#### 7.3. Measures of Treatment Adherence

The number of completed injections will be determined for each participant, and divided by the total number of expected injections (up to 13) given the amount of time in the study. The proportion of completed injections will be summarized by treatment arm and overall. Each injection, injection dose, baseline age, age at clinical visit, and weight will be listed by participant ID, visit, and by treatment arm.

#### 8. ENDPOINT EVALUATION

#### 8.1. Overview of Efficacy Analysis Methods

#### 8.1.1. Multicenter Studies

Although this is a multicenter study, the data is intended to be collected and analyzed as a whole. There are too few participants enrolled in the study relative to the number of sites to perform formal analyses stratified by site.

#### 8.1.2. Assessment Time Windows

Mepolizumab/placebo injections were scheduled as close as possible to the every 4-week target date as outlined in the Schedule of Events (Section 15.1). Any data collected outside of a visit window will still be included in any analyses of the scheduled visit.

At the onset of the COVID-19 pandemic, the following procedures were restricted, and were site-specific: Impulse oscillometry, spirometry, FeNO, nasal lavage samples, nasal blow samples, nasal epithelial cell collection, and sputum samples. Exacerbation visits were conducted only via telephone and cold visits were suspended. If participants were unable to come into the study center for visits, the visits were conducted via telephone.

#### 8.1.3. Multiple Comparisons/Multiplicity

Adjustment for multiplicity will not be performed for the primary or secondary endpoints.

### 8.2. Primary Endpoint

#### 8.2.1. Computation of the Primary Endpoint

For participants who completed the study, the primary endpoint is the number of asthma exacerbations between randomization and the end of participant follow-up (Visit 14), or four weeks from the final injection--whichever comes first. For participants who terminated from the study early, the primary endpoint is number of exacerbations between randomization and their last known completed visit.

Exacerbations are defined as a prescription of a course of systemic corticosteroids by a clinician, initiation of a course of systemic corticosteroids by a participant, or as a hospitalization for asthma. If a participant initiated and completed a course of systemic corticosteroids without clinician involvement, this course will be counted only if the study clinician agrees the treatment was warranted, and it meets the following dosage: the course for prednisone, prednisolone, or methylprednisolone will be at least 20 mg daily dose for 3 of 5 consecutive days. The course for dexamethasone will be at least a 10 mg single daily dose. If a corticosteroid burst for the treatment of an asthma exacerbation was prescribed by a non-ICAC clinician, it was counted regardless of dose.


#### 8.2.2. Primary Analysis of the Primary Endpoint

The primary analysis will compare the rate of exacerbations during the treatment period using a negative binomial model applied to the mITT sample. The model will include an offset term to account for differential follow-up among participants. To account for adaptive randomization, the model will also be adjusted for study site, number of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils (< or ≥400 cells/µl), BMI (< or ≥95th percentile for age), total serum IgE (< or ≥540 kUA/L) and treatment dose (40 mg or 100 mg). Such a model will allow us to estimate the adjusted relative rate and corresponding 95% CI between the mepolizumab and placebo arms. A two-sided significance level of 0.05 will be used for this analysis.

Although the primary version of the primary analysis will be conducted on the mITT sample, the same analysis of the primary endpoint will be performed for the PP population.

#### 8.2.3. Sensitivity Analyses of the Primary Analysis

At the time of the COVID-19 pandemic and subsequent quarantine period, observable exacerbation rates decreased relative to observed rates in the prior years of the study. In order to account for the unknown effects of the pandemic on the primary endpoint, the exacerbation rate will be analyzed using the same model as specified in section 8.2.2, but only including participants who were randomized, received at least one injection, and who had at least one follow-up visit prior to March 16, 2020. For participants who met this definition, only exacerbations that occurred between randomization and March 16, 2020 will be analyzed in the model. All subsequent exacerbations and follow-up time will be censored after March 16, 2020. The offset variable used in the model will be defined as the length of time, in years, from randomization to the end of a participant's follow-up, or March 16, 2020, whichever occurs first.

The same analysis will be applied to the PP population.

#### 8.2.4. Secondary Analyses of the Primary Endpoint

Analyses for the primary endpoint may be supported by several analyses.

One disadvantage of a covariate adaptive randomization strategy is that Type I error may be inflated in certain circumstances (e.g., time trends). Consequently, rather than adjusting the model for the variables used in the adaptive randomization as discussed in Section 8.2.2, a permutation test will be used for inference instead as it involves fewer assumptions. Under a permutation model, the observed relative rate between the mepolizumab and placebo arms will be assessed with reference to all possible permutations that the treatment arms could have been assigned to participants, or up to 5000 iterations.

Rather than adjusting the model for the variables used in the adaptive randomization, the model will instead adjust for study site (as a random or fixed effect), number of exacerbations in year prior to study (2, 3 or 4+), BMI percentile (treated as a continuous variable), total serum IgE (treated as a continuous variable and log-transformed, if appropriate) peripheral blood


eosinophils (treated as a continuous variable and log-transformed, if appropriate), and treatment dose (40 or 100 mg).

#### 8.3. Secondary Endpoints

#### **8.3.1.** Endpoint 1

Variable: Composite Asthma Severity Index (CASI) at Visits 4, 7, 10, 13, and 14.

Analysis: A generalized linear mixed model will be used to model CASI during the treatment period. The model will include a fixed effect for treatment arm as the primary exposure but will also adjust for baseline CASI, study site, number of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils (above or below 400 cells/µl), BMI (above or below 95th percentile for age) and total serum IgE (above or below 540 kUA/L) to account for adaptive randomization. Visit will be treated as a categorical variable in the model, and an interaction term between treatment arm and visit will be used to estimate the least square mean CASI for each treatment arm for each timepoint of measurement. The difference in least square mean, the corresponding 95% CI and the p-values will be provided for the comparison of mepolizumab vs placebo. The model will be fit using restricted maximum likelihood, and each fixed effect will be tested using an F-test statistic, the Kenward-Roger approximation for the degrees of freedom, an unstructured covariance matrix, and a two-sided significance level of 0.05. If the model assuming an unstructured covariance matrix does not converge, other covariance structures, such as a spatial power covariance structure, will be considered. Descriptive statistics including the number of participants, mean, and standard deviation will also be presented. This analysis will be conducted on the mITT population.

As sites were restricted to limited visit assessments due to COVID-19, lung function assessments were not performed and FEV1 (% predicted), a domain of the CASI score, was not collected. In these cases, the last known FEV1 (% predicted) value, from Visit 4 or onward, will be used to calculate a participant's CASI at subsequent visits. Additionally, sites were discouraged from stepping down participants' asthma controller therapy during the pandemic, another domain of the CASI score, which could bias the results towards the null.

#### **8.3.2.** Endpoint 2

Variable: Quality of life, as measured by physician-patient global assessment, at Visit 14

Analysis: A generalized logit model will be used to analyze the physician-patient global assessment at Visit 14 for the mITT population. The model will include treatment arm as a fixed effect as the primary exposure but will also adjust for study site, number of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils (above or below 400 cells/µl), BMI (above or below 95th percentile for age) and total serum IgE (above or below 540 kUA/L). A table will summarize the observed quality of life measurements, as recorded in the CRF at Visit 14, by treatment arm. No imputation of missing data will be used for participants who were not assessed for quality of life measurements at Visit 14.


#### **8.3.3.** Endpoint 3

Variable: Lung function as assessed by spirometry and impulse oscillometry

Analysis: A generalized mixed model as described in section 8.3.1 will be used to analyze each spirometry and impulse oscillometry parameter, separately, at each visit where the lung function was collected for the mITT population. It is noted that lung function data was not collected during the limited assessment visits during the COVID-19 pandemic and is considered missing completely at random. No imputation of missing data will be used in the analysis of lung function data.

#### **8.3.4.** Endpoint 4

Variable: Time to first asthma exacerbation

Analysis: Kaplan-Meier curves and a Cox PH model will also be used to model the time to first asthma exacerbation during the treatment period. The Cox PH model will include treatment arm as the primary exposure but will also adjust for study site, number of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils (above or below 400 cells/µl), BMI (above or below 95th percentile for age) and total serum IgE (above or below 540 kUA/L). The analysis will be conducted for the mITT population ignoring the COVID-19 intercurrent event

#### 8.3.5. **Endpoint 5**

**Variable:** Rate of exacerbations (mepolizumab vs. placebo) during the treatment period for participants in the mITT sample who do not fit the FDA-approved dosing table for omalizumab therapy and for participants who do fit the FDA-approved dosing table.

**Analysis:** A negative binomial model, as specified in section 8.2.2, will be used to estimate the effect of mepolizumab on the rate of exacerbation, as compared to the placebo group, in the omalizumab-eligible and omalizumab-ineligible sub-groups. A treatment and a treatment by omalizumab-eligibility interaction term will be used to estimate the exacerbation rates.

#### **8.3.6.** Endpoint 6

Variable: Adverse Events

Analysis: Safety will be summarized treatment arm in the safety sample by the number and percentage of serious and non-serious adverse events stratified by grade and relationship to treatment as well as the number and percentage of participants who have a serious and non-serious adverse event stratified by grade and relationship to treatment. See Section 9 for further details and definitions.

## 8.4. Other Endpoints

#### **8.4.1.** Exploratory Analysis of the Primary Endpoint


To test if the effect of mepolizumab on the rate of asthma exacerbations during the treatment period is modified by particular sub-groups, separate negative binomial models of the rate of asthma exacerbations during the treatment period will be developed to test the two-way interaction between treatment arm and:

- BMI percentile at baseline (continuous or categorical)
- Peripheral blood eosinophils at baseline (continuous or categorical and log-transformed, if appropriate)
- Bronchodilator responsiveness at baseline (continuous or categorical)
- Number of exacerbations in year prior to study (2, 3 or 4+)
- Total serum IgE at baseline (continuous or categorical and log-transformed, if appropriate)
- Dose at baseline (40 mg or 100 mg)
- FeNO (continuous or categorical) at baseline

To test if the effect of mepolizumab on the rate of asthma exacerbations during the treatment period is modified by both number of exacerbations in year prior to study as well as peripheral blood eosinophils, a separate negative binomial model of the rate of asthma exacerbations during the treatment period will be developed to test the three-way interaction between treatment arm, peripheral blood eosinophils (treated as either a piecewise linear spline or non-linear spline and log-transformed, if appropriate) and number of exacerbations in year prior to study (2, 3 or 4+).

#### **8.4.2.** Exploratory Endpoints

Analyses of exploratory endpoints and outcomes will be conducted as described in section 13.4.5 of the protocol.

#### 9. SAFETY EVALUATION

#### 9.1. Overview of Safety Analysis Methods

The safety analyses will be performed in the safety population defined in Section 5. Safety assessment summaries will include:

- AEs, defined in Protocol Section 12.2.1.
- Suspected Adverse Reactions (SARs), defined in Protocol Section 12.2.1.1.
- Unexpected Adverse Event, defined in Protocol Section 12.2.2
- AEs leading to discontinuation of study drug
- AEs leading to discontinuation from study
- Serious adverse events (SAEs), defined in Protocol Section 12.2.3.
- Deaths
- Clinical laboratory results
- Vital signs

Adverse events were collected from the time of consent until a participant completes study participation or until 30 days after he/she prematurely withdraws (without withdrawing consent) or is withdrawn from the study.

For this analysis, a treatment-emergent adverse event (TEAE) will be defined as any AE not present prior to the initiation of study drug or any AE already present that worsens in either intensity or frequency following exposure to study drug. TEAEs will be summarized in the safety population.

Partial dates will be imputed for the purposes of defining TEAEs as follows:

- For a missing start day where the month and year are present, the start day will be set to the first day of the month, unless: 1) the first day of the month is before the date of administration of study drug and the month and year are the same as the month and year of the date of administration of study drug; and 2) the end date is on or after the date of administration of study drug or the end date is completely missing, in which case the start day will be set to the day of administration of study drug.
- For a missing start day and month where the year is present, the start day and month will be set to January 1<sup>st</sup>, unless: 1) January 1<sup>st</sup> is before the date of administration of study drug and the year is the same as the year of the date of administration of study drug; and 2) the end date is on or after the date of administration of study drug or the end date is completely missing, in which case the start day and month will be set to that of the date of administration of study drug.


- For a missing end day where the month and year are present, the end day will be set to the last day of the month, unless the month and year are the same as the month and year of the last contact date for the participant, in which case the end day will be set to that of the participant's last contact date.
- For a missing end day and month where the year is present, the end day and month will be set to the participant's last contact date, unless the year of the participant's last contact date is greater than the end year, in which case the end day and month will be set to December 31st.

Unless otherwise specified, a data listing for all measurements in Section 9 will be provided for the safety population and sorted in order of treatment arm, participant ID, and time of assessment (e.g., visit, time, and/or event).

#### 9.2. Adverse Events

All AEs will be classified by system organ class (SOC) and preferred term, according to a standardized thesaurus (Medical Dictionary for Regulatory Activities [MedDRA]). MedDRA V20.0 or later will be used to classify all AEs.

The severity of AEs will be classified, as applicable, using the following criteria and complies with *ICH Guideline E-6: Guidelines for Good Clinical Practice*:

- Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (published September 2007) for local reactions to study procedures.
- Grading System of Severity of Anaphylaxis adapted, from the grading scale of Brown et al. (3) for anaphylaxis and systemic reactions to study procedures.
- National Cancer Institute *Common Terminology Criteria for Adverse Events Version 4.03* (published June 14, 2010) for all other reactions. (This document is referred to herein as the "NCI-CTCAE manual.")

The relationship, or attribution, of an adverse event to the study therapy regimen or study procedure(s) will initially be determined by the study clinician and recorded on the appropriate AE/SAE eCRF. Final determination of attribution for safety reporting will be determined by DAIT NIAID. The relationship of an adverse event to study therapy regimen or procedures will be determined using the descriptors and definitions provided in Table 12.3.2 of the protocol.

Overall summary tables will be developed using the safety population to report the number of events and the number and percentage of participants having at least one treatment-emergent event in the following categories:

- AEs
- AEs by maximum grade for each of the following:
  - Skin Testing
  - Anaphylaxis


- Injection Site Reactions
- CTCAE

TEAEs classified by treatment arm, MedDRA SOC, and preferred term will be summarized in the Safety Population for each of the following categories:

- AEs
- AEs by relationship to study drug

Summary tables will present the total number of events as well as the number and percentage of participants experiencing the events. If a participant experiences the same AE on multiple occasions, the event will be counted once for each occurrence when reporting the number of AEs. When reporting the number of participants experiencing the events, a participant will only be counted once if they experience an event within the particular SOC or preferred term. Percentages will be based on the number of participants in the safety population.

Similar summaries will be generated for SARs (defined in Protocol Section 12.2.3), AEs leading to discontinuation of study drug, and AEs leading to study withdrawal separately.

Data listings will be provided separately for AEs, SARs, AEs leading to discontinuation of study drug, and cases of COVID-19.

#### 9.3. Deaths, Serious Adverse Events

SAEs will be listed and summarized in the same manner described in Section 9.2. Separate displays listing death, including time to death and primary cause of death, will also be created.

## 9.4. Clinical Laboratory Evaluation

Clinical laboratory measurements will be performed at Screening and at various visits throughout the study and include a complete blood count with differential (CBC). Results will be converted to standardized units where possible. For numeric laboratory results, descriptive statistics of laboratory values will be presented for each treatment arm and overall. For categorical laboratory results, the number and percentage of participants reporting each result will be presented for each treatment arm and overall. A data listing of all laboratory measurements including an indication of any abnormal values and clinical significance will be provided.

## 9.5. Vital Signs and Growth Parameters, Physical Findings, and Targeted Pulmonary Exam Results

#### 9.5.1. Vital Signs and Growth Parameters

Vital sign measurements (including temperature, heart rate, respiratory rate, systolic blood pressure, and diastolic blood pressure) and growth parameters will be collected at each clinic visit.

A data listing of all vital sign and growth parameter measurements will be provided.


#### 9.5.2. Physical Examinations

A study clinician performed a physical examination at Visit 0. Additional examinations may have been completed at the remainder of the visits, but at the study clinician's discretion. Significant findings that met the definition of an adverse event (AE) were recorded on the AE form.

#### 9.5.3. Targeted Pulmonary Exam

Targeted pulmonary exams were conducted at randomization; Asthma Evaluation and Management Visits 4, 7, 10, 13; Cold Visits; Exacerbation Follow-up Visits; and at the Final Visit. Chest auscultation results, including inspiratory wheeze, retractions, rhonchi, and crackles, will be listed by ID and study visit. Evidence of oral candidiasis, any significant findings, and participant's discontinuation from the study will also be reported in the listing.

| ICAC | | | |
|-----------------|----------|--------|------------|
| $\{Statistical$ | Analysis | Plan - | Protocol # |

## 10. OTHER ANALYSES

No formal interim analyses of efficacy data were performed for this study.

### 11. INTERIM ANALYSES AND DATA MONITORING

The DSMB received annual periodic safety reports on enrolled and randomized participants. However, no formal interim analysis of safety data was conducted.

| ICAC {Statistical Analysis Plan - Protocol #} | |
|---|---|
| 12. | CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL |

## 13. REFERENCES

| 1. | Wildfire JJ, Gergen PJ, Sorkness CA, et al. Development and validation of the Composite Asthma Severity Indexan outcome measure for use in children and adolescents. J Allergy Clin Immunol 2012;129:694-701. |
|---|---|
| 2. | Ortega HG, Liu MC, Pavord ID, et al. Mepolizumab Treatment in Patients with Severe Eosinophilic Asthma. The New England journal of medicine 2014. |
| 3. | Brown SG. Clinical features and severity grading of anaphylaxis. J Allergy Clin Immunol 2004;114:371-6. |
| 4. | Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics 1975;31:103-15. |

ICAC

{Statistical Analysis Plan - Protocol #}

- 14. APPENDIX
- 14.1. Study Flow Chart
- 14.2. Schedule of Events

ICAC {Statistical Analysis Plan - Protocol #}

| | Scree-<br>ning | Rand<br>omiz<br>ation | omiz ation Treatment Phase (12 months) | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Asthma N | /lanageme | nt | | | | | | |
| Week | 0 | 4 | 8 | | | | | | | | | | | | | PRN | |
| Visit | V0 | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12 | V13 | V14 | Cold+ | EX# |
| Consent/Assent | + | | | | | | | | | | | | | | | | |
| Medicalhistory | + | | | | | | | | | | | | | | | | |
| Asthma Eval & Mgt | + | + | | | + | | | + | | | + | | | + | + | | |
| Asthma Counseling | + | + | | | + | | | + | | | + | | | + | + | | |
| Spirometry | + | + | | | + | | | + | | | + | | | + | + | + | + |
| IOS | | + | | | + | | | | | | | | | + | | + | + |
| Bronchodilator<br>reversibility (Spiro &<br>IOS) | | + | | | + | | | | | | | | | + | | | |
| CASI | + | + | | | + | | | + | | | + | | | + | + | | |
| ACT/c-ACT | + | + | | | + | | | + | | | + | | | + | + | | |
| Physician-patient global assessment tool | | | | | | | | | | | | | | | + | | |
| Physical Exam | + | | | | | | | | | | | | | | | | |
| Targeted pulmonary exam | | + | | | + | | | + | | | + | | | + | + | + | + |
| Lungsassessment | | | + | + | | + | + | | + | + | | + | + | | | | |
| FeNO | | + | | + | | | | + | | | + | | | | + | + | |
| SQ study drug/plaœbo | | + | + | + | + | + | + | + | + | + | + | + | + | + | | | |
| Pregnancy test | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | | |
| Urinary cotinine | | + | | + | | | | | | | | | | | + | + | + |
| Blood collection | + | + | | + | | | | | | | + | | | | + | + | + |
| CBC with differential | + * | + | | + | | | | | | | + | | | | + | + | + |
| Blood chemistry | + | | | + | | | | | | | | | | | + | | |
| Serum total IgE & specific IgE | + | | | | | | | | | | | | | | + | | |
| Blood markers<br>(plasma/RNA/DNA) | | + | | + | | | | | | | | | | | + | + | + |
| Antibodiesto drug | | + | | + | | | | | | | | | | | + | | |
| Skin Testing | +* | | +* | +* | +* | | | | | | | | | | | | |

## 

ICAC {Statistical Analysis Plan - Protocol #}

| Nasal lavage | | + | | + | | | | | | | | | | | + | + | + |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Nasosorption | | | | | | | | | | | | | | | + | + | + |
| Nasal blow | | + | + | + | + | + | + | + | + | + | + | + | + | + | + | | |
| Nasal resp virus | | + | + | + | + | + | + | + | + | + | + | + | + | + | + | | |
| Nasal ECP | | + | + | + | + | | | + | | | | | | | + | | |
| Nasal swab collection^ | | | | | | | | | | | | | | | | + | + |
| Nasal epithelial cell collection | | | | | | | | | | | | | | | +** | | |
| Sputum Induction | | | | | | | | | | | | | | | +** | | |
| Vital signs and growth parameters | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + |
| Adverse event assessment | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + |
| Concomitant medication assessment | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + | + |